#### Bond Avillion 2 Development LP

#### **Clinical Study Protocol**

Drug Substance Budesonide/Albuterol Sulfate

(BDA)

Study Code AV003

EudraCT Number 2018-003673-10

Version Version 4.0, Final

Date 08 April 2021

A Long-term, Randomized, Double-blind, Multicenter, Parallel-group,
Phase III Study Evaluating the Efficacy and Safety of PT027 Compared
to PT007 Administered as Needed in Response to Symptoms in
Symptomatic Adults and Children 4 Years of Age or Older with Asthma

Sponsor: Bond Avillion 2 Development LP,

#### VERSION HISTORY

#### Version 4.0, 08 April \$2021

Global amendment to clarify analysis of all efficacy parameters within the primary database lock and following of remaining pediatric patients exposure up-to 24 weeks for safety only within the final database lock. Removal of reversibility requirement at Visit 1 for 4 to 11 year olds. Adjustment to presentation of Inhaled Corticosteroids and administrative changes.

#### Version 3.0, 21 July 2020

Collaboration of the control of the

to incorporate temporary measures taken to protect subject and site staff safety during the COVID-19 pandemic (Appendix N). Details are provided in the Summary of Changes.

#### Version 2.0, 29 July 2019

...d provide n
...on of the de fact
...onal Conference on H.
...dhe Asthma Quality of Life
...de Questionnaire, and Asthma C
...ded in the Summary of Changes.
...ded in the Sum clarifications and updates to the study, including the addition of the de facto estimand at treatment policy strategy defined in the draft International Conference on Hamiltonian and analysis.

#### CLINICAL STUDY PROTOCOL SYNOPSIS

A Long-term, Randomized, Double-blind, Multicenter, Parallel-group, Chapter and Safety of PT027 Company To07 Administered as Needed in Response to Chapter A No. Phase III Study Evaluating the Efficacy and Safety of PT027 Compared to PT007 Administered as Needed in Response to Symptoms in Symptomatic Adults and Children 4 Years of Age or Older with Asthma (MANDALA)

## International coordinating investigators

Study site(s) and number of subjects planned

Approximately 380 study sites are anticipated to randomize approximately 3000 adult and adolescent subjects with noderate to severe asthma to 1 of 3 treatment groups (approximately 1000 subjects per group. In addition, up to 100 subjects in the 4 to 11-year age group with moderate to severe asthma will be randomized with approximately 50 subjects randomized to the albuterol sulface (here after referred to as albuterol) metered-dose inhaler (AS MDI) and 50 subjects randomized to the low dose budesonide/albuterol metered-dose inhaler (BDA) MDI) groups only. Approximately 6000 subjects will need to be screened, assuming an estimated Freen failure rate of 30% to 50%.

This hase III study is planned to be conducted globally.

#### Study design

This is a randomized, double-blind, multicenter, parallel-group, variable-length, event-driven study with a treatment period of at least 24 weeks for each subject. The purpose of this study is to compare 2 doses of BDA MDI with AS MDI on the time to first severe asthma exacerbation in adult, adolescent, and pediatric subjects with moderate to severe asthma defined by Global Initiative for Asthma (GINA). Subjects will administer randomized investigational product (IP) as needed (prn) in response to asthma symptoms.

Subjects meeting all entry criteria at the screening visit (Visit 1/1a, as applicable) will enter a 14-to 28-day screening period. (Subjects may consent for the study in advance of Visit 1 and if required, request for medical records to support evidence of prior exacerbations without triggering the 28-day screening period.) If a severe exacerbation event occurs during the screening period, the screening period may be extended to a maximum of 9 weeks. Screened subjects will continue to take their regular asthma maintenance therapy throughout the study (from Visit 1 through the treatment period). At Visit 1, eligible subjects will discontinue their usual prn inhaled product used as-needed for symptom relief and begin Sponsor-provided Ventolin to be used prn in response to symptoms or prior to exercise during the screening period only. Subjects will be asked to turn in their own is trailed reliever products to the investigational sites for storage until the individual subject last study visit. Eligible subjects will be randomized at Visit 2.

#### Objectives

| Primary Objective: | Primary Endpoint: |
|---|---|
| To evaluate the efficacy of budesonide/albute of metered-dose inhaler 80/180 μg and 160(180 μg administered prn in response to symptotic compared to albuterol metered-dose inhaler 180 μg | Time to first severe asthma exacerbation |
| Secondary Objective: | Secondary Endpoint: |
| To characterize the effect of udesonide/albuterol metered-dose inhaler 80/180 µg and 160/180 µg administered prn in response to symptoms compared to albute of metered-dose inhaler 180 µg | <ul> <li>Severe exacerbation rate (annualized)</li> <li>Total systemic corticosteroid exposure over the treatment period</li> <li>Asthma Control Questionnaire -5 (ACQ-5) change from baseline and responder analysis at Week 24</li> <li>Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12)/Pediatric Asthma Quality of Life Questionnaire (PAQLQ) change from baseline and responder analysis at Week 24</li> </ul> |
| offety Objective: | Safety Endpoints: |

To evaluate the safety and tolerability of Adverse events/serious adverse events budesonide/ albuterol metered-dose inhaler Vital signs 80/180 µg and 160/180 µg administered prn in Clinical chemistry and hematology parameters response to symptoms compared to albuterol Electrocardiogram metered-dose inhaler 180 μg Exploratory Objective: **Exploratory Endpoints:** To characterize the effect of budesonide/albuterol Asthma Control Questionnaire -5 change from metered-dose inhaler 80/180 µg and 160/180 µg baseline and responder analysis at Week d administered prn in response to symptoms Asthma Control Questionnaire-5 change compared to albuterol metered-dose inhaler 180 baseline and responder (3-factor) and vsis at Week 12 and Week 24 Asthma Quality of Life Questionnaire for 12 years and older/Pediatric Asthma unality of Life Questionnaire change from baseline and responder analysis at Week 12 d∰hma (annualized rate and time Change from Saseline in prebronchodilator forced expiratory blume in 1 second at Week 12 and Week ng and evening peak expiratory flow Asthma daytime/night-time symptoms

Time to treatmont 2:of investigational product (reliever therapy) Time to treatment discontinuation or change in maintenance therapy Asthma Control Test (ACT) or Childhood Asthma Control Test (C ACT) change from baseline and responder analysis at Week 24 Percentage of "as needed"-free days Percentage of symptom-free days Percentage of asthma control days Inhaled corticosteroid exposure over the treatment period

#### Target subject population

The study will enroll subjects ≥4 years of age in all countries with the exception of the following:

- In Serbia, only subjects ≥12 years of age will be enrolled.
- In Germany, Slovakia and Ukraine, only subjects ≥18 years of age will be enrolled.

Age-specific assessments will be implemented where relevant for the population enrolled.

Duration of study/treatment

The study will consist of 3 periods:

Screening period (14 to 28 days), except where a severe asthma as the ast of more than a severe asthma as a policial of the screening period more than the screening period more than the severe asthma as a policial of the severe asthma exacerbation within the previous at least 1 severe asthma exacerbation within the previous are provided to severe as the severe asthma exacerbation within the previous are provided to severe as the severe

- consent for the study in advance of Visit 1 and if required, request for medical records to support evidence of prior exacerbations without triggering the 28-day screening period.)
- Treatment period of at least 24 weeks. The study treatment period will continue (extension phase) until the required 570 first severe; accerbation events, as defined per protocol, have been reached and the last adult subject has completed 24 weeks of treatment, which will be defined as the prinary completion date (PCD). Paediatric subjects will continue until 24 weeks of treatment have been reached for each paediatric patient, defined as the final completion date.
  - In the event 570 events are captured before the last adult patient has had 24 weeks of treatment, alk subjects on treatment for ≥24 weeks will have their endof-study (EOS) visit at their next scheduled clinic visit. All subjects on treatment for < 24 weeks will continue until 24 weeks at which point they will complete their EOS isit
  - In the event 570 events will be captured after the last subject has had 24 weeks of treatment, each subject will return to complete the EOS visit at their next scheduled ckinic visit
- Safety follow-up period: where a safety follow-up telephone contact will occur 2 weeks (±4 days) after EOS or premature discontinuation visit (PDV), whichever occurs firs

The study will be completed when the last subject has completed his or her post-study follow-up telephone contact. Subjects who discontinue IP will complete a PDV, and adverse will be or first subject enrolled: Q4 2018.

Frommated date of last subject completed: Q1 2022. events (AEs)/serious adverse events (SAEs) will be followed up if medically indicated.

#### Investigational product, dosage, and mode of administration

BDA MDI is formulated as both micronized budesonide and micronized albuterol co-suspended with spray-dried porous particles in a hydrofluoroalkane (HFA) propellant. The co-suspension formulation ensures that subjects receive a consistent delivery of the drug from each actuation of the MDI.

Investigational product will be used in response to asthma symptoms as they would normally take their reliever medication. If subjects take IP in advance of exercise for the prevention of exercise induced symptoms, IP usage in relation to exercise will be captured within the eDiary. No other reliever products will be used during the treatment period.

At randomization (Visit 2), adolescents and adults (aged ≥12 years) who meet the eligibility criteria will be randomly assigned to 1 of the following 3 treatment grows in a 1:1:1 ratio as reliever therapy on top of usual care. Children aged 4 to 11 years will be randomized in a 1:1 ratio only to the lower BDA MDI dosage or AS MDI:

- BDA MDI 80/180 μg (given as 2 actuations of BDA MDI 40/90 μg per puff) prn
- BDA MDI 160/180 μg (given as 2 actuations of BDA MDI 80/90 μg per puff) prn
- AS MDI 180 μg (given as 2 actuations of ΔS MDI 90 μg per puff) prn

The maximum daily dosage of IP should not exceed 12 puffs per day.

Subjects will be recommended not to take prove than 8 puffs per day and advised to contact the study site/investigator if their symptotic necessitate more than 8 puffs in a day.

In order to ensure safety and monitor daily teatment status, all subjects will be provided with an electronic diary (eDiary: AM3 decice). The eDiary transfers data every 24 hours across a range of asthma symptom scores and daily usage (ie, number of puffs inhaled) to assess a subject's asthma status. Subjects will use the eDiary for reporting daily use of IP and any symptoms. If symptoms and/or daily dosage exceed a protocol-specified threshold, the eDiary will generate an alert to the subject and the investigational site. In this way, daily IP usage will be monitored closely by the investigators and medical monitors to assess any worsening of subject status. Action will be taken where clinically indicated.

#### Statistical methods

#### Sample size calculation

A sample size of 1000 adult and adolescent subjects per treatment group and observation of the 570 first severe exacerbation events provides this study with 87% power to observe a 25% reduction in the risk of severe exacerbation with at least 1 dose of BDA MDI versus AS MDI assuming the Hochberg procedure (Hochberg 1988) for multiple testing and a 2-sided argnificance level of 5%.

In addition, up to 100 subjects in the 4 to 11-year age group with moderate to severe asthma will be randomized with approximately 50 subjects randomized to the AS MDI group and 50 subjects randomized to the low dose BDA MDI group only.

#### Primary efficacy analysis

The primary variable, time to first severe asthma exacerbation, will be analyzed using a Cox proportional hazards regression model to compare treatment arms. The model will be adjusted for the randomization stratification factors (age group [≥ 4 to 11, ≥12 to 17, ≥18] Pregion (North America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to screening (Visit 1) plus any severe exacerbation event experienced during the screening period and key covariates of interest with more detail to be provided in the statistical adalysis plan (SAP). The 2 primary treatment comparisons will be 2-sided with the 5% overall alpha level controlled using the Hochberg procedure. The primary efficacy analysis will include all data up to the primary outcome database lock (pDBL), scheduled to occur following the PCD and once all randomized adults have attended their EOS visit.

#### Secondary efficacy analyses

Annualized severe asthma exacerbation rate will be analyzed using negative binomial regression to compare treatment groups. The reasonse variable in the model will be the number of severe asthma exacerbations. The model will adjust for (age group  $[\ge 4$  to  $11, \ge 12$  to  $17, \ge 18]$ ); region (North America Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to screening (Visit 1) plus any severe exacerbation event experienced during the screening period and key covariates of interest with more detail to be provided in the SAP.

Responder variables for Asthraa Control Questionnaire-5 (ACQ-5) and Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12)/ Pediatric Asthma Quality of Life Questionnaire (PAQLQ) at Week 24 will each be analyzed using a logistic regression model to compare treatment groups. The model will be adjusted for the randomization stratification factors and key covariates as described above.

The total systemic corticosteroid (SCS) exposure as total annualized dose of SCS (mg/year) will be presented descriptively by treatment. A comparison in total annualized SCS dose between EDA MDI 80/180 vs AS MDI 180 and BDA MDI 160/180 vs AS MDI 180 will be analyzed using a Wilcoxon rank sum test and associated p-values will be presented along with the descriptive summary.

If both doses of BDA MDI are statistically superior to AS MDI for the primary endpoint, the full alpha will be available to pass to the family of secondary endpoints.

The type-I error will be controlled for secondary endpoints.

estimand in the following sequential order, grouped by secondary endpoint:

Annualized severe exacerbation rate

- BDA MDI 160/180 μg versus AS MDI 180 μg
- BDA MDI 80/180 μg versus AS MDI 180 μg

Total annualized dose of systemic corticosteroid

- 3. BDA MDI 160/180 μg versus AS MDI 180 μ
- BDA MDI 80/180 μg versus AS MDK 8

Asthma Control Questionnaire-5 (AC hange from baseline responder analysis at Week 24

- BDA MDI 160/180 μg versus MDI 180 μg
- BDA MDI 80/180 μg verχ AS MDI 180 μg

Asthma Quality of Life Questonnaire for 12 years and older (AQLQ+12) change from baseline responder analysis at Week 24

- BDA MDI 1669180 μg versus AS MDI 180 μg
- 8. BDA MD 80/180 μg versus AS MDI 180 μg

Statistical tests for the secondary analyses will be conducted at the 5% level of significance (2-sided) Inference for a test in the defined order is dependent on statistical significance having been achieved in the preceding tests, if this is not achieved then nominal p-values will exclude the exclude all ages. be provided. As per the primary analysis, comparisons of BDA MDI 160/180 versus AS MDI exclude the pediatric population, whilst comparisons of BDA 80/180 versus AS MDI will

Statistical significance can only be claimed on the key secondary endpoints if a statistically significant treatment effect is observed on both BDA MDI 160/180  $\mu g$  and BDA MDI 80/180  $\mu g$  versus AS MDI for the primary endpoint of time to first severe exacerbation. The secondary efficacy analyses will include all data up to the pDBL.

#### Estimands

Three estimands are of interest in this study:

The primary estimand of interest is the efficacy estimand, defined as the effect of the randomized treatment in all subjects assuming continuation of randomized treatment for the duration of the study, regardless of actual usage and assuming that maintenance therapy is not changed. This estimand could be considered as a while-on-treatment strategy or a hypothetical strategy as defined in the draft International Conference on Harmonization (ICH) E9 Addendum.

The second estimand of interest is the attributable estimand, defined as the effect of treatment in subjects attributable to the randomized treatment assuming that maintenance therapy is not changed. For this estimand, discontinuation of randomized treatment for tolerability or change in maintenance therapy for lack of asthma control is considered a negative outcome. This estimand is a mixture of composite and hypothetical strategies as defined in the draft ICH E9 addendum.

The third estimand of interest is the effectiveness estimand which is a combination of the hypothetical and treatment policy strategies as defined in the draft ICH E9 addendum. The strategy is hypothetical in that the treatment effect will be estimated without collecting data post the intercurrent event of discontinuation from randomized treatment. However, the strategy is consistent with the treatment policy strategy in that the treatment effect is estimated irrespective of the occurrence of the intercurrent event of a change in the maintenance therapy.

The fourth estimand of interest is the de facto estimand, defined as the effect of a treatment policy regardless of occurrence of intercurrent event; changes in maintenance therapy or premature discontinuation of randomized treatment. This estimand is considered a treatment policy strategy as defined in the draft ICH E9 addendum.

#### TABLE OF CONTENTS

| Clinical St | udy Protocol | 1 |
|---|---|---|
| TITLE PA | GE | 1 |
| VERSION | HISTORY | . 6 |
| CLINICAL | HISTORY STUDY PROTOCOL SYNOPSIS F CONTENTS BBREVIATIONS AND DEFINITION OF TERMS INTRODUCTION Background and rationale for conducting this study Rationale for study design, doses, and control groups Benefit/risk and ethical assessment Study design Study governance and oversight Independent data monitoring committee Adjudication committee STUDY OBJECTIVES Primary objective Secondary objective Safety objective Exploratory objective SUBJECT SELECTION, ENROLLMENT, RANDOMIZATION, RESTRICTIONS, TREATMENT DISCONTINUATION, AND STUDY TERMINATION Inclusion criteria | VO3 |
| TABLEO | F CONTENTS. | 0 |
| TABLE OF | PROPERTY THOUGH AND DEED HERON OF TERMS | 11 |
| LIST OF A | BBREVIATIONS AND DEFINITION OF TERMS | 17 |
| 1 | INTRODUCTION O | 19 |
| 1.1 | Background and rationale for conducting this study | 19 |
| 1.2 | Rationale for study design, doses, and control groups | 20 |
| 1.3 | Benefit/risk and ethical assessment | 21 |
| 1.4 | Study design | 22 |
| 1.5 | Study governance and oversight | 24 |
| 1.5.1<br>1.5.2 | Independent data monitoring committee | 24 |
| 1.5.2 | Adjudication commune 2 | 23 |
| 2 | STUDY OBJECTIVES | 25 |
| 2.1 | Primary objective | 25 |
| 2.2 | Secondary objective | 25 |
| 2.3 | Safety objective | 26 |
| 2.4 | Exploratory objective | 26 |
| 3 | SUBJECT SELECTION, ENCOLLMENT, RANDOMIZATION, | |
| | RESTRICTIONS, TREATMENT DISCONTINUATION, AND STUDY TERMINATION | 27 |
| 3.1 | Inclusion criteria | 27 |
| 3.2 | ^ | |
| 3.3 | Exclusion criteria | |
| | Procedures for Randling incorrectly enrolled or randomized subjects | |
| 3.4 | Methods for assigning treatment groups | 33 |
| 3.5 | . 🗸 | |
| 3.6 | Methods for ensuring blinding | |
| 3.7 | Methods for unblinding | |
| 3.8 | ~ | |
| 3.9 | Reatment discontinuation by subject and/or Sponsor | |
| 3.10 | Study termination | |
| 3.10 11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | Screen failures | |
| 4100 | STUDY PLAN AND TIMING OF PROCEDURES | |
| <b>€</b> M | Screening and run-in period | |
| 4.2 | Randomization/treatment period/extension phase | 43 |

| 4.3 | End-of-study visit | 44 |
|---|---|---|
| 4.4 | Unscheduled visit and premature discontinuation visit | 45 |
| 4.5 | Safety follow-up period | 45 |
| 4.6 | Follow-up | 45 |
| 5 | STUDY ASSESSMENTS Efficacy assessments Asthma exacerbation definition Definition of asthma signs/symptoms worsening Investigator-justified asthma exacerbations Severe asthma exacerbations Treatment for severe asthma exacerbations Onset and duration of asthma exacerbations Approach for capturing asthma exacerbations Asthma Quality of Life Questionnaire+12/Pediatric Asthma Quality of Life Questionnaire | .46 |
| 5.1 | Efficacy assessments | 96 |
| 5.1.1 | Asthma exacerbation definition | 46 |
| 5.1.1.1 | Definition of asthma signs/symptoms worsening | 46 |
| 5.1.1.2 | Investigator-justified asthma exacerbations | 47 |
| 5.1.1.3 | Severe asthma exacerbations | 47 |
| 5.1.1.4 | Treatment for severe asthma exacerbations | 47 |
| 5.1.1.5 | Onset and duration of asthma exacerbations | 48 |
| 5.1.1.6 | Approach for capturing asthma exacerbations | 48 |
| 5.1.2 | Asthma Quality of Life Questionnaire+12/Pediatric Asthma Quality of Life | |
| | Questionnaire | 49 |
| 5.1.2.1 | Asthma Quality of Life Questionnaire+12 | 49 |
| 5.1.2.2 | Pediatric Asthma Quality of Life Questionnaire | 50 |
| 5.1.3 | Asthma Control Questionnaire-5 and -7 | 50 |
| 5.1.4 | Asthma Control Test | 51 |
| 5.1.5 | Pediatric Asthma Quality of Life Questionnaire— Asthma Control Questionnaire—5 and -7 Asthma Control Test Childhood Asthma Control Test eDiary Peak expiratory flow Use of investigational product (relieved therapy) | 51 |
| 5.1.6 | eDiary | 51 |
| 5.1.6.1 | Peak expiratory flow | 51 |
| 5.1.6.2 | Use of investigational product (relieve wherapy) | 52 |
| 5.1.6.3 | eDiary maintenance therapy compliance | 52 |
| 5.1.6.4 | eDiary maintenance therapy computative eDiary recording of asthma symptoms Deterioration of asthma Lung function measurement by spirometry Reversibility Test | 52 |
| 5.1.7 | Deterioration of asthma | 53 |
| 5.1.8 | Lung function measurement spirometry | 53 |
| 5.1.8.1 | Reversibility Test | 54 |
| 5.1.8.2 | COVID-19 and Pulmonary Function Testing | 54 |
| 5.2 | Safety assessments | 54 |
| 5.2.1 | Laboratory safety assessments | 55 |
| 5.2.2 | Resting 12-lead Dectrocardiogram | |
| 5.2.3 | Vital sign measurements | 56 |
| 5.2.4 | Adverse event assessments | 56 |
| 5.3 | Other assessments | 56 |
| 5.3.1 | Physica examination | 56 |
| 5.3.2 | Concomitant medications | 57 |
| 5.4 | Parmacokinetics | 57 |
| 5.5 | Pharmacodynamics | 57 |
| 5.6 KIN | Genetics | 57 |
| 5.7 | Biomarker analysis | 57 |
| Silve | Other assessments Physical examination Concomitant medications Pharmacokinetics Pharmacodynamics Genetics Biomarker analysis SAFETY REPORTING AND MEDICAL MANAGEMENT Definition of adverse events | 58 |
| <b>3</b> 6.1 | Definition of adverse events | 58 |

| 6.2 | Definitions of serious adverse event | 58 |
|---|---|---|
| 6.3 | Recording of adverse events | 59 |
| 6.3.1 | Period for collection of adverse events | 59 |
| 6.3.2 | Follow-up of unresolved adverse events | 59 |
| 6.3.3 | Variables | 59 |
| 6.3.4 | Causality collection | <b>6</b> 6 |
| 6.3.5 | Deteriorations of asthma and severe asthma exacerbations | Y0 |
| 6.3.6 | Adverse events based on signs and symptoms | 60 |
| 6.3.7 | Adverse events based on examinations and tests | 61 |
| 6.3.8 | Hy's Law | 61 |
| 6.3.9 | COVID-19 Adverse Events | 62 |
| 6.4 | Variables Causality collection Deteriorations of asthma and severe asthma exacerbations Adverse events based on signs and symptoms Adverse events based on examinations and tests Hy's Law COVID-19 Adverse Events Reporting of serious adverse events Overdose Pregnancy Maternal exposure Paternal exposure Medication error | 62 |
| 6.5 | Overdose | 63 |
| 6.6 | Pregnancy | 63 |
| 6.6.1 | Maternal exposure | 63 |
| 6.6.2 | Paternal exposure | 64 |
| 6.7 | Medication error | 64 |
| 7 | INVESTIGATIONAL PRODUCT AND THE TREATMENTS Identity of investigational product(s) Dose and treatment regimens Labelling Storage Compliance Accountability Metered dose inhaler: handling and cleaning | 66 |
| 7.1 | Identity of investigational product(s). | 66 |
| 7.2 | Dose and treatment regimens | 66 |
| 7.3 | Labelling C. :A | 67 |
| 7.4 | Stornes | 07 |
| 7.4 | Storage | 00 |
| 7.5 | Compliance | 68 |
| 7.6 | Accountability | 68 |
| 7.7 | victored-dose limited. Hallening and creating | |
| 7.8 | Concomitant and other teatments | 69 |
| 7.8.1 | Maintenance therapies | |
| 7.8.2 | Medications that may affect reversibility and FEV1 testing | |
| 7.8.3 | Prohibited medications | |
| 7.8.4 | Other concompant treatment | 71 |
| 8 | STATISTIÇAL ANALYSES | 72 |
| 8.1 | Statistice considerations | 72 |
| 8.1.1 | Estimonds | 72 |
| 8.1.2 | Prisary outcome analysis | 73 |
| 8.1.3 | Tope 1 error control | 73 |
| 8.2 | Sample size estimate | 74 |
| 8.3 | Definitions of analysis sets | 74 |
| 8.3.1 | Full analysis set | 74 |
| 8.30 | Safety analysis set | 75 |
| <b>8</b> 24 | Statistical considerations Estimates Princerry outcome analysis Tope 1 error control Sample size estimate Definitions of analysis sets Full analysis set Safety analysis set Violations and deviations | 75 |

| 8.5 | Outcome measures for analyses | 75 |
|---|---|---|
| 8.5.1 | Primary efficacy analysis | 75 |
| 8.5.1.1 | Derivation of time to first severe asthma exacerbation | |
| 8.5.2 | Secondary efficacy analyses | 75 |
| 8.5.2.1 | Derivation of annualized severe asthma exacerbation rate | 76 |
| 8.5.2.2 | Derivation of total systemic corticosteroid exposure | 7€ |
| 8.5.2.3 | Derivation of total systemic corticosteroid exposure | <b>.</b> |
| 8.5.2.4 | Derivation of Asthma Quality of Life Questionnaire +12 and Pediatric | Asthona |
| | Ouality of Life Ouestionnaire variables | |
| 8.5.3 | Exploratory analyses | 78 |
| 8.5.3.1 | Quality of Life Questionnaire variables Exploratory analyses Derivation of deterioration of asthma variables Derivation of time to treatment discontinuation or change in maintenance. | <del>78</del> |
| 8.5.3.2 | Derivation of time to treatment discontinuation or change in maintenant | ce therapy |
| | for lack of asthma control | 78 |
| 8.5.3.3 | Derivation of Asthma Control Test responder variable | 78 |
| 8.5.3.4 | Derivation of other eDiary variables | 78 |
| 8.5.3.5 | Inhaled corticosteroid exposure | 79 |
| 0.5.5.5 | Derivation of deterioration of asthma variables. Derivation of time to treatment discontinuation or change in maintenar for lack of asthma control Derivation of Asthma Control Test responder variable Derivation of other eDiary variables. Inhaled corticosteroid exposure Methods for statistical analyses Analysis of the primary variable Analysis of the secondary efficacy variables Severe asthma exacerbation rate Asthma Control Questionnaire-5 Asthma Quality of Life Questionnaire 12 and Pediatric Asthma Quality of Life Questionnaire Total systemic corticosteroid exposure. Analysis of safety variables Adverse events Vital signs Clinical chemistry and hematology | 70 |
| 8.6 | Methods for statistical analyses | 79 |
| 8.6.1 | Analysis of the primary variable | /9 |
| 8.6.2 | Analysis of the secondary efficacy variables | 80 |
| 8.6.2.1 | Severe asthma exacerbation rate | 80 |
| 8.6.2.2 | Asthma Control Questionnaire-5 | 81 |
| 8.6.2.3 | Asthma Quality of Life Questionnaire ₩12 and Pediatric Asthma Quality | ity of Life |
| | Questionnaire | 82 |
| 8.6.2.4 | Total systemic corticosteroid exposure | 82 |
| 8.6.3 | Analysis of safety variables | 82 |
| 8.6.3.1 | Adverse events | 82 |
| 8.6.3.2 | Vital signs | 82 |
| 8.6.3.3 | | |
| 8.6.3.4 | Concomitant medication | 83 |
| 8.6.4 | Analysis of exploratory ariables | 83 |
| 8.6.4.1 | Deterioration of asthrea | 83 |
| 8.6.4.2 | Prebronchodilator PEV1 | 83 |
| 8.6.4.3 | Morning peak expratory flow | 84 |
| 8.6.4.4 | Other eDiary variables | 84 |
| 8.6.4.5 | Time to treatment discontinuation or change in maintenance therapy for | or lack of |
| | asthma compol | 84 |
| 8.6.4.6 | Asthma@ontrol Test | |
| 8.6.4.7 | Inhale corticosteroid exposure | 85 |
| 8.6.5 | Subgroup analysis | 85 |
| 8.6.6 | Sensitivity analysis | 85 |
| 8.6.6.1 | Tipping point analysis | 85 |
| 8.6.62 | Attributable estimand | 85 |
| 8668 | Subgroup analysis Sensitivity analysis Tipping point analysis Attributable estimand Effectiveness estimand | 85 |
| 8 6.604 | De facto estimand | 86 |
| 8665 | COVID-19 pandemic impacts | |
| 8.6. <b>6</b> .4<br>8 <b>3</b> 5.6.5 | • | |
| 79 | STUDY AND DATA MANAGEMENT | 87 |

| 9.1 | Training of study site staff | 87 |
|---|---|---|
| 9.2 | Monitoring of the study | 87 |
| 9.2.1 | Source data | |
| 9.2.2 | Study agreements | |
| 9.2.3 | Archiving of study documents | 88<br> |
| 9.3 | Study timetable and end-of-study | <b>&amp;</b> 8 |
| 9.4 | Data management | \$.89 |
| 10 | Data management | 91 |
| 10.1 | Ethical conduct of the study | 91 |
| 10.2 | Subject data protection | 91 |
| 10.3 | Ethics and regulatory review | 91 |
| 10.4 | Informed consent/assent | 92 |
| 10.5 | Changes to the clinical study protocol and informed consent assent form | 92 |
| 10.6 | 71 | 93 |
| 11 | | 94 |
| 12 | SUMMARY OF CHANGES | 96 |
| 12.1 | Changes made to Version 3.0 | 96 |
| 12.2 | Changes made to Version 2.0 | 99 |
| 12.3 | Changes made to Version 1.0 | .105 |
| APPENDE | LIST OF REFERENCES SUMMARY OF CHANGES Changes made to Version 3.0 Changes made to Version 2.0 Changes made to Version 1.0 X A, AVILLION PROTOCOL SIGNATURE PAGE | .112 |
| APPENDD | X B, PRIMARY INVESTIGAÇORSIGNATURE PAGE | .113 |
| APPENDE | X C, GLOBAL INITIATIVE FOR ASTHMA (GINA, 2018) | .114 |
| APPENDE | X D, ADDITIONAL SAFETT INFORMATION | .116 |
| APPENDE | X E, HY'S LAW | .119 |
| APPENDE | X F, ASTHMA QUALTY OF LIFE +12 QUESTIONNAIRE | .124 |
| APPENDE | X G, PEDIATRIC ASTHMA QUALITY OF LIFE QUESTIONNAIRE | .130 |
| APPENDE | X H, ASTHMACONTROL QUESTIONNAIRE-5 AND -7 | .135 |
| APPENDE | XI, ASTHMA CONTROL TEST | .144 |
| APPENDE | X J, CHIEDHOOD ASTHMA CONTROL TEST | .145 |
| APPENDE | X K, LIST OF E-DIARY QUESTIONS | .146 |
| APPENDE | X & METERED-DOSE INHALER HANDLING AND CLEANING | .148 |
| APPEND | M, SPIROMETRY ASSESSMENT CRITERIA | .155 |
| APPENDE | X N, COVID-19 EMERGENCY MEASURES PERMITTED TO ENSURE | |
| nentin | SUBJECT SAFETY | .157 |

# 

#### LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

The following abbreviations and special terms are used in this Clinical Study Protocol.

| Abbreviation or special term | Asthma Control Questionnaire-5 Asthma Control Questionnaire-7 Asthma Control Test adverse event |
|---|---|
| ACQ-5 | Asthma Control Questionnaire-5 |
| ACQ-7 | Asthma Control Questionnaire-7 |
| ACT | Asthma Control Test |
| AE | adverse event allergy immunotherapy alanine aminotransferase (or alanine transaminase) |
| AIT | allergy immunotherapy |
| ALT | alanine aminotransferase (or alanine transaminase) |
| AQLQ+12 | Acthma Quality of Life Questionnaire for 12 years and older |
| AS MDI (PT007) | albuterol sulfate metered-dose inhaler aspartate aminotransferase |
| AST | aspartate aminotransferase |
| BDA | budesonide/albuterol |
| BDA MDI (PT027) | budesonide/albuterol metered-dose inhatel |
| β-hCG | β-human chorionic gonadotroκία 🔊 |
| BMI | body mass index |
| C ACT | Childhood Asthma Control T-9 |
| EC | aspartate aminotransferase budesonide/albuterol budesonide/albuterol metered-dost inhatel β-human chorionic gonadotrotuit body mass index Childhood Asthma Control Test Ethics Committee adionactions to Institutional Review Board (IRB) and Independent Ethics Committee (IEC) |
| ECG | electrocardiogram |
| eCRF | electronic case port form |
| EOS | end-of-study. |
| ePRO | electronic patient reported outcome |
| FAS | full analysis set |
| FEV <sub>1</sub> | fored expiratory volume in 1 second |
| _ | Corred vital capacity |
| GCP 50 | Good Clinical Practice |
| GCP<br>GINA | Global Initiative for Asthma |
| GMP © | Good Manufacturing Practice |
| HFA 💍 | hydrofluoroalkane |
| HL & | Hy's Law |
| ICF KN | informed consent form |
| ICIFC | International Conference on Harmonization |
| GINA GMP HFA HL ICF ICF ICS | inhaled corticosteroid |
| IDMC | Independent Data Monitoring Committee |

| Abbreviation or special term | Explanation |
|---|---|
| International<br>Coordinating investigator | If a study is conducted in several countries, the International Coordinating Investigator is the investigator coordinating the investigators and/or activities internationally. |
| IP | investigational product |
| IWRS | Interactive Web Response System |
| LABA | long-acting β2-agonist |
| LAMA | long-acting muscarinic antagonist |
| LTRA | leukotriene receptor antagonist |
| MDI | metered-dose inhaler |
| med | medium |
| MID | metered-dose inhaler medium minimal important difference |
| MMRM | mixed model repeated measures oral corticosteroids |
| OCS | oral corticosteroids |
| PAQLQ | Pediatric Asthma Quality of Life Question are |
| PCD | primary completion date |
| PDV | premature discontinuation visit |
| PEF | Pediatric Asthma Quality of Life Questioning primary completion date premature discontinuation visit peak expiratory flow pulmonary function test Potential Hy's Law as needed |
| PFT | pulmonary function test |
| PHL | Potential Hy's Law |
| Pm | as needed |
| SABA | short/rapid-acting \$2-adrenoreceptor agonist |
| SAMA | short-acting mascarinic antagonist |
| SAE | serious adverse events |
| SAP | Statistical Analysis Plan |
| SCS | systemic corticosteroids |
| SMART | mbicort is approved for maintenance and reliever therapy |
| TBL | ototal bilirubin |
| TC & | telephone call |
| ULN 5 | upper limit of normal |
| TBL TC ULN WBDC | Web Based Data Capture |

#### 1 INTRODUCTION

#### 1.1 Background and rationale for conducting this study

Bond Avillion 2 Development LP (Sponsor) is developing budesonide/albuterol sulfate (PT027) hereafter referred to as budesonide and albuterol metered-dose inhaler [BDA MDI] and albuterol sulfate (hereafter referred to as albuterol [AS MDI]) pressurized inhalation suspension products in adults and children 4 years of age or older with asthma. Please refer to the current Investigator Brochure (2019) for additional information.

Albuterol is a short/rapid-acting β2-adrenoreceptor agonist (SABA), inducing airway smooth muscle relaxation and reducing or preventing bronchoconstriction. Albuterol is approved in many countries in multiple formulations for treatment or prevention of bronchoconstriction, and is also known under the generic name of salbutamol. In clinical practice, albuterol is used as an as needed (prn) reliever therapy (Global Initiative for Asthma [GINALV018).

Budesonide is a well-established anti-inflammatory corticosteroid that exhibits potent glucocorticoid and weak mineralocorticoid activity and is approved worldwide in orally inhaled formulations for the treatment of asthma and chronic obstructive pulmonary disease both as a mono-product and in combination with a long/rapid-seting 32-agonist (LABA, formoterol).

In vitro studies have demonstrated that inhaled strong (ICS) agents potentiate the effects of SABAs in reducing airway smooth muscle fone (Mendes 2008) and can reverse adrenergic receptor tolerance and desensitization (Cooler and Panettieri 2008). Clinically, similar functional potentiation with combined ICSs and attacked has been observed in patients with asthma for functional measures of airway smooth muscle and airway blood flow (Mendes 2015). An analysis of 425 asthma exacerbations in attents from the FACET study (Tattersfield 1999) revealed that asthma symptoms and acreased reliever therapy use were noted over several days before the start of an asthma exacerbation. Combining the use of a SABA (albuterol) with budesonide in the proposed budesonide and albuterol metered-dose inhaler (BDA MDI) combination product should not only provide rapid bronchodilation, but also treat worsening airway inflammation by the addition of the budesonide component. Per current treatment guidelines (GINA 2013), ICS/formoterol maintenance and reliever can be used in patients with moderate or severe ashma. Studies of budesonide and a rapid-acting LABA (formoterol) as reliever have demonstrated enhanced protection from severe exacerbations in patients already receiving combination therapy for maintenance without an increase in adverse effects (Rabe 2006; O'Byp 2005). In addition, budesonide/formoterol as maintenance and reliever significantly reduced severe exacerbation risk in pediatric patients (O'Byrne 2007).

In some markets, Symbicort Turbuhaler (hereafter referred to as Symbicort) is approved for maintenance and reliever therapy (SMART). With SMART application, patients with asthma use symbicort as maintenance inhalation medication and also prn in response to symptoms. The simultaneous administration of budesonide with formoterol when symptoms occur ensures that

patients with asthma receive both a rapid-acting bronchodilator for symptom relief and antiinflammatory medication to treat their persistent airway inflammation. It is important to note that
the prn administration of ICS in this treatment regimen is not expected to significantly increase
overall steroid load (mostly because of a reduction in the number of severe exacerbation
episodes, resulting in fewer patients requiring systemic corticosteroid (SCS) doses as acute
treatment). BDA MDI is proposed to be available prn for symptom control to all patients with
asthma, regardless of maintenance therapy.

When patients use the BDA MDI products as needed in response to asthma symptoms, it is expected that their risk of experiencing an asthma exacerbation will be lower than in subjects using albuterol alone.

#### 1.2 Rationale for study design, doses, and control groups

The study will compare BDA MDI at 2 different doses with AS MDI adults and children 4 years of age or older with moderate to severe asthma.

The clinical standard of care for subjects with moderate to severe asthma is a medium-to-high-dose ICS or low-to-high-dose ICS incombination with LABA, with a SABA such as albuterol to use prn in response to symptoms (ie reliever therapy). When subjects require frequent reliever therapy, additional anti-inflammators medication may provide benefit by early reaction to increased asthma symptoms that are reflective of an incipient severe exacerbation. BDA MDI would prevent or reduce bronche constriction and provide additional anti-inflammatory medication when needed at the same of symptoms. Safety and efficacy of BDA MDI will be compared with AS MDI because albuterol is the standard of care reliever therapy in response to symptoms.

The objective of this randomized, dealer-blind, multicenter, parallel-group study is to evaluate, within a typical design for the development of new asthma therapies, the benefit of BDA MDI administered prn in response to symptoms in adults and children 4 years of age or older with moderate to severe asthma receiving medium-to-high-dose ICS or low-to-high-dose ICS in combination with LABA, with or without an additional controller therapy (leukotriene receptor antagonist [LTRA], long-acting muscarinic antagonist [LAMA] or theophylline).

The primary endpoint is the time to first severe asthma exacerbation, and secondary endpoints include the annualized severe exacerbation rate and asthma symptom control as measured by Asthma Control Questionnaire-5 (ACQ-5).

The treatment duration for the study will be at least 24 weeks for each subject to support the subject exposure data. The study treatment period will continue (extension phase) until the required 570 first severe exacerbation events, as defined per protocol, have been reached and the sist adult subject has completed 24 weeks of treatment, which will be defined as the primary

completion date (PCD). Not all pediatric subjects will have 24 weeks of treatment at time of PCD.

Two dosage levels of BDA MDI, 80/180 µg and 160/180 µg (given as 40/90 µg and 80/90 µg, respectively, per actuation), are included in this study to support final dose selection for approval. Children aged 4 to 11 years will only be randomized to the lower dosage level of MDI, 80/180 µg, or AS MDI (90 µg per actuation).

BDA MDI and AS MDI are IPs. The dose chosen for AS MDI (albuterol) is in line with the approved label for Proventil® with which AS MDI has been demonstrated to be equivalent in the D6930C00002 cumulative dose study and D6930C00001 dose finding study. Budesonide doses were assessed in the dose-ranging Study PT008001. The budesonide doses whosen for BDA MDI will allow assessment of the potential to provide therapeutic benefit in provide while avoiding excessive steroid dosing within the applicable age ranges.

#### 1.3 Benefit/risk and ethical assessment

BDA MDI may provide benefit in subjects in terms of potential reduction in the risk of asthma exacerbation and improvement in the control of asthma symptoms and lung function beyond what is typically seen with albuterol alone (Rabe 2006; Seyme 2005; O'Byrne 2007). In addition, the Sponsor believes that the administration of BDA MDI to subjects with asthma will achieve the rapid improvement in lung function from albuterol, the anti-inflammatory effect attributable to budesonide, and potentially additional benefits attributable to the combination of albuterol and budesonide.

The risk of adrenal suppression, particularly during a period of stress (infection, surgery, etc) has been noted in the Canadian product methograph for Pulmicort Turbuhaler<sup>®</sup>. The Sponsor considers it is relevant to monitor steroid effects in subjects. As such, routine tests of adrenal cortisol function have been built into this study to monitor for adrenal suppression risk: morning serum cortisol will be assessed.

Further, height (cm) measurements will be assessed more frequently in subjects ≤18 years of age, to monitor for any possible effects on growth.

#### COVID-19

Recent information from the American Academy of Allery Asthma and Immunology (AAAAI) published on their website (https://www.aaaai.org/conditions-and-treatments/library/asthma-library/co.ad-asthma) in indicates that currently there is no evidence of increased infection rates in patients with asthma and that best practice is to ensure that a patient's asthma is controlled. In the MANDALA study, subjects are maintained on a stable asthma treatment regimen and closely monitored while staying in the study. The sponsor believes that the benefit risk assessment for trial participants to enroll and continue in the study is positive.

#### 1.4 Study design

This is a randomized, double-blind, multicenter, parallel-group, variable-length, event-driven study with a treatment period of at least 24 weeks for each subject. The purpose of this study is to compare 2 doses of BDA MDI with AS MDI on the time to first severe asthma exacerbation (Section 5.1.1) in adult, adolescent, and pediatric subjects with moderate to severe asthma as defined by GINA. Subjects will administer randomized investigational product (IP) prince response to asthma symptoms. See Figure 1 for a graphical presentation of the study screen and Table 1 for a list of study assessments.

Subjects attending screening (Visit 1) will enter a 14- to 28-day screening and run-in period. The screening period may be extended to a maximum of 9 weeks for subjects who have a severe asthma exacerbation after Visit 1. Subjects may consent for the study in advance of Visit 1 and if required, request for medical records to support evidence of prior exacerbations without triggering the 28-day screening period. Screened subjects will continue to take their regular asthma maintenance therapy throughout the study (from screening Visit 1/1a, as applicable)) through the treatment period). At Visit 1, eligible subjects will discontinue their usual print inhaled product used for symptom relief and begin Sponsor provided Ventolin to be used print response to symptoms or prior to exercise during the creexing period only. Subjects will be asked to turn in their own inhaled reliever products to the investigational sites for storage until the individual subject last study visit. Eligible and jects will be randomized at Visit 2.

At randomization (Visit 2), adult and adolescent subjects (aged ≥12 years) who meet the eligibility criteria will be randomly assigned to 1 of the following 3 treatment groups in a 1:1:1 ratio as reliever therapy on top of usual case. Children aged 4 to 11 years will be randomized in a 1:1 ratio only to the lower BDA MDI desage or AS MDI:

- BDA MDI 80/180 μg (given as actuations of BDA MDI 40/90 μg per puff) prn
- BDA MDI 160/180 μg (given as 2 actuations of BDA MDI 80/90 μg per puff) prn
- AS MDI 180 μg (given 2 actuations of AS MDI 90 μg per puff) prn

The maximum daily dosage of IP should not exceed 12 puffs per day. Subjects will be recommended not to take more than 8 puffs per day and advised to contact the investigator if their symptoms necessitate more than 8 puffs in a day.

The maximum daily dosage is 12 puffs (BDA MDI 480/1080 µg or 960/1080 µg, or AS MDI 1080 µg). In order to ensure safety and monitor daily treatment status, all subjects will be provided with an electronic diary (eDiary: AM3 device). The eDiary transfers data every 24 hours across a range of asthma symptom scores and drug usage (ie, number of puffs inhaled) to assess a subject's asthma status. Subjects will use the eDiary for reporting daily use of IP and any symptoms. If symptoms and/or daily dosage exceed a protocol-specified threshold, the eDiary will generate an alert to the subject and the investigational site. In this way, daily IP

usage will be monitored closely by the investigators and medical monitors to assess any worsening of subject status. Action will be taken where clinically indicated.

The study will consist of 3 periods:

- Screening period (14 to 28 days) except where a severe exacerbation event occurs during the screening period, and this may be extended to a maximum of 9 weeks. (Subjects may consent for the study in advance of Visit 1 and if required, request for medical records to support evidence of prior exacerbations without triggering the 28-day screening period.)
- Treatment period of at least 24 weeks. The study treatment period will continue extension
  phase) until the required 570 first severe exacerbation events, as defined perprotocol, have
  been reached and the last adult subject has completed 24 weeks of treatment, which will be
  defined as the PCD. Not all pediatric subjects will have 24 weeks of treatment at time of
  PCD.

In the event 570 events will be captured before the last subject has had 24 weeks of treatment, all subjects on treatment for ≥24 weeks will have their end-of-study (EOS) visit at their next scheduled clinic visit. All subjects on treatment for <24 weeks will continue until 24 weeks at which point they will complete their EOS visit

In the event 570 events will be captured after the last subject has had 24 weeks of treatment, each subject will return to complete the EQS vision at their next scheduled clinic visit

Safety follow-up period: where a safety follow is telephone contact will occur 2 weeks
 (±4 days) after the subject's EOS visit or previous discontinuation visit (PDV), whichever
 occurs first

The study will be completed when the last subject has completed his/her post-study follow-up telephone contact. Subjects who discontinue IP will complete a PDV, and adverse events (AEs)/serious adverse events (SAEs) will be followed up if medically indicated.

Figure 1 Study design



ICS=inhaled corticosteroid; LABA=long-acting  $\beta Z$  agonit, N=number; PRN=as needed; R=randomization; SABA=short-acting β2-adrenoreceptor agonist somening visit; W=week.

#### 1.5 Study governance and

#### 1.5.1 Independent data Monitoring committee

An independent data monitoring committee (IDMC) will be established to assess the ongoing safety of the study. The IDNEC will review blinded data (open session) and unblinded safety data (closed session) to assess any safety related reasons why the study should continue, be modified, or stopped. Glosed sessions will be supported by the unblinded statistician and responsibilities of the IDMC will be clarified within a charter before initiation of the study.

The IDMC chair and all committee members will be independent investigators/specialists separate from the study team or contract research organization.

All decisions made by the IDMC will be documented within written records of meetings and recommendation made to the Sponsor.

#### 1.5.2 Adjudication committee

An independent adjudication committee will adjudicate centrally and in a blinded fashion after medical monitoring review, cases where a reported death, emergency room visit, urgent care visit and/or hospitalization, change in medication and/or other sign/symptom is indicative of worsening of asthma but has not been recorded as such in the electronic case report form, (eCRF). For any event that qualifies for adjudication, study sites will be asked to provide deidentified (anonymized) clinical documentation such as discharge summaries, to suggest the external event adjudication. The tasks and responsibilities of the adjudication committee will be filed in a charter before initiation of the study and will contain written operating procedures. The adjudication committee will maintain the adjudication results in writing and will enter details of events not recorded within the eCRF into an adjudicated platform. This data will be reported alongside the eCRF data in the Clinical Study Region.

#### 2 STUDY OBJECTIVES

#### 2.1 Primary objective

| Primary Objective: | Priparty exterpoint: |
|---|---|
| To evaluate the efficacy of budesonide/albuterol metered-dose inhaler 80/180 μg and 160/180 μg administered prn in response to symptoms compared to albuterol metered-dose inhaler 180 μg | Third toofirst severe asthma exacerbation |

#### 2.2

| <u> </u> | |
|---|---|
| 2.2 Secondary objective: Secondary endpoint: | |
| Secondary Objective: | Secondary endpoint: |
| To characterize the effect of bude bnide/albuterol metered-dose inhaler 80/180 kg and 160/180 µg administered prn in response to symptoms compared to albuterol metered-dose inhaler 180 µg | <ul> <li>Severe exacerbation rate (annualized)</li> <li>Total systemic corticosteroid exposure over the treatment period</li> <li>Asthma Control Questionnaire-5 (ACQ-5) change from baseline and responder analysis at Week 24</li> <li>Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12)/Pediatric Asthma Quality of Life Questionnaire (PAQLQ) change from baseline and responder analysis at Week 24</li> </ul> |

#### 2.3 Safety objective

| Safety Objective: | Safety Endpoints: |
|---|---|
| To evaluate the safety and tolerability of<br>budesonide/ albuterol metered-dose inhaler<br>80/180 µg and 160/180 µg administered prn in<br>response to symptoms compared to albuterol<br>metered-dose inhaler 180 µg | Adverse events/serious adverse events Vital signs Clinical chemistry and hematology parameters Electrocardiogram |

#### 2.4 Exploratory objective

| Zapiorator, objective | |
|---|---|
| Other Objective: | Exploratory Endpoints: |
| To characterize the effect of budesonide/albuterol<br>metered-dose inhaler 80/180 µg and 160/180 µg<br>administered prn in response to symptoms<br>compared to albuterol metered-dose inhaler 180<br>µg | <ul> <li>Asthma Control Question aire-5 change from baseline and responder analysis at Week 12</li> <li>Asthma Control Questionnaire-5 change from baseline and responder (3-factor) analysis at Week 12 and Beek 24</li> </ul> |
| ć. | <ul> <li>Asthma Control Questionnaire-3 change from baseline and responder analysis at Week 12</li> <li>Asthma Control Questionnaire-5 change from baseline and responder (3-factor) analysis at Week 12 and Seek 24</li> <li>Asthma Quality of Life Questionnaire for 12 years and older Pediatric Asthma Quality of Life Questionnaire change from baseline and responder analysis at Week 12</li> <li>Seteriorations of asthma (annualized rate and time to first)</li> <li>Change from baseline in prebronchodilator forced expiratory volume in 1 second at Week 12 and Week 24</li> <li>Morning and evening peak expiratory flow</li> <li>Use of investigational product (reliever therapy)</li> <li>Asthma daytime/night-time symptoms</li> <li>Time to treatment discontinuation or change in maintenance therapy</li> <li>Asthma Control Test (ACT) or Childhood Asthma Control Test (C ACT) change from baseline and responder analysis at Week 24</li> <li>Percentage of "as needed"-free days</li> <li>Percentage of symptom-free days</li> <li>Percentage of asthma control days</li> <li>Inhaled corticosteroid exposure over the treatment period</li> </ul> |
| at Pai | Change from baseline in prebronchodilator forced expiratory volume in 1 second at Week 12 and Week 24 |
| Milate | <ul> <li>Morning and evening peak expiratory flow</li> <li>Use of investigational product (reliever therapy)</li> <li>Asthma daytime/night-time symptoms</li> </ul> |
| Eros, | Time to treatment discontinuation or change in maintenance therapy |
| A to supp | Asthma Control Test (ACT) or Childhood Asthma Control Test (C ACT) change from baseline and responder analysis at Week 24 |
| ્રું<br>જે | Percentage of "as needed"-free days |
| | Percentage of symptom-free days |
| 200 | Percentage of asthma control days |
| nist ni | Inhaled corticosteroid exposure over the treatment<br>period |

#### 3 SUBJECT SELECTION, ENROLLMENT, RANDOMIZATION, RESTRICTIONS, TREATMENT DISCONTINUATION, AND STUDY TERMINATION

Each subject must meet all of the inclusion criteria and none of the exclusion criteria for this study. No waivers will be granted from the Sponsor for any subject not meeting inclusion exclusion criteria.

No study-related procedures may be performed before the subject has signed the thics Committee (EC) approved Informed Consent Form (ICF)/assent form.

#### 3.1 Inclusion criteria

For inclusion in the study, subjects must fulfill the following criteria within the screening period:

- Able and willing to provide written informed consent or sign age-appropriate forms, subjects below legal age of consent must have parent(sor guardian sign the ICF before participation
- Female or male aged ≥4 years at the time of participated consent in all countries with the exception of the following: in Serbia, only subjects ≥12 years old will be enrolled; in Germany, Slovakia, and Ukraine, only subjects ≥18 years old will be enrolled.
- 3 Diagnosis of asthma as defined by Criteria at least 1 year before Visit 1
- 4 Receiving 1 of the following schedules asthma maintenance therapies for 3 months with stable dosing for at least the last 4 weeks before Visit 1:
  - (a) Medium-to--high-dose ICS (Appendix C; GINA 2018)
  - (b) Medium-to-high-dose ICS and 1 additional maintenance therapy from the following: LTRA, LAMA, or the phylline
  - (c) Low-to-high-dose KS in combination with LABA with or without 1 additional maintenance thereby from the following: LTRA, LAMA, or theophylline
    - Up to 20% of all randomized subjects (on ICS alone or ICS in combination with LABA) will be permitted to have an additional maintenance medication (seephylline, leukotriene receptor antagonist, or LAMA).

The below defines the minimally acceptable documentation required to support inclusion criterion 4:

Signed and dated notes from a referring physician, including name, dose, and duration of the ICS or ICS/LABA inhaler (or names and doses, if used as separate inhalers) and LTRA, LAMA, or theophylline, if applicable, and/or

- Evidence of prescriptions for an ICS, ICS/LABA, and LTRA, LAMA, or theophylline if applicable, medications that demonstrate coverage for the duration specified in inclusion criteria
- Prebronchodilator forced expiratory volume in 1 second (FEV<sub>1</sub>) of ≥40 to <90% predicted normal value for adults, and >60% predicted normal value for subjects aged 4 to 17 years after withholding the medications specified in Table 4. If FEV<sub>1</sub> values are not within the permitted range at Visit 1, 1 re-test must be performed at Visit 1a before advancing to Visit 2 or confirming screen failure. Note: Subjects 4 to 17 years of age who previously failed inclusion criterion 5 due to the previous upper FEV1 limit will be permitted to rescreen once and will be required to meet all other eligibility criteria upon e-screening.
- Subjects aged ≥12 years of age must demonstrate reversibility at VisiQ, with an increase in FEV<sub>1</sub> ≥12% (and ≥200 mL for subjects aged ≥18 years) relative baseline after administration of Sponsor-provided Ventolin via central spirometry. If reversibility is not demonstrated at Visit 1, 1 re-test for reversibility testing must be done at Visit 1a before advancing to Visit 2 or confirming screen failure. Subjects@ged 4 to 11 years of age will perform the reversibility test, but do not require demonstration of reversibility during Visit 1 and may enroll provided documented historica reversibility within 1 year is available. Subjects aged 4 to 11 years who previously failed inclusion criterion 6 will be permitted to rescreen. Each subject may rescreen only once.
- Demonstrate acceptable spirometry performance (ie, meet American Thoracic Society/European Respiratory Society acceptability/repeatability criteria) (Appendix M, Spirometry Assessment Criteria), Subjects 4 to 11 years will be eligible if they provide 2 acceptable/repeatable measurements
- A documented history of at least severe asthma exacerbation within 12 months before Visit 1

For inclusion, a severe exacerbation is considered to be any deterioration of asthma that led to at least 1 of the following conditions:

- A temporary bolus/burst of SCS for at least 3 consecutive days; a single depoinjectable dose of corticosteroids will be considered equivalent to a 3-day course
- An in-patient hospitalization (definevaluation and treatment in asthma

  The below definestudy: An emergency room or urgent care visit (defined as evaluation and treatment for 624 hours in an emergency department or urgent care center) because of asthma

An in-patient hospitalization (defined as admission to an in-patient facility and/or evaluation and treatment in a healthcare facility for ≥24 hours) because of

The below defines what is acceptable to document exacerbations for inclusion in this

- Discharge summaries from a hospital, emergency room, or an urgent care facility indicating that a subject was hospitalized or treated with SCS for an asthma exacerbation
- Signed and dated notes from a referring physician, including information regarding diagnosis and treatment of an exacerbation with SCS
- Subjects can provide evidence of prescriptions for SCS used during an exacerbation
- Asthma Control Questionnaire-7 (ACQ-7) score ≥1.5 assessed at Visit 1
- 10 ACQ-5 score >1.5 assessed at Visit 2
- 11 Use of Sponsor-provided Ventolin prn medication because of asthma Symptoms on at least 3 days during the last week of the run-in period before Visit 2,0
- 12 Demonstrate acceptable MDI administration technique as assessed by the investigator; use of spacers prohibited
- 13 Able to perform acceptable and reproducible peak expiratory flow (PEF) measurements as assessed by the investigator
- 14 Body mass index <40 kg/m<sup>2</sup>
- 15 Willing to remain at the study site as required exprotocol and complete all visit assessments

  16 Negative pregnancy test (serum at Visit Y) for female subjects of childbearing potential
- 17 Women of childbearing potential and sexually active in heterosexual relationships must agree to 1 of the following options to prevent pregnancy:
  - (a) Practice complete abstinence desided as refraining from heterosexual intercourse during the entire period of ris@associated with the study treatments. Periodic abstinence is not acceptable. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Therefore complete abstinence is an acceptable method of contraception only if it is consistent with the preferred and usual lifestyle of the subject.
  - (b) If a female of childbearing potential agrees to prevent pregnancy by using 1 of the following methods of birth control from the date the ICF is signed until 2 weeks after the final dose of IP is taken:
    - Hormonal contraception (eg, oral contraceptive, contraceptive implant, or injectable hormonal contraceptive)
      - Double-barrier birth control (ie, a combination of male condom with either cap, diaphragm, or sponge with spermicide, a condom with spermicide, intrauterine device [IUD] and intrauterine hormone-releasing system [IUS])
    - Maintenance of a monogamous sexual relationship with a male partner who has been surgically sterilized by vasectomy provided that the male partner is the

sole sexual partner of the female (of childbearing potential) participant and that the vasectomized partner has received medical assessment of the surgical success (ie, documented history of medical confirmation of success of vasectomy).

Note: Women are considered to be of nonchildbearing potential if they are physiologically incapable of becoming pregnant, including any female who is 2 years postmenopausal (a postmenopausal state is defined as no menses for 12 months; without an alternative medical cause), or surgically sterile, defined as having a bilateral salpingectomy, bilateral oophorectomy, or hysterectomy. Tubal ligation with the considered an acceptable permanent birth control measure for this protocol. For purposes of this protocol, menopausal women are defined as women who are an enorrheic for 12 consecutive months or more after cessation of all exogenous hospital treatment. Adolescent specific recommendations: If subject is female and has reached menarche, or has reached Tanner stage 3 breast development (even if not having reached menarche), the subject will be considered a female of child bearing potential.

Contraceptive methods may be recommended for adolescent females only if they are already sexually active. Use of hormonal contraceptives in adolescent females must always be in consultation with a gynecologist.

Male subjects who are sexually active in better sexual relationships must be surgically sterile or agree to use a double-barrier method of contraception (ie, a combination of male condom with either cap, diaphragm or spronge with spermicide) from the first dose of randomized IP until 2 weeks after their last dose. Male subjects must not donate sperm during their study participation period.

#### 3.2 Exclusion criteria

Subjects must not enter the stady if any of the following exclusion criteria are fulfilled within the screening period:

- 1 Chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, entalitysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulationary dysplasia), including regular or occasional use of oxygen
- Oral/SCS use (any dose and any indication) within 6 weeks before Visit 1
  Subjects who have experienced an asthma exacerbation requiring oral/systemic glucocorticosteroid in the 6 weeks before Visit 1 cannot be enrolled in the study because of the 6 weeks wash out of the oral/SCS, but can enter Visit 1 once the wash out period has been met

Chronic use of oral corticosteroids (OCS, ≥3 weeks use in 3 months prior to Visit 1)

- 4 Having received any marketed (eg, omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab) or investigational biologic within 3 months or 5 half-lives before Visit 1, whichever is longer, or any other prohibited medication
- 5 Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months before Visit 1 (including all forms of tobacco, e-cigarettes) [vaping], and marijuana)</p>
- 6 Life-threatening asthma defined as any history of significant asthma episode(s) equiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, asthma-related syncopal episode(s) within 5 years of Visit 1
- 7 Completed treatment for lower respiratory infection or asthma exacerbation within 6 weeks of Visit 1
- 8 Upper respiratory infection involving antibiotic treatment not respect within 7 days before Visit 1
- 9 Clinically significant laboratory abnormalities, in the opinion of the investigator, or having any of the following results at Visit 1:
  - (a) a serum creatinine value >1.5 times the upper limit of the reference range
  - (b) a serum total bilirubin value >1.5 times the upper limit of the reference range
  - (c) a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2.5 times the upper limit of the reference range

Note: Laboratory tests may be repeated once: if laboratory tests have to be repeated, the results must be available for review before Visit 2 (randomization).

- 10 Having any of the following results at Visit 1:
  - (a) an abnormal electrocardiogram (ECG) that is, in the investigator's opinion, clinically significant
  - (b) a QTCF interval >480 fms (subjects aged ≥12 years)/ ≥460 ms (subjects aged 4 to 11 years, based on the Fridericia correction where QTCF=QT/RR0.33)
- Historical or currence vidence of a clinically significant disease including, but not limited to: cardiovascular (eg, congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia, coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine (eg, uncontrolled diabetes mellitus, uncontrolled thyroid disorder. Addison's disease, Cushing's syndrome), or gastrointestinal (eg, poorly controlled peptic ulcer, gastroesophageal reflux disease) disorders. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject which through study participation, or that could affect the efficacy or safety analysis if the disease/condition exacerbated during the study

Cancer not in complete remission for at least 5 years before Visit 1

History of psychiatric disease, intellectual deficiency, poor motivation, or other conditions if their magnitude is limiting informed consent validity.

Significant abuse of alcohol or drugs in the cancer are eligible, if in the opinion cancer are eligible, if in the opinion cancer are eligible, if in the opinion and the subject's concern.

Hospitalization for psychiatric disorder or attempted suicide within 1 year of Visit 18 subject of Visi

- 16 Having a known or suspected hypersensitivity to albuterol/salbutamol, obbudesonide and/or their excipients

  17 Having a scheduled/planned hespitalization during the study.
- 17 Having a scheduled/planned hospitalization during the study
- 18 Inability to abstain from protocol-defined prohibited medications during the study
- 19 Using any herbal products by inhalation or nebulizer within weeks of Visit 1 and not agreeing to stop during the study duration
- 20 Having received a live attenuated vaccination within Mays of Visit 1.
- Currently pregnant or breastfeeding
   Study investigators, subinvestigators, coordinators, and their employees or immediate family members, or employees of the Sponsor
- 23 Treatment with any investigational treatment or device in another clinical study within the last 30 days (or 5 half-lives, which were longer) of Visit 1
- 24 Currently participating in any interventional study
- 25 Having previously been randomized in this study or any other PT007 or PT027 clinical
- 26 Subjects who experience stathma exacerbation during the screening period

Procedures for withdraw of incorrectly enrolled subjects are described in Section 3.4.

#### Subjectenrollment and randomization

Approximately 3500 adult and adolescent subjects with moderate to severe asthma will be randomized to 1 of 3 treatment groups (approximately 1000 subjects per group). In addition, up to 100 subjects in the 4 to 11-year age group with moderate to severe asthma will be randomized with approximately 50 subjects randomized to the AS MDI and 50 subjects randomized to the low dose BDA MDI groups only. Approximately 6000 subjects will need to be creened, assuming an estimated screen failure rate of 30% to 50%. This Phase III study is manned to be conducted globally.

The investigator(s) and/or study personnel will:

- Obtain signed informed consent/assent (as applicable) from the potential subject and/or their guardian/legal representative before any study specific procedures are performed
- 2 Enter the subject data into the enrollment module in Rave Web Based Data Capture (WBDC) eCRF to enable the allocation of subject identification (Ecode)
- 3 Determine subject eligibility (see Sections 3.1 and 3.2)
- 4 Enter the information required to enable the Interactive Web Response System (IWRS) to initiate randomization and generate the randomization code

Randomization codes will be assigned through IWRS strictly sequentially to subjects eligible for randomization. If a subject withdraws from participation in the study, then his/her randomization code cannot be reused.

### 3.4 Procedures for handling incorrectly enrolled or andomized subjects

Subjects who fail to meet the eligibility criteria should not, under any circumstances, be randomized or receive IP. There can be no waivers granted from the Sponsor for any subject not meeting inclusion or exclusion criteria. Subjects who are enrolled, but subsequently found not to meet all the eligibility criteria must not be randomized or initiated on treatment, and must be screen-failed and withdrawn from the study.

Where a subject does not meet all the eligibility enteria but is randomized in error, or incorrectly started on treatment, the investigator should inform the medical monitor assigned to the project immediately, and a discussion should occur between the medical monitor assigned to the project and the investigator regarding whether to continue or discontinue the subject from treatment. The Sponsor's medical monitor assigned to the project must ensure all decisions and protocol deviations, any, are appropriately documented.

#### 3.5 Methods for a signing treatment groups

A randomization schedule will be generated by a designated statistical representative performing statistical support for the study. This schedule will be prepared before the start of the treatment period of the designated statistical representative will follow their established standard operating procedures regarding generation, security, and distribution of the randomization schedule.

Randomization will be centralized. Adult and adolescent subjects (aged ≥12 years) will be randomized in a 1:1:1 ratio into 1 of the 3 treatment groups as reliever therapy on top of usual care (BDA MDI 80/180 μg, or BDA MDI 160/180 μg, or AS MDI 180 μg) according to a SACS-generated randomization schedule. Children aged 4 to 11 years will be randomized in a 1:1 ratio only to the lower BDA MDI dosage (80/180 μg) or AS MDI 180 μg. Randomization for adolescents and adults will be stratified by age group (≥12 to 17, ≥18); region (North

America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to screening (Visit 1) plus any severe exacerbation event experienced during the screening period. Randomization for children will not be stratified.

Upon enrollment, subjects will be assigned a unique subject identification code (Ecode) which is automatically generated by the electronic data capture system (Rave WBDC) based on the order of entry. Once it has been determined that a subject meets all eligibility criteria, the subject information will be integrated into the IWRS (Randomization and Trial Supply Management) for randomization.

#### 3.6 Methods for ensuring blinding

The study blind is to be maintained until all subjects have completed the treatment period and until after the database has been locked. The study site receives documentation of subject study identification and kit allocation through the IWRS. The randomization code will not be available, with the exception of unblinding procedures described in Section 3.7, to the study team, study center personnel, Sponsor monitors, Sponsor project statisticians, or any other personnel employed or affiliated with the Sponsor as well as investigators and subjects until after the database has been locked.

The 3 different kit types of study IP are visually identical, protecting the blind through their similarity in appearance.

#### 3.7 Methods for unblinding

The treatment blind should not be broken except in medical emergencies and based on the investigator's clinical judgment when the appropriate management and welfare of the subject requires knowledge of the treatment allocation. Individual treatment details, for each subject, will be available to the investigator(s) or pharmacists from the IWRS, if needed. If unblinding occurs, the investigator must notify the Sponsor as soon as possible, but without revealing the treatment assignment of the unblinded subject. Routines for this will be described in the IWRS user manual that will be provided to each center. The IWRS provides unblinding procedures, if needed.

The designated representative retains the right to break the code for SAEs that are unexpected and are suspected to be causally related to an IP and that potentially require expedited reporting to regulatory authorities. Treatment codes will not be broken for the planned analyses of data until all decisions on the evaluability of the data from each individual subject have been made and documented.

With the exception of emergency unblinding as described above, all members of the study team, investigators, and site staff will be blinded. The only individuals who will have access

to unblinded information during the conduct of the study in advance of the primary outcome database lock will be the unblinded statistician supporting the IDMC closed session review which will be performed in accordance with the IDMC charter.

#### 3.8

Restrictions

Subjects should be advised that marketed (eg, omalizumab, mepolizumab, reslizumab benralizumab, dupilumab) or investigational biologic treatments or other investigational treatments other than the IPs are not allowed during the treatment power.

Subjects requiring chronic OCS are excluded. All and locumented at baseline, should recognize the pinion, if a subopinion, if a subject requires a change in their asthma maintenance therago, this should be discussed with the medical monitor.

Changes to maintenance therapy doses would be permissible in specific circumstances and when clinically indicated. In the event that the investigator considers the introduction of additional maintenance therapy or intensification of the existing maintenance therapy (change) is required, the medical monitors should be contacted.

#### Treatment discontinuation by Subject and/or Sponsor 3.9

Subjects may be withdrawn from the study at any sime at their own request, upon request of the investigator, or by the Sponsor at any time of for any reason. The subject or his/her parent/legal representative is free to discontinue treatment at any time, without prejudice to further treatment. Other reasons for discontinuation may include:

- Adverse event
- Subjects who suffer ≥3 severe exacerbations within a 3-month period or ≥5 total severe exacerbation events, or a single severe exacerbation event longer than 20 days in duration should be considered for discontinuation if Sponsor and the investigator decide that it is in the best interest of the subject to discontinue randomized treatment and withdraw from the study (an exace bation alone does not require subject discontinuation)
- In the opinion of the investigator, the subject is noncompliant with the Clinical Study Protocol (eggost-enrollment eligibility violation) or is lost to follow-up and no alternative contact information is available (this implies that at least 2 documented attempts have been made to contact the subject)
- If famale subject becomes pregnant, the subject will automatically be discontinued from
- In subjects who have elevated liver enzymes AST and/or ALT  $\geq$ 3 times the upper limit of normal (×ULN) and total bilirubin (TBL) ≥2×ULN (ie, meeting the criteria of at least Potential Hy's Law), IP will be suspended until the liver test values return to the normal

range. If the AST, ALT, or TBL reach these elevated levels again, after recommencement of IP, the subject will be discontinued from IP and withdrawn from the study.

The study will be completed when the last subject has completed his/ or her post- study follow-up telephone contact. Subjects who discontinue IP will complete a PDV, and AEs/SAEs will be followed up if medically indicated.

A subject that decides to discontinue IP will always be asked about the reason(s) and the presence of any AEs. If possible, they will be seen and assessed by an investigator(s). Adverse events and SAEs will be followed up (See Section 6); eDiary and all IPs should be returned by the subject.

Subjects who discontinue study treatment prior to EOS will be encouraged to remain in the study to complete all remaining study visits during the treatment/extension phase period. Treatment discontinuation subjects will return to appropriate maintenance asthma medications, per the investigator's discretion. For subjects recorded as Treatment Discontinuations who do not complete at least 1 post-treatment data collection, a telephone follow-up call is required at least 14 days after last 12 days.

If a subject chooses not to continue with study assessments, at a minimum the subject will complete the PDV (as indicated in Table 1). These subjects will return to appropriate maintenance medications, per the investigators discretion. A follow-up telephone call (TC) will be performed at least 14 days after the last IP dose. In the event the PDV is performed >14 days post last IP dosing, a follow-up PC will not be required. These subjects who do not withdraw consent for follow-up will be followed for survival/death, severe exacerbations, AEs/SAEs, and concomitant medications including asthma treatment (maintenance and rescue therapies) at quarterly intervals until EOS.

#### 3.10 Study termination

If the Sponsor, investigator, study monitor, IDMC, or regulatory officials discover conditions arising during the study that indicate that the subject's safety and/or scientific value of the study and/or quality of the IPs have been compromised, the study may be halted or the study center's participation may be terminated. Ongoing subjects will be discontinued from the study and assigned to receive treatment as per local standard of care.

Conditions that may warrant termination of the study include, but are not limited to, the following list:

The study may be stopped if, in the judgment of the Sponsor, study subjects are placed at undue risk because of clinically significant findings that:

are considered significant
- are assessed as causally related to IP
- are not considered to be consistent with continuation of the study
- The discovery of an unexpected, serious, or unacceptable risk to the subjects enrolled in
- A decision on the part of the Sponsor to suspend or discontinue testing, evaluation, development of the IP for any reason

Conditions that may warrant termination of a study center's participation include, but are not limited to, the following list:

- Failure of the investigator to enroll subjects into the study at an acceptable rate or within an agreed timeline
- Failure of the investigator to comply with pertinent governing both regulations
- Submission of knowingly false information from the research facility to the Sponsor, study monitor, medical officer, or regulatory official
- Insufficient adherence to protocol requirements

Regardless of the reason for termination, all data available for the subject at the time of discontinuation of follow-up must be recorded in the eCRF. All reasons for discontinuation of treatment must be documented.

essure that adequate consideration is given to the In terminating the study, the Sponsor protection of the subjects' interests.

Study termination and follow-up will be performed in compliance with applicable governing body regulations.

## Screen failures 3.11

Screening failures are subjects who do not fulfill the eligibility criteria for the study, and therefore must not be andomized. These subjects should have the reason for study withdrawal recorded as "Screen failure". Subjects who screen fail will not be rescreened except for children and adolescents who screen failed because they did not meet the now obsolete upper FEV<sub>1</sub> % predicted limit. Children and adolescents who previously failed to meet the upper FEV<sub>1</sub> % predicted threshold, but who met all other eligibility requirements, may re-screen once. Upon re-screening, these subjects must meet all eligibility requirements in order to be

, will be purpose the state of

Table 1 Study Assessments and Procedures

| Z 2 0 4 1 X X X X X UITING | 3<br>4<br>28±2<br>X | AL ST | 5 | 6° | 7<br>36<br>252 ±4<br>00<br>X | Extension Phase (every 124) weeks ±8days until the PCD) X | X<br>X<br>X<br>X <sup>f</sup><br>X | PDV c (if applicable) X Xf X | Safety Follow-up IC (2 weeks [±4 days]after EOS o PDV) |
|---|---|---|---|---|---|---|---|---|---|
| 2<br>0<br>4<br>1<br>X | 4<br>28 ±2 | 8<br>56±2 | 12 | 24 | 36 | (every 12+<br>weeks ±4 days<br>until the PCD) | visit) X X <sup>f</sup> | X<br>X | (2 weeks [±4<br>days]after EOS o<br>PDV) |
| 0<br>4<br>1<br>X | 4<br>28 ±2 | 8<br>56±2 | 12 | 24 | 36 | weeks ±&days<br>until the PCD) | X<br>X <sup>f</sup> | X<br>Xf | days]after EOS o<br>PDV) |
| 0<br>4<br>1<br>X | 4<br>28 ±2 | 56±2 | | | | weeks ±&days<br>until the PCD) | X f | X <sup>f</sup> | PDV) |
| 4 1<br>X | 28 ±2 | 56±2 | | | | until (to PCD) | X f | X <sup>f</sup> | X |
| 4 1<br>X | 28 ±2 | 56±2 | | | | x<br>x | X f | X <sup>f</sup> | X |
| x | x | all do | A CONTRACTOR | Xf X | x x | x | X f | X <sup>f</sup> | X |
| x | x | all de | ED Sir | X <sup>f</sup> X | x x | x<br>x | X f | X <sup>f</sup> | X |
| | x | att of | ED air | X <sup>f</sup><br>X | x | x<br>x | X f | X <sup>f</sup> | х |
| | x | all of | Strong Raise | X <sup>f</sup><br>X | x | x<br>x | X f | X <sup>f</sup> | x |
| | x | ALL SO | Strox Strox | Xf<br>X | x | x<br>x | X f | X <sup>f</sup> | x |
| | x | ALIN S | inortair | X <sup>f</sup><br>X | x | x<br>x | X f | X <sup>f</sup> | x |
| | x | ALI OF | in X | X <sup>f</sup><br>X | X | x | | | x |
| | Х | OFFIGE STATE | jtr <sup>O</sup> X | X | X | x | x | x | x |
| T x | | Ser 9 | , | | | | | | |
| х | | , dill | | | | | | | |
| X | | ~ | | | | | | | |
| | X C | Ø X | X | X | X | X | X | X | |
| X | E. F. | | | X | | | X | X | |
| X | ok x | X | X | X | X | X | X | X | X |
| uring | urine h | urine h | urine h | serum | urine h | urine <sup>h</sup> | serum | serum | |
| No. | | | | X | | | X | X | |
| gP | | | | | | | | Ļ | |
| | | | | X | | | X | X | |
| | | | - | X | | | x | X | |
| | | | | | | | | | X X X X 39 of 159 |

| | Screening<br>and run-<br>in | | Double | e-blind T | reatment | Period | | Extension<br>Phase | EOSO (last clinic | PDV e<br>(if<br>applicable) | Safety Follow-up<br>TC<br>(2 weeks [±4 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit a | 1/1a b | 2 | 3 | 4 | 5 | 6° | 7 | (every 12- | Prisit) | аррисавте) | days]after EOS or |
| | | | | | | | | weeks ±4 day | | | PDV) |
| Week | -4 to -2 | 0 | 4 | 8 | 12 | 24 | 36 | until the P (50) | | | |
| Day | -28 to -14 | 1 | 28 ±2 | 56 ±2 | 84 ±4 | 168 ±4 | 252 ±4 | 3 | | | |
| Efficacy measurements :6 | | | | | | | | | | | |
| Collection/review of exacerbations i | X | X | X | X | X | X | X | 70 X | X | X | |
| ACQ-5 j | | X | X | X | X | X | ΧQ | x | X | X | |
| ACQ-7 k | X | | | | | | ×0. | | | | |
| ACT/C ACT | | X | X | X | X | , x,o | X | X | X | X | |
| AQLQ+12/PAQLQ | | X | X | X | x | 1 Sollie | X | X | X | X | |
| Review of PEF, use of IP (reliever therapy), asthma daytime/night-time symptoms, night-time awakenings due to asthma symptoms <sup>1</sup> | X | X | X | x<br>.c | A STAN | ₹ <sub>ØX</sub> | X | х | X | Х | |
| Spirometry (FEV1) <sup>m</sup> | x | X | | SOF | <b>₹</b> CX | X | | | | | |
| eDiary | d | | | 4,0 | , | | | | с | С | |
| Review compliance with eDiary | | X | X | JOHN TO SERVICE SERVIC | X | X | $\mathbf{x}$ | X | X | X | |
| Collection/review of exacerbations i X X X X X X X X X X X X X X X X X X | | | | | | | | | | | |
| Randomization | | X | 470 | | | | | | | | |
| IP (dispense/collect) | | d | or old | c/d | c/d | c/d | c/d | c/d | С | с | |
| Ventolin (dispense) | d | <sub>E</sub> NO | * | | | | | | | | |

Abbreviations: ACQ-5/7=Asthma Control Questionnaire for 12 years and older; β-hCG=β-human chorionic gonadotropin; BM body mass index; c=collect; C ACT=Childhood Asthma Control Test; d=dispense; ECG=electrocardiogram; EOS=end-of-study; FEX = forced expiratory volume in 1 second; IP=investigational product; LABA=long-acting β2-agonist; PAQLQ=Pediatric Asthma Quality of Life Questionnaire; PCD=primary completion date; PDV=premature discontinuation visit; PEF=peak expiratory flow; TC=telephone call; V=visit TC=telephone call; V=visit

a Repeat assessments/visits, if needed will be captured in unscheduled visits.

 40 of

- Visit 1 will be split and used for repeated assessments, if needed (ie, Visit 1a will be needed for the repeat assessment of abouterol/salbutamol reversibility test and FEV<sub>1</sub>, if applicable). Subjects may consent for the study in advance of Visit 1 and if required, request for medical periods to support evidence of prior asthma exacerbations without triggering the 28-day screening period. Where a severe exacerbation event occurs during the screening period, this may be extended to a maximum of 9 weeks (to account for a course of systemic corticosteroids of up to 1 week duration followed by a 4-week washout period). In the event of an extension to the screening period due to a severe exacerbation event, the following will be repeated: safety laboratory assessments, ECG, vital signs, concomitant medications, and medical/surgical history.
- The treatment duration for the study will be at least 24 weeks for each subject to support the subject exposure data. The study treatment period will continue (extension phase) until the required 570 first severe exacerbation events, as defined per protocol, have been eached; and the last adult subject has completed 24 weeks of treatment, which will be defined as the PCD. After Visit 6, visits will be scheduled every 12 weeks with the assessments from Visit 7 to be performed in all of them.
- The EOS visit will be planned once the first 570 severe exacerbation events occur. If a subject 8 treatment lasts ≥24 weeks then the subject's EOS visit will occur at their next scheduled clinic visit. Once the PCD has been reached, any ongoing subject will return to complete an EOS visit at their next scheduled clinic visit.
- Subjects who prematurely withdraw from the study will undergo a PDV. In the event he PDV is performed >14 days post last IP dosing, a follow-up TC will not be required. These subjects who do not withdraw consent for follow-up will be believed for survival/death, severe exacerbations, AEs/SAEs, and concomitant medications including asthma treatment (maintenance and rescue paragres) at quarterly intervals until EOS.
- Additional height (cm) assessments to be collected for subjects \le 18 years of age ONLY. Assessments of height will continue in accordance with a subject's age at the time of signed informed consent/assent (where a subject changes age outing the study).
- Demonstrate reversibility at Visit 1, with an increase in FEV<sub>1</sub> $\ge$ 12% (and  $\ge$ 200 mL for subjects  $\ge$ 18 years) relative to baseline after administration of Sponsor-provided Ventolin via central spirometry at either Visit 1 or Visit 1 or Visit 1 or Visit 1 or Visit 1 a must be used for re-testing, if needed; with only 1 reversibility re-test permitted an advance of randomization (Visit 2).
- h A serum pregnancy test (β-hCG) will be performed at Visit 1, and EOS/PDV; urine β-hCG test will be performed at all other clinic visits (for women of childbearing potential only). (In Argentina, women of childbearing potential will have additional pregnancy testing at monthly time points.)
- Asthma exacerbations data will be reviewed, and severe exacerbations identified as per Section 5.1.1. Subjects are to be reminded not to take any albuterol product except for the IP.
- Asthma Control Questionnaire-5 self-administered adult version to be used for adults and adolescents 11 years and older; the interviewer-administered version should be used for children 4 to 10 years. Subject will need to satisfy ACQ-5 (≥1.5) entry requirements at Visit 2.
- Subject will need to satisfy ACQ-7 (≥1.5) enty requirements at Visit 1.
- The AM3 device will be dispensed at screening and PEF measurements will be taken through the screening period in advance of Visit 2.

Prebronchodilator FEV1 will be measured in the morning between 06:00 and 11:00 AM at Visits 1, 2, 5, and 6. Prebronchodilator FEV1 of ≥40 to <90% predicted normal value for adults and ≥60% predicted normal value for subjects aged 4 to 17 years after withholding SABA thours (and at Visit 1 and Visit 1a [used for repeated assessments, if needed], if applicable, as confirmed by centralized spirometry). Sponsor-provided Ventolin should be withheld ≥6 hours at Visit 2 At subsequent treatment visits, IP should be withheld ≥6 hours before Visit 5 and Visit 6. At all visits where Eevi is measured (Visits, 1, 2, 5, and 0), subjects whose maintenance therapy includes LABA should be instructed not to use their maintenance therapy without the timeframe specified in Table 4 in advance of the visit as these are considered bronchodilators. If these medications were taken within the restricted time periods, visits should be re-scheduled.

The period of the visit as these are considered bronchodilators. If these medications were taken within the restricted time periods, visits should be re-scheduled. The period of the visit as these are considered bronchodilators. If these medications were taken within the restricted time periods, visits should be re-scheduled. The period of the visit as these are considered bronchodilators. If these medications were taken within the restricted time periods, visits should be re-scheduled. The period of the visit as these are considered bronchodilators. If these medications were taken within the restricted time periods, visits should be re-scheduled. Visit 2. At subsequent treatment visits, IP should be withheld ≥6 hours before Visit 5 and Visit 6. At all visits where FEV₁ is measured (Visits, 1, 2, 5, and 6), subjects whose maintenance therapy includes LABA should be instructed not to use their maintenance therapy with the timeframe specified in Table 4 in

## 4.1 Screening and run-in period

Procedures will be performed according to study assessments and procedures presented in Table 1. Subjects may consent for the study in advance of Visit 1 and if required, request for medical records to support evidence of prior exacerbations without triggering the 28-day screening period. The screening period will be 14 to 28 days except where a severe asthmatex exacerbation event occurs during this period. Where a severe asthmatex exacerbation occurs during the screening period, the period may be extended to a maximum of 9 weeks (to account for a course of SCS of up to 1 week in duration followed by a 4-week washout period). In the event of an extension to the screening period due to a severe exacerbation event, the following assessments and procedures will be repeated following washout of SCS before Visit 2: safety laboratory assessments, ECG, vital signs, concomitant medications, and medical/surgical history.

At screening, consenting subjects are assessed to ensure that they need eligibility criteria at Visit 1 or Visit 1a, as applicable. Subjects who do not meet these criteria must not be enrolled in the study.

The study procedures carried out during this period will pictude medical and surgical history, demographics, physical examination (including body mass index [BMI], weight and height), concomitant medications review, Sponsor-provided ventolin reversibility test (reversibility must be demonstrated at either Visit 1 or Visit 1a Wisit 1a will be used for re-testing, if needed; with only 1 reversibility re-test permitted in advance of randomization [Visit 2]), vital signs, 12-lead ECG, AEs, pregnancy test, blood samples for hematology and clinical chemistry (1 re-test is permitted in advance of Visit 3); and morning serum cortisol assessment, collection/review of exacerbations, spinemetry (if needed, FEV<sub>1</sub>, must be re-tested once at Visit 1a; only 1 re-test is permitted) ACQ-7, PEF, and dispensing eDiary.

Subjects aged 4 to 11 years of see who previously failed inclusion criterion 6 will be permitted to rescreen.

Demographic data and wher characteristics will be recorded and will include the age and year of birth; gender, race, and/or ethnicity according to local regulations; alcohol consumption; and smoking history.

A standard medical, medication, and surgical history will be obtained with review of the selection coloria for the subject. Previous asthma related treatments and duration of asthma related treatments will be recorded.

## Randomization/treatment period/extension phase

Procedures will be performed according to study assessments and procedures presented in Table 1.

Subjects should not administer Sponsor-provided Ventolin on the morning of their randomization visit (Visit 2). Subjects taking ICS, LABA, or other maintenance medications that can impact the performance of spirometry should refer to Table 4 for medications that can interfere with pulmonary function tests (PFTs).

At randomization (Visit 2), eligible subjects will enter a 24-week double-blind treatment period.

The study treatment period will continue (extension phase) until the required 570 first severe exacerbation events, as defined per protocol, have been reached and the last adult sobject has completed 24 weeks of treatment, which will be defined as the PCD.

- In the event 570 events will be captured before the last adult subject has had 24 weeks of treatment, all subjects on treatment for ≥24 weeks will have their EQS visit at their next scheduled clinic visit. All subjects on treatment for < 24 weeks will continue until 24 weeks at which point they will complete their EOS visit.</li>
- In the event 570 events will be captured after the adult last subject has had 24 weeks of treatment, each subject will return to complete the EOS visit at their next scheduled clinic visit.
- Children and adolescents ongoing in treatment after the PCD will continue in follow-up until they have completed 24 weeks of treatment.

The study procedures carried out during this period will include: randomization, concomitant medications review, height (for subjects 218 tears of age at time of informed consent), vital signs, 12-lead ECG, AEs, pregnancy test, thood samples for hematology, and clinical chemistry; and morning serum cortisol assessment, collection/review of exacerbations, spirometry, ACQ-5, asthma control test (ACT)/childhood esthma control test(C ACT), Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12)/Pediatric Asthma Quality of Life Questionnaire (PAQLQ) (where populations are approved), PEF, use of IP (reliever therapy), asthma daytime/night-time symptoms, night-time awakenings due to asthma symptoms, eDiary/IP compliance, and dispensing and/or collection of IP.

## 4.3 End-of-ctudy visit

Procedures will be performed according to study assessments and procedures presented in Table 1. The EoS visit will be planned once the 570 first severe exacerbation events occur. If a subject's treatment is ≥24 weeks then the subject's EOS visit will occur at their next scheduled clinic visit. Once the PCD has been reached, any ongoing subject will return to complete their EOS visit at their next scheduled clinic visit.

The study procedures carried out during this visit will include: physical examination (including weight), concomitant medications review, height (for subjects ≤18 years of age at time of informed consent), vital signs, 12-lead ECG, AEs, pregnancy test, blood samples for

hematology, and clinical chemistry, and morning serum cortisol assessment, review of asthma exacerbations, ACQ-5, ACT/C ACT, AQLQ+12/PAQLQ, review of PEF, use of IP (reliever therapy), asthma daytime/night-time symptoms, night-time awakenings due to asthma symptoms, eDiary/IP compliance, and collection and final reconciliation of the IP.

#### 4.4 Unscheduled visit and premature discontinuation visit

Repeat assessments/visits, if needed, will be captured in unscheduled visits and the procedures carried out during an unscheduled visit will be decided by the investigator.

Procedures will be performed according to study assessments and procedures presented in Table 1.

The study procedures carried out during the PDV visit will include: physical examination (including weight), height (for subjects ≤18 years of age), concomitant medications review, vital signs, 12-lead ECG, AEs, pregnancy test, blood samples for hematology, and clinical chemistry; and morning serum cortisol assessment, review of asthma exacerbations, ACQ-5, ACT/C ACT, AQLQ+12/PAQLQ, review of PEF, use of IP (reliever theraps), asthma daytime/night-time symptoms, night-time awakenings due to asthma symptoms, eDiary compliance, randomization, and collection and reconciliation of the IP.

#### 4.5 Safety follow-up period

tue assessments and procedures presented in Procedures will be performed according to Table 1. The safety follow-up telephoxic connect will occur 2 weeks (±4 days) after EOS or PDV, whichever occurs first.

The study procedures carried out during this period will include: recording of concomitant medications and AEs.

## 4.6

If a subject chooses not to continue with study assessments, at a minimum the subject will complete the PDV (as fadicated in Table 1). These subjects will return to appropriate maintenance medications, per the investigators discretion. A follow-up TC will be performed at least 14 days after the last IP dose.

In the event the PDV is performed >14 days post last IP dosing, a follow-up TC will not be required. These subjects who do not withdraw consent for follow-up will be followed for survivableath, severe exacerbations, AEs/SAEs, concomitant medications including asthma treatment (maintenance and rescue therapies) at quarterly intervals until EOS.

used for data collection and query handling. The investigator will ensure that data are recorded on the eCRF and in accordance with the instructions provided.

The investigator ensures the accuracy, completeness, and timeliness of the data recorded and of the provision of answers to data queries according to the Clinical Trial Agreement. The investigator will sign the completed eCRF. A copy of the completed eCRF will be archived at the study site.

The laboratory safety assessments will be sent for analysis to a central laboratory.

The spirometry and ECG assessments will be performed at site using MosterScope equipment provided by eResearch Technology including an AM3 device which will also be used to collect ACQ-5, ACQ-7, PEF, and eDiary data. In addition to this, a tablet will be used to collect the AQLQ+12 and ACT/C ACT questionnaire data using the Study Works software. This data will be recorded in the vendor's central database and transferred conciled with the eCRF data as summarized in Section 9.4.

#### 5.1 Efficacy assessments

Efficacy assessments include asthma exacerbations, AQLQ+12/PAQLQ, ACQ-5, ACT/C ACT, PEF, use of IP (reliever therapy), asthma vaytime/night-time symptoms, night-time awakenings due to asthma symptoms, and review Kel ary compliance.

### Asthma exacerbation definition 5.1.1

An asthma exacerbation is defined to deterioration of asthma which includes:

- Worsening of asthma signs/symptoms (see Section 5.1.1.1)
- Increased use of "as needed" reliever therapy
- Deterioration of lung function (ie, decreased PEF and/or decreased FEV<sub>1</sub>)
- A medical intervention as described below (see Section 5.1.1.3)

These descriptions above are provided for definition, however, only severe asthma exacerbation will be assessed during this study (Section 5.1.1.3).

## Definition of asthma signs/symptoms worsening

The worsening/onset of symptoms must include at least 1 of the following:

Shortness of breath

Wheezing

Clinical Study Protocol, Version 4.0 Budesonide/albuterol (BDA) – AV003

- Chest tightness
- Cough
- Sputum
- Night-time awakening due to asthma
- Activity limitation due to asthma
- Decreased PEF
- Decreased FEV<sub>1</sub>

## 5.1.1.2 Investigator-justified asthma exacerbations

A vast majority of asthma exacerbations are associated with worsening of the signs/symptoms described in Section 5.1.1.1. Clinical presentations may, however, vary among subjects. If a subject's symptoms and the overall clinical findings support the diagnosis of an asthma exacerbation, but the symptomatic worsening does not meet the definition in Section 5.1.1.1, the investigator must justify the decision for defining the event as an exacerbation and document the reasoning in the eCRF.

### 5.1.1.3 Severe asthma exacerbations

All protocol-defined severe asthma exacerbations need to fulfill the symptom criteria as defined in Section 5.1.1.1 and be supported by an eDiary alest or an investigator justification.

An asthma exacerbation will be considered severe if it results in at least 1 of the following:

- A temporary bolus/burst of SCS for at least 3 consecutive days to treat symptoms of asthma
  worsening; a single depo-injectable considered equivalent to
  a 3-day bolus/burst of SCS
- An emergency room or urgent care visit (defined as evaluation and treatment for <24 hours in an emergency department or urgent care center) due to asthma that required SCS (as per the above)
- An in-patient hospitalisation (defined as admission to an in-patient facility and/or evaluation and treatment in a healthcare facility for ≥24 hours) due to asthma

Note: all deaths will be adjudicated to determine if they meet the criteria for severe exacerbation events.

## 5.1.1.4 Treatment for severe asthma exacerbations

The treatment for a severe asthma exacerbation is at least 3 consecutive days of SCS.

• The recommended treatment (GINA 2018) for a severe exacerbation is prednisolone (1 mg/kg/day up to 50 mg for adults and adolescents) once per day (preferably in the morning) for 5 to 7 days

exension of such application Tapering the prednisolone dose is not needed if the treatment has been given for less than 2 weeks (GINA 2018)

Treatment for less than 3 days does not constitute a severe asthma exacerbation.

#### 5.1.1.5 Onset and duration of asthma exacerbations

For severe exacerbations, the duration is defined by the prescribed treatment.

For severe exacerbations:

- The start date will be defined as the start date of prescribed treatment with a SCS.
- The stop date will be defined as the last day of prescribed treatment with a SCS.
- If the timeframe between successive SCS use is  $\geq 7$  days, the event of severe asthma exacerbation will be considered as 2 separate events of severe sthma exacerbation. An event of severe asthma exacerbation is considered "singular" if SCS use is <7 days.
- A single depot injectable dose of corticosteroids will be considered equivalent to a 3-day course of SCS. The corresponding stop date for this treatment will consequently be determined as the date of administration plus Odays
- If multiple treatments are prescribed for the same exacerbation, the earliest start date and the latest stop date will be used.
- For a severe asthma exacerbation requiring hospitalization with no documented corticosteroid treatment, hospitalization admission/discharge dates, or emergency visit date will be used as start/stop dates.

#### Approach for capturing sthma exacerbations 5.1.1.6

#### 5.1.1.6.1 Severe Asthma Exacecontion eCRF

All screening and post-random attion severe asthma exacerbations (including investigatorjustified asthma exacerbations) must be captured using the Severe Asthma Exacerbation eCRF.

Severe asthma exacerbations will be considered expected study endpoints and will not be reported as AEs unless they also meet the criteria for an SAE (Section 6.3.5).

#### Symptom Reporting 5.1.1.6.2

The subject will use the eDiary for daily symptom reporting, entering symptoms twice daily.

If symptoms meet the below threshold, the eDiary generates an alert to the subject and the investigational site:

Decrease in morning peak flow ≥20% on at least 2 consecutive days compared with baseline, and/or

- An increase in rescue medication use of ≥4 puffs on at least 2 consecutive days compared with the average use during baseline and/or
- >12 puffs of rescue medication in 1 day, and/or
- A night-time asthma symptom score of >baseline night-time score and ≥2 for at least 2 consecutive days, and/or
- A daytime asthma symptom score of 3 for at least 2 consecutive days

This alert should generate contact between the subject and the investigational site. The investigator then makes the decision whether or not to initiate (or escalate, as appropriate) treatment (ie, with inhaled or SCS and/or hospitalization).

### NB: An eDiary alert is not an asthma exacerbation per se.

Although the eDiary alert may initiate contact between the subject and the investigational site, the investigator or designee will always assess the subject's symptoms and determine whether to treat the subject for an exacerbation. Subjects will also be recommended not to take more than 8 puffs per day and advised to contact the study site/investigator if their symptoms necessitate more than 8 puffs in a day.

Asthma signs or symptoms will be recorded as AEs only when: the sign or symptom is serious, causes the subject to discontinue IP, or is new to the subject or inconsistent with the subject's pre-existing asthma history (Section 6.3.6)

# 5.1.2 Asthma Quality of Life Questionnaire+12/Pediatric Asthma Quality of Life Questionnaire

## 5.1.2.1 Asthma Quality of Life Questionnaire+12

The AQLQ+12 will be used in subjects 12 years and older. The AQLQ+12 will be selfadministered using an ePRO device during site visits as indicated in Table 1. Linguistically validated translations of the AQLQ+12 into local languages will be used.

The Asthma Quality of Life Questionnaire (AQLQ, Appendix F, Asthma Quality of Life +12 Questionnaire) was developed to measure the functional problems (physical, emotional, social, and occupational) that are most troublesome to adults with asthma.

There are 32 Questions in the AQLQ+12 and they are in 4 domains (symptoms, activity limitation comotional function, and environmental stimuli). The activity domain contains 5 subject specific questions. This allows subjects to select 5 activities in which they are most limited and these activities will be assessed at each follow-up. Subjects are asked to think about how they have been during the previous 2 weeks and to respond to each of the 32 questions on a point scale (7=not impaired at all; to 1=severely impaired). The overall AQLQ+12 score is the

The PAQLQ will be self-administered during site visits as indicated in Table 1 in subjects aged 7 to 11 years. Subjects aged 4 to 6 years will complete the questionnaire with the hold caregiver. As the PAQLQ is not validated for children less than 7 who are aged 4 to 6 years will be excluded 6

The subject/caregiver will complete the PAQLQ on paper and responses will be transcribed to the eCRF by site staff. Linguistically validated translations of the PAQLQ into local languages will be used.

The PAQLQ, (Appendix G, Pediatric Asthma Quality of Life Questionhaire) was developed to measure the functional problems (physical, emotional, and social) that are most troublesome to children with asthma.

The PAQLQ has 23 questions in 3 domains (symptoms, activity limitation, and emotional function). The activity domain contains 3 subject-secific questions. Children (subjects aged 7 to 11 years) are asked to think about how they the ve Geen during the previous week and to provide responses to each of the 23 questions a spoint scale (7=not bothered at all; 1=extremely bothered). The overall PAQL scotte is the mean of all 23 responses and the individual domain scores are the means of the terms in those domains.

### Asthma Control Question aire-5 and -7 5.1.3

The ACQ-5 will be administered using an ePRO device during site visits as indicated in Table 1. The ACQ-5 self-administered adult version will be used for adults and adolescents 11 years and older. As the ACQ is not validated for children less than 6 years old, the interviewer-administered version will be implemented for children aged 4 to 10 years. The questions take approximately 2 to 3 minutes to complete. Linguistically validated translations of the ACQ-5 into local languages will be used.

International guide the for the treatment of asthma have identified that the primary clinical goal of asthma management is to optimize asthma control (minimization of symptoms, activity limitation, broachoconstriction, and rescue β2-agonist use) and thus reduce the risk of life-threateting exacerbations and long-term morbidity. The Asthma Control Questionnaire (5-item persion; Appendix H, Asthma Control Questionnaire-5 and -7) was developed to meet these Arteria. It measures both the adequacy of asthma control and change in asthma control, which occurs either spontaneously or as a result of treatment.

The ACQ-5 questionnaire will be self-administered for adults and adolescents 11 years and older. The interviewer-administered version will be used for children aged 4 to 10 years.

Subjects will be asked to complete the ACQ-5, consisting of 5 questions on symptom control; each of the questions will be scored on a 7-point scale (0=excellent asthma control; 6=extremely poor control).

Note: The ACQ-7 will be completed once at screening only and consists of the top scoring 5 symptoms from the ACQ-5, with the addition of FEV<sub>1</sub>% predicted value and daily rescree bronchodilator use. Subjects are required to score ≥1.5 for eligibility to the study.

### 5.1.4 Asthma Control Test

The ACT will be self-administered using an ePRO device during site visits as indicated in Table 1. Linguistically validated translations of the ACT into local languages will be used.

The ACT (Appendix I, Asthma Control Test) is a 5-question health survey used to measure asthma control in subjects aged 12 and older. The survey measures the elements of asthma control as defined by the National Heart, Lung, and Blood Institute The ACT is an efficient, reliable, and valid method of measuring asthma control, with or without lung functioning measures such as spirometry.

The development of the ACT follows a paradigm shift in the treatment of asthma, from a focus on asthma severity to asthma control. Specifically, ACT helps identify and detect asthma subjects who are not well controlled. It was designed with input from asthma experts who helped establish cut-point scores to improve the chinical utility of the survey.

## 5.1.5 Childhood Asthma Control Pest

The C ACT will be self-administered using an ePRO device during site visits as indicated in Table 1. Linguistically validated translations of the C ACT into local languages will be used.

The C ACT report (Appendix J Childhood Asthma Control Test) is a validated tool for subjects aged 4 to 11 years to assess a shima control and identify children with inadequately controlled asthma.

## 5.1.6 eDiary

The eDiary will be attilized by all subjects enrolled in the study including children. Children, as necessary, will be assisted by a caregiver for the performance of assessments and navigation of the applicable questions.

## 5.1.6.1 Peak expiratory flow

Subjects will be trained at Visit 1. Throughout the study, subjects will record the best of 3 PEF measures on rising in the morning and before going to bed in the evening prior to taking any asthma therapy.

eDiary maintenance therapy compliance

Monitoring of compliance for medium-to-high-dose ICS or low-to-high-dose ICS combination with LABA will be done only through the eDiary question "have you taken regular maintenance therapy today?" (Appendix K, List of e-Diary question "have you taken collection of the actual devices for measurement/assessment vill be assessed by subject reported response " iken as compliant to dose and recombination to dose and recomb

#### 5.1.6.4 eDiary recording of asthma symptoms

The subject will use the eDiary for daily symptom reporting; intering symptoms twice daily.

The device will be programmed to alert both the subject and study center when the below prespecified alert thresholds are crossed. The purpose of the alerts is to trigger a documented contact between the site and subject for further valuation if deemed necessary by the investigator. Sponsor will also receive programmed alerts to monitor subject follow-up.

- subjects to signs of change of asthma and to contact their physician.
- A dedicated person from the Sporsor will review the ePRO and compliance alerts (2 consecutive days of missing data) and contact the site.
- In case of ePRO or compliance alerts, a qualified person from the site will contact the subject. For ePRO alerts the subject's asthma status should be evaluated and it will be determined if a clinic visit is necessary.

## An eDiary alert is not an asthma exacerbation per se.

Although the enter may initiate contact between the subject and the investigational site, the investigator or designee will always assess the subject's symptoms and determine whether to treat the subject for an exacerbation.

symptoms should be captured in (Appendix K, List of e-Diary questions). Asthraa symptoms should be captured in the eDiary by the subject every morning and evening

#### 5.1.7 Deterioration of asthma

In this study, deterioration of asthma is defined as 1 or more of the following items for ≥2. consecutive days:

- PEF: a decline of ≥20% from baseline
- Reliever therapy use: >4 puffs/day and  $\geq 2 \times baseline$
- Symptoms: night-time score that is >baseline and ≥2 OR a daytime score that is baseline and =3

Daytime is defined as the period between the morning lung function assessment (upon rising in the morning) and the evening lung function assessment.

Night-time is defined as the period between the evening lung function assessment (at bedtime) and the morning lung function assessment.

Severe asthma exacerbations will also be considered to be degrioration of asthma and included in the analyses of this endpoint.

# Lung function measurement by Spirometry 5.1.8

Prebronchodilator spirometry will be performed on a MasterScope provided for the study by the central reader at screening (Visit 1 and/or Visit 3 a, as applicable), Visit 2 (baseline), Visit 5 and Visit 6 (endpoint measurements). It is proportant that all spirometry assessments are performed after 06:00 and no later than 11:00 AM and that the spirometry at Visits 5 and 6 are performed ±1 hour in relation to the time of spirogetry at Visit 2. Preferably, the same study personnel should test the subject's lung function throughout the study to reach optimal performance and to enhance reproducibility. The subject should rest at least 15 minutes prior to the test. For repeated measurements eg, to assess best of 3, a short pause (1 minute) between measurements is recommended.

The measurements are to be made with the subject seated in an upright position (preferably), or if not comfortable standing position is also acceptable. The same position should be used for all spirometry measures during the entire study. The head must not be tilted during measurements. During the breathing maneuvers, the thorax should be able to move freely; hence tight clothing should be logsened.

Subjects should have previously discontinued bronchodilator medications as specified in Section 7.8.2 for reversibility tests as these can affect bronchodilation. If these medications west taken within the restricted time periods, visits should be re-scheduled.

Measurement procedures should be performed in accordance with the user manual for the study.

### 5.1.8.1 Reversibility Test

To fulfill the reversibility inclusion criterion, the increase in FEV₁ relative to baseline must be ≥12% (and ≥200 mL for subjects ≥18 years) approximately 30 minutes after inhalation of Sponsor-provided Ventolin.

Reversibility testing will be performed as follows:

- Determine if morning doses of all maintenance asthma medications (Table 4) were withheld and that short-acting bronchodilators were not administered within 6 hours of testing (if applicable).
- Perform prebronchodilator PFTs after at least 15 minutes of rest, and before administration of Ventolin.
- Subjects aged ≥12 years should administer 4 puffs of Ventolia. Subjects aged <12 years should administer 2 puffs of Ventolin.</li>
- 4. Perform post-bronchodilator PFTs approximately 30 monutes after the administration of Ventolin.

The reversibility is calculated as follows:

Reversibility=([Post FEV<sub>1</sub>-Pre FEV<sub>4</sub>)×100.

Pre-and postbronchodilator FEV<sub>1</sub> measurements will be captured within the MasterScope. If the reversibility inclusion criterion is not met as Visit 1, the reversibility test must be repeated at Visit 1a in advance of Visit 2 (randomization).

## 5.1.8.2 COVID-19 and Pulmosary Function Testing

In-clinic spirometry assessments should not be performed for subjects exhibiting signs and symptoms for COVID-19. Any suspected prior or active cases should have a diagnostic test to confirm COVID-19 status any subjects with confirmed COVID-19 should not perform spirometry assessments within 14 days of the cessation of symptoms and until the PI considers the subject is no longer infectious. Device cleaning and hygiene guidance should be followed at all times.

## 5.2 Safety assessments

Safety assessments include clinical laboratory (hematology, chemistry, morning serum cortisol, and presenancy tests for females of childbearing potential) parameters, 12-lead ECG readings, vital sign measurements, and collection of AEs.

Additional safety samples may be collected if clinically indicated, at the discretion of the investigator.

The clinical chemistry, hematology, serum cortisol assessments will be performed using a centralized laboratory. Sample tubes and sample sizes may vary depending method used and routine practice at the site. Table 2 Laboratory Safety Variables

| Hematology/Hemostasis (whole blood) | Clinical Chemistry (serum or plasma) |
|---|---|
| Basophils (%) | Albumin |
| Basophils Abs | Alanine transaminase |
| Eosinophils (%) | Alkaline phosphatase |
| Eosinophils Abs | Aspartate transaminase |
| Hemoglobin Hematocrit Mean Corpuscular Hemoglobin Mean Corpuscular Hemoglobin Concentration Mean Corpuscular Volume Monocytes (%) Monocytes Abs | Alirubin, total |
| Hematocrit Control | Calcium, total |
| Mean Corpuscular Hemoglobin | Chloride |
| Mean Corpuscular Hemoglobin Concentration | Cholesterol, total |
| Mean Corpuscular Volume | Creatinine |
| Monocytes (%) | Creatine kinase |
| Monocytes Abs | Gamma-glutamyl transpeptidase |
| Neutrophils (%) | Glucose (random) |
| Neutrophils Abs | Magnesium |
| Red blood cells (erythrocytes) | Phosphate |
| White blood cells (leukcoytes) | Potassium |
| Platelet count | Protein, total |
| Lymphocytes (%) | Sodium |
| Lymphocytes Abs | Triglycerides |
| 200 | Morning (serum) cortisol |
| Urine | Urea |
| Unite β-hCG pregnancy (Visit 2) a | Serum β-hCG pregnancy (Visit 1, 6 and EOS/PDV) |

\_ pregative previations: Abs=
Notes: Subreviations: Abs=absolute; β-hCG=β-human chorionic gonadotropin; EOS=end-of-study; PDV=premature

If a subject shows an AST or ALT ≥3× ULN and total bilirubin (TBL) ≥2×ULN please refer to a Section 3.9 and Appendix E, Hy's Law for further instructions.

5.2.2 Resting 12-lead electrocardiogram

A 12-lead ECG will be performed at the visits detailed in Table 1. The ECGs may be adjusted in Table 1.

ECGs may be adjusted in response to the emerging safety profile.

Twelve-lead ECGs will be obtained using a centralized laboratory after the subject has been resting semi-supine for at least 10 minutes. All ECGs should be recorded with the subject in the same physical position. A standardized ECG machine should be used and the subject should be examined using the same machine throughout the study, where feasible.

After paper ECGs have been recorded, the investigator or designated physician will review each of the ECGs and may refer to a local cardiologist, if appropriate. A paper copy should be filed in the subject's medical records. If an abnormal ECG finding at screening/baseline is considered to be clinically significant by the investigator, it should be reported as an AE. For all ECGs, details of rhythm, PR, RR, QRS, and QT intervals, an overall evaluation will be recorded.

5.2.3 Vital sign measurements

Vital signs including resting pulse and book pressure should be assessed at the visits detailed in Table 1. Measurements should be taken in the sitting position after at least 10 minutes of rest.

Any clinically significant changes in Stal signs should be recorded as an AE if applicable.

### 5.2.4 Adverse event assessments

Adverse events will be collected from time of signature of informed consent/assent through to the follow-up period as described in Section 6.

#### 5.3 Other assessments

### 5.3.1 Physical examination

A complete physical examination will be performed at screening and EOS/PDV as detailed in Table 1. Table will include an assessment of the following items: BMI (height in centimeters [for all subjects at Visit 1 and for subjects ≤18 years of age only at Week 24 (Visit 6) and EOS/QDV, as detailed in Table 1] and weight), general appearance, respiratory system, capstovascular system, abdomen, skin, head and neck (including ears, eyes, nose, and throat), Simph nodes, thyroid, musculoskeletal system (including spine and extremities), and neurological system.

### 5.3.2 Concomitant medications

The collection and recording of all concomitant medications, including all asthma therapies, will be performed at the visits detailed in Table 1. Permitted and restricted concomitant medications are descried in Section 7.8.

All prescription drugs, herbal products, vitamins, minerals, and over-the-counter medications taken within 3 months before screening will be recorded as previous medications. Astuma medication history will be recorded for 12 months before screening. All medications taken after screening and through the EOS/PDV visit will be recorded as concomitant therapy:

All asthma therapies taken during the study (Visit 1 through EOS/PDV) including SCS for exacerbations as well as concomitant ICSs will be recorded in the concomitant medication form in the subject's eCRF. Asthma maintenance therapy (ie, an ICS, or ICSCABA  $\pm$  1 of LTRA, LAMA, or theophylline) must be recorded at baseline. Any changes to the maintenance therapy presented at screening (Visit 1/1a, as applicable), including changes in dosing, will also be collected on the concomitant medication page in the eCRF.

Subjects will be maintained, after Visit 1, on their current maintenance regimen. Changes to maintenance therapy are discouraged unless clinically indicated. Investigators should contact the medical monitor assigned to the project in advance of any proposed change to maintenance therapy for study subjects; considerations should be made to subject drug compliance and other factors in advance of making changes to maintenance therapy.

For restrictions relating to concomitation medications see Sections 3.1 and 3.2.

## 5.4 Pharmacokinetics

Not applicable.

## 5.5 Pharmacodymamics

Not applicable.

## 5.6 Genetičš

Not applicable.

## 5.7 Biomarker analysis

Not appačable.

## 6 SAFETY REPORTING AND MEDICAL MANAGEMENT

The investigator is responsible for ensuring that all staff involved in the study is familiar with the content of this section.

Severe asthma exacerbations will be considered study efficacy endpoints and will not be reported as AEs unless considered an SAE. SAEs will be reported as per standard reporting guidance. Associated symptoms of asthma are considered as symptoms of disease under study and will not be recorded as AEs unless considered an SAE.

## 6.1 Definition of adverse events

An AE is the development of any untoward medical occurrence in a subject or clinical study subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, nausea, chest pain), or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

The term AE is used to include both serious and not serious AEs and can include a deterioration of a pre-existing medical occurrence. An AE may occur at any time, including the screening period, even if no IP has been administered.

# 6.2 Definitions of serious adverse event

An SAE is an AE occurring during and study phase (ie, after the signing of the informed consent/assent through to the safety follow-up visit), that fulfills 1 or more of the following criteria:

- Results in death
- Is immediately life-threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization.
- Results in persistent or significant disability or incapacity
- Is a congenital abnormality or birth defect
- Is an important medical event that may jeopardize the subject or may require medical intervention to prevent 1 of the outcomes listed above

For further guidance on the definition of an SAE, see Appendix D to the Clinical Study Protocol.

Adverse events and SAEs will be collected from time of signature of informed consent/assent through the safety follow-up period.

6.3.2 Follow-up of unresolved adverse events

Any AEs that are unresolved at the subject's last assessment visit in the study are follow-up by the investigator for as long as medically indicated that eCRF. The Sponsor content is subjected to the subject of the study are follow-up as medically indicated that eCRF. eCRF. The Sponsor or a Safety and Pharmacovigilance Department representative retains the right to request additional information for any subject with ongoing AE(s)/SAE(s) at the end of the study (after the subject's final study visit) and capture that information in the eCRF, if judged necessary.

#### 6.3.3 Variables

The following variables will be collected for each AE:

- The date when the AE started and stopped Maximum severity
- Seriousness
- Investigator causality rating against
- Action taken with regard to IP
- Outcome

In addition, the following variables will be collected for SAEs:

- Date AE met criteria for serious AE
- Date investigator became aware of serious AE
- Reason why the AE is considered serious
- given for the SAE
- Date of hospitalization
- Date of discharge
- Robable cause of death.
- Date of death.
  - Whether autopsy is performed.
- Causality assessment in relation to study procedure(s).

- Causality assessment to other medication.
- Description of AE.

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria in Section 6.2. An AE of severe intensity need not necessarily be considered serious. For example, nausea that persists for several hours may be considered severe nausea, but not an SAE unless it meets the criteria shown in Section 6.2. On the other hand, a stroke that results in only a limited degree of disability may be considered a mild stroke but would be an SAE when it satisfies the criteria shown in Section 6/2

The severity of the event should be assessed as mild, moderate, or severe.

The investigator and the Sponsor will assess causal relationship between IP and each AE, and answer "yes" or "no" to the question "Do you consider that there is a reasonable possibility that the event may have been caused by the IP?"

For SAEs, causal relationship will also be assessed for other medication and study procedures. Note that for SAEs that could be associated with any study procedure the causal relationship is implied as "yes".

existion is found in Appendix D of this Clinical A guide to the interpretation of the causa Study Protocol.

### Deteriorations of asthma and severe asthma exacerbations 6.3.5

All severe asthma exacerbations (Section 5.1.1.3) must be captured on the eCRF. Deterioration of asthma (Section 5.1.7) will be captured on the basis of symptoms as recorded by the subject in the eDiary. Severe asthma exacerbations will be considered expected study endpoints and will not be reported as AEs unless the Cilso meet the criteria for an SAE (Section 6.2).

### Adversegvents based on signs and symptoms 6.3.6

All AEs spontane sly reported by the subject or care provider or reported in response to the open question from the study site staff: "Have you/ your child had any health problems since the previous visit@ou (or your child) were last asked?" or revealed by observation will be collected and recorded in the eCRF. When collecting AEs, the recording of diagnosis is preferred (when ot signs and sympto other signs or symptoms that are not gene each sign or symptom will be recorded separately. possible over recording a list of signs and symptoms. However, if a diagnosis is known and there are other signs or symptoms that are not generally part of the diagnosis, the diagnosis and

Asthma symptoms or signs, such as wheeze, cough, chest tightness, dyspnea, breathlessness, and phlegm, will be recorded as AEs only when:

- The sign or symptom is serious.
- The subject discontinues IP due to the sign or symptom.
- The sign or symptom is new to the subject or not consistent with the subject's pre-existing asthma history (defined as within 1 year of Visit 1) as judged by the investigators.

### 6.3.7 Adverse events based on examinations and tests

The results from the Clinical Study Protocol mandated laboratory tests, ECOs, vital signs, and other safety assessments will be summarized in the Clinical Study Report. Deterioration from baseline in these parameters should therefore only be reported as an AE if it fulfills any of the AE criteria or is the reason for discontinuation of treatment with the IP or is considered "clinically significant".

The criteria for determining whether the mandated laboratory tests, ECGs, vital signs, and other safety assessments are clinically significant and should be reported as AEs are generally:

- Test result is associated with accompanying symptoms or signs, and/or
- Test result requires additional diagnostic testing or medical/surgical intervention, and/or
- Test result leads to a change in study downg or discontinuation from the study, significant
  additional concomitant drug treatment or other therapy, and/or
- Test result is considered to be an by the investigator or Sponsor.

If deterioration in a laboratory value, ECG, vital sign, or other safety assessment is associated with clinical signs and symptoms; the sign or symptom will be reported as an AE and the associated laboratory result/cital sign will be considered as additional information. Wherever possible, the reporting investigator uses the clinical, rather than the laboratory term (eg, anemia versus low hemoglobins value). In the absence of clinical signs or symptoms, clinically relevant deteriorations in nonmandated parameters should be reported as AE(s).

Any new or aggradated clinically relevant abnormal medical finding at a physical examination as compared with findings at the baseline assessment will be reported as an AE.

## 6.3.8 Thy's Law

Cases where a subject shows elevations in liver biochemistry may require further evaluation and occarrences of AST and/or ALT  $\ge 3 \times \text{ULN}$  combined and with TBL  $\ge 2 \times \text{ULN}$  may require IP suppension/discontinuation and study withdrawal, and may need to be reported as SAEs. Please refer to Section 3.9 and Appendix E, Hy's Law for further instruction on cases of increases in liver biochemistry and evaluation of Hy's Law.

#### 6.3.9 COVID-19 Adverse Events

For subjects experiencing signs and symptoms indicating respiratory infection, confirmatory testing for COVID-19 is expected in line with national guidelines.

Non-serious confirmed COVID-19 AEs will be recorded within the clinical database but additional information may be collected within the safety database and/or narratives as required.

If an SAE of COVID-19 infection is confirmed via testing, it should be reported witten diagnosis "COVID-19 confirmed" in the SAE report form. If COVID-19 infection is suspected, symptoms (eg, cough, fever, etc.) should be recorded in the SAE report form until diagnosis is confirmed. If test is not available and signs and symptoms, as judged by the investigator, are highly suspicious of COVID-19 infection, "COVID-19 suspected" should be reported.

All SAEs in relation to COVID-19 shall be reported in line with the instructions for SAE reporting described in Section 6.4.

Reporting of serious adverse events

All SAEs have to be reported, whether or not considered sousally related to the IP or to the study procedure(s). All SAEs will be recorded in the early

If any SAE occurs in the course of the study then it westigators or other site personnel should Safety and Pharmac Department within 1 day ie, immediately inform but no later than 24 hours of when he she becomes aware of it.

Should the eCRF system become nonoperational, SAEs shall be sent in paper form to:



Safety an Pharmacovigilance Department works with the investigator to ensure that all the necessary information is provided.

For fatal or life-threatening SAEs where important or relevant information is missing, active follow-up is wedertaken immediately.

Investigators or other site personnel should inform the Pharmacovigilance Department of any follow-up information on a previously reported SAE within 1 calendar day ie, immediately, but no later than 24 hours of when he or she becomes The Sponsor will also report to all applicable health authorities within 7 days of awareness for a fatal or life-threatening reaction or within 15 days for a reaction neither fatal nor life-threatening of any serious unexpected adverse drug reaction related to the drug which occurred during the study.

### 6.5 Overdose

For the purpose of this study, an accidental or deliberate intake of blinded treatment of more than 12 puffs during 1 day is defined as an overdose and must be reported as such as described below.

All overdoses must be recorded on the Overdose/Medication Error eCRF. Any associated AEs should also be recorded as the AE diagnosis/symptom on the relevant AE/SAE modules in the eCRF.

Investigators and the medical monitors will receive a safety notification alert from the subject's eDiary on a daily basis from any subject whose dosage exceeds & puffs in a single day. Upon receipt of alerts, the investigator will contact the subject to remaind them that they should not take more than 12 puffs per day. If indicated, the investigator will arrange an unscheduled clinic visit with the subject.

If an overdose occurs during the course of the study which has an associated SAE, then the investigator or other site personnel will inform the Safety and Pharmacovigilance Department immediately, or no later that 24 hours of when he or she becomes aware of the overdose.

The Safety and Pharmacovigilance Department works with the investigator to ensure that all relevant information is provided to the Safety and Pharmacovigilance Department representative.

For overdoses associated with an SAE, the standard SAE reporting timelines apply, see Section 6.4.

## 6.6 Pregnagor

All pregnancies and outcomes of the pregnancy should be reported to the study subject has received any IP.

Safety and Pharmacovagilance Department representative except if the pregnancy is discovered before the study subject has received any IP.

## 6.6.1 🖋 Maternal exposure

If a subject becomes pregnant during the course of the study, IP should be discontinued in mediately and "Pregnancy" recorded as the reason for discontinuation on the eCRF.

Pregnancy itself is not regarded as an AE unless there is a suspicion that the IP under study may have interfered with the effectiveness of a contraceptive medication. Congenital abnormalities/birth defects and spontaneous miscarriages should be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs. The outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal bank, or congenital abnormality) should be followed up and documented even if the subject was discontinued from the study.

If any pregnancy occurs in the course of the study, then the investigator or other specific personnel will inform the Safety and Pharmacovigilance Department within day ie, immediately, but no later than 24 hours of when he or she becomes aware of it. Any conception occurring from the date of dosing through the EOS/PDV should be reported.

The Safety and Pharmacovigilance Department will work with the investigator to ensure that all relevant information is provided.

The same timelines apply when outcome information is available.

## 6.6.2 Paternal exposure

Pregnancy of a subject's partner is not considered to be an AE. However, any conception occurring from the date of dosing through the EOS DV should be reported to the Safety and Pharmacovigilance Department representative and followed up for its outcome.

## 6.7 Medication error

For the purposes of this clinical study, a medication error is an unintended failure or mistake in the treatment process for the Sponsor's IP that either causes harm to the subject or has the potential to cause harm to the subject.

A medication error is not keek of efficacy of the drug, but rather a human or process related failure while the drug is in control of the study site staff or subject.

Medication error includes situations where an error:

- Occurred
- Was identified and intercepted before the subject received the drug
- . Disnot occur, but circumstances were recognized that could have led to an error

Kamples of events to be reported in clinical studies as medication errors:

- Drug name confusion
- Dispensing error eg, medication prepared incorrectly, even if it was not actually given to the subject
- Drug not administered as indicated, eg, wrong route or wrong site of administration
- Drug not taken as indicated
- Drug not stored as instructed eg, kept in the fridge when it should be at room temperature Wrong subject received the medication (excluding IWRS errors)
- Wrong drug administered to subject (excluding IWRS errors)

Examples of events that do not require reporting as medication errors in whical studies:

- Errors related to or resulting from IWRS-including those which lead to 1 of the above listed events that would otherwise have been a medication error
- Accidental overdose (will be captured as an overdose)
- Subject failed to return unused medication or empty packaging
- Errors related to background medication, or standard of care medication in open-label studies, even if it is a Sponsor's product

Ès may occur as a consequence of the Medication errors are not regarded as A medication error.

All medication errors must be recorded in the Overdose/Medication Error eCRF. Any associated AE should also be recorded as the AE diagnosis/symptom on the relevant AE/SAE modules in the eCRF. If a medication error occurs during the course of the study which has an associated SAE, then the investigator or other site personnel will inform the Safety and Pharmacovigilance Department immediately, or no later than 24 hours of when he or she becomes aware of the medication error.

Sety and Pharmacovigilance Department will work with the investigator to ensure that all relevant information is provided to the Pharmacovigilance Department representative. For medication errors associated with an SAE, the standard SAE reporting timelines apply (see Section 6.4).

## Management of investigational product-related toxicities

In the absence of a specific antidote, management of toxicities can be dealt with on the basis of symptoms.

BDA MDI is formulated (Table 3) as both micronized budesonide and micronized albuterol co-suspended with spray-dried porous particles in a hydrofluoroalkane (HFA) propellant. The co-suspension formulation ensures that subjects receive a consistent delivery of the drug each actuation of the MDI.

Investigational Product Strength and Dosage Form Table 3

| Investigational product name and dose | Product strength | Dosage Form/ Fill<br>Count | Administration | Manufacturer |
|---|---|---|---|---|
| BDA MDI<br>80/180 μg | BDA MDI<br>40 µg budesonide and<br>90 µg albuterol per<br>puff | MDI/120 actuations | Taken as 2<br>setuations | |
| BDA MDI<br>160/180 μg | BDA MDI<br>80 µg budesonide and<br>90 µg albuterol per<br>puff. | MDI/120 actuations | Taken as 2 actuations | |
| AS MDI 180 μg | AS MDI<br>90 μg albuterol per<br>puff <sup>a</sup> | MDN20; equations | Taken as 2<br>actuations | |
| Additional study medication | | | | |
| Ventolin HFA <sup>b</sup> | 108 μg albuterol sulfate (90 μg albuterol base) as an aerosol formulation | Albaterol (salbutamol)<br>sulfate inhalation<br>aerosol. 200 puffs per<br>canister | Use as needed<br>during screening<br>period | |

Albuterol sulfate (salbutamol sulfate) is a not investigational medicinal product since it is taken as directed for reversibility testing (Visit 1 and repeat Whit 1a, if necessary) and as needed for symptoms during the Screening Period.

### Dose and Treatment regimens 7.2

Investigational product will be used in response to asthma symptoms as subjects would normally take their reliever medication. If subjects take IP in advance of exercise for the prevention of exercise induced symptoms, IP usage in relation to exercise will be captured within the Diary. No other reliever products will be used during the treatment period.

At randomization (Visit 2), adolescents and adults (aged ≥12 years) who meet the eligibility criteria will be randomly assigned to 1 of the following 3 treatment groups in a 1:1:1 ratio as Riever therapy on top of usual care. Children aged 4 to 11 years will be randomized in a 1:1 ratio only to the lower BDA MDI dosage or AS MDI:

<sup>&</sup>lt;sup>a</sup> Each puff contains 108 μg albuterol soffate corresponding to 90 μg albuterol base per actuation

b Table represents commercially available Ventolin formulation for the United States, each country will utilize commercially available Ventolina that country, product strength may differ

- BDA MDI 80/180 µg (given as 2 actuations of BDA MDI 40/90 µg per puff) prn
- BDA MDI 160/180 μg (given as 2 actuations of BDA MDI 80/90 μg per puff) prn
- AS MDI 180 μg (given as 2 actuations of AS MDI 90 μg per puff) prn

Randomization for adolescents and adults will be stratified by age group (≥12 to 17, ≥18) region (North America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior screening (Visit 1plus any severe exacerbation event experienced during the screening period. Randomization for children will not be stratified.

The maximum daily dosage of IP should not exceed 12 puffs per day and subjects will be advised to contact the investigator if their symptoms necessitate more than 8 puffs per day (see Section 6.5 for overdose).

Handling instructions for the MDI device will be available for the site to train subjects and also for the subjects to retain throughout the study.

## 7.3 Labelling

Labels will be prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfill the prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfill the prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfill the prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfill the prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfill the prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines. The labels will fulfill the prepared in accordance with Good Manufacturing Practice (GMP) and local regulatory guidelines.

The subject will receive a kit contained 2 will devices, individually wrapped in foil bags held within a carton. The MDI devices provided in this study and the packaging and labelling of the kits are visually identical to maintain the blind. A kit will be dispensed for every 4 weeks of treatment. Each kit will contain the bollowing blinded labels:

- Single panel canister laber English only)
- Single panel actuator Bel (United States only) or multilanguage actuator booklet label
- MDI device shield abel (single panel, English only)
- Foil bag label (single panel, English only)
- Single panel arton label (United States only) or multilanguage carton booklet label

The labes will include the following information:

 Name of Sponsor (Bond Avillion 2 Development LP – Clinical Development Company: Avillion LLP)

- ion of such application Investigational product dosage form, route of administration, and quantity of dosage units (blinded across all arms)
- Storage conditions
- Study Trial Reference
- Medication ID number
- Directions for use
- The name of the investigator, where applicable (this will be added on the label annually when the IP is dispensed)

The label will include the following standard statements:

## 7.4

"For clinical study use only" (or the required local statement) of the "Keep out of reach of children"

Storage

's should be kept in a secure place under appropriate storage trainer readings of "

g der" All IPs should be kept in a secure place under appropriate storage conditions. The IP label on the carton specifies the appropriate storage are minimum/maximum) should be recorded on every working day at a minimum.

### 7.5 Compliance

The administration of all IPs will be captured in the subject's eDiary dose indicator readings and will be captured within the appropriate sections of the eCRF. Data from the dose counter will be compared with the subject's eDiary entries and any discrepancies will be used to help in training the subject to acceptately capture all IP administration in the eDiary.

The subject will be asked to record in their eDiary whether or not they have taken their maintenance theragy today via a yes/no question, which will be captured in the appropriate sections of the

### **Accountability** 7.6

The Ipprovided for this study will be used only as directed in the Clinical Study Protocol.

will be returned to the a will be returned to the will will be returned to the approved study returns vendor for destruction after accountability

document, which will cover all aspects of the trial with regards to IP. An "Instructions For Use" document can be found in Appendix L, Metered-dose Inhaler Handling and Cleaning for the IP MDI device.

The importance of the device cleaning and priming requirements should be emphasized to subjects. Device priming should not be conducted in the same room as spirometry, assessments are being conducted.

#### 7.8 Concomitant and other treatments

#### 7.8.1 Maintenance therapies

Inhaled corticosteroids (ICS)/LABA, LTRA, theophylline, and LAMAs are permitted to be used as maintenance therapy on study as specified in the inclusion criteria. No subject can be on >3 maintenance therapies.

During the study, subjects should maintain stable doing of their maintenance therapies as presented at screening (Visit 1/1a, as applicable). Ose Changes to maintenance therapy are discouraged unless clinically indicated in accordance with GINA guidelines. Investigators should notify the study medical monitors of the change to maintenance therapy for study subjects; considerations should be made to subject drug compliance and other factors in advance of making changes to maintenance therapy.

Subjects receiving maintenance allergy communotherapy (AIT) are allowed to continue their AIT; the initiation of AIT during the study is not allowed.

### 7.8.2 Medications that may affect reversibility and FEV1 testing

The medications presented in Table 4 may affect reversibility assessments. Investigators should notify the study medical pointors of any change to maintenance therapy for study subjects. If subjects have taken any of the medications below within the timeframe indicated of the planned reversibility test, the test should not be carried out and the subject should return to perform the reversibility testing

Table 4 Medications Restricted Time Limit Prior to any Lung Function Testing (reversibility and FEV1)

| | Restricted time limit before lung function |
|---|---|
| Medication | testing |
| SABA/Sponsor-provided Ventolin/Study | 6 hours |
| IP | 20 |
| Inhaled LABA | , io |
| Formoterol | 12 hours |
| Salmeterol | 12 hours |
| Olodaterol | 24 hours |
| Indacaterol | 24 hours |
| Vilanterol | 24 hours |
| LTRA | 24 hours |
| Theophylline twice daily | 12 hours |
| Theophylline once daily | 24 hours |
| LAMA | 24 hours 💥 |

Abbreviations: IP=investigational product; LABA=long-acting 62-agonist; LAMA=long-acting muscarinic antagonist; LTRA=leukotriene receptor antagonist.

#### 7.8.3 Prohibited medications

cotudy include: Prohibited concomitant medications during

- teresids (except if required to treat severe asthma Oral, parenteral, or rectal corticos exacerbation)
- Any other asthma medication except stable doses of maintenance therapy taken at entry into the study and provided by the Sponsor
- Inhaled disodium cromog vcate or inhaled nedocromil sodium
- 5-lipoxygenase inhibitors (ie, zileuton)
- Inhaled short-acting anticholinergics (or short-acting muscarinic antagonists [SAMA], ie, ipratropium)
- Inhaled long acting anticholinergies (LAMA), except those that were started before screening and continued as part of maintenance treatment (see inclusion criterion 4).
- Phosphodiesterase inhibitors (ie, roflumilast)
- monoclonal or polyclonal antibody therapy for any reasmonoclonal or polyclonal antibody therapy is allowed)

  Beta2-adrenergic blockers including and low daily doses Omalizumab, benralizumab, mepolizumab, reslizumab, dupilumab, or any other monoclonal or polyclonal antibody therapy for any reason (intra-ocular administration of

Beta2-adrenergic blockers including eye-drops (specific cardio-selective beta-blockers in low daily doses, eg, metoprolol in doses up to 100 mg/d, are allowed)

mitant treatment

And described in Section 7.8.1, which is considered in wellbeing, including short-term concomitant treatment win. to treat severe exacerbations, may be given at the discretion of the ecreption Other concomitant treatment

Medication other than that described in Section 7.8.1, which is considered necessary for the subject's safety and wellbeing, including short-term concomitant treatment with prohibited asthma treatments to treat severe exacerbations, may be given at the discount investigator and recorded in the appropriate sections of the section of the section of

All personnel involved with the analysis of the study will remain blinded until database lock and identification of Clinical Study Protocol violators.

Analyses will be performed by the Sponsor or its representatives.

The IDMC will have access to unblinded data in closed sessions with an unblinded statistician upon their request (see IDMC charter).

A comprehensive statistical analysis plan (analysis for the study will remain blinded until database lock and identification of Clinical Study Protocol violators.

Analyses will be performed by the Sponsor or its representatives.

analysis for IDMC and any subsequent amendments will be documented with final amendments completed before the unblinding of the data.

#### 8.1.1 Estimands

Three estimands are of interest in this study:

The primary estimand of interest is the efficacy estimand defined as the effect of the randomized treatment in all subjects assuming continuation of randomized treatment for the duration of the study, regardless of actual usage and assuming that maintenance therapy is not changed. This estimand could be considered as while-on-treatment strategy or a hypothetical strategy as defined in the draft International Conference on Harmonization (ICH) E9 addendum.

The second estimand of interest is the attributable estimand, defined as the effect of treatment in subjects attributable to the randomize reatment assuming that maintenance therapy is not changed. For this estimand, discontinuation of randomized treatment for tolerability or change in maintenance therapy for lack of asthma control is considered a negative outcome. This estimand is a mixture of composite and hypothetical strategies as defined in the draft ICH E9 addendum.

The third estimand of interest is the effectiveness estimand which is a combination of the hypothetical and treatment policy strategies as defined in the draft ICH E9 addendum. The strategy is hypothetical in that the treatment effect will be estimated without including data post the intercurrent event of discontinuation from randomized treatment. However, the strategy is consistent with the treatment policy strategy in that the treatment effect is estimated irrespective of the occurrence of the intercurrent event of a change in the maintenance therapy.

The fourth estimand of interest is the de facto estimand, defined as the effect of a treatment poor regardless of changes in maintenance therapy or premature discontinuation of andomized treatment. This estimand is considered a treatment policy strategy as defined in the draft ICH E9 addendum.
# 8.1.2 Primary outcome analysis

Primary outcome database lock (pDBL) will commence once all randomized adults (≥18 years) have attended their EOS visit at the PCD. The analyses of primary, secondary, exploratory and safety objectives will include all data up to the pDBL, which may include data for children (450 11 years) who are still on-going in the trial and have not yet completed the 24-week treatment period.

A final data base lock will occur after the pDBL, once all children have completed the EOS visit and safety follow-up.

Patient level listings of data for children who were on-going at the pDBL will be reported at the final database lock. No efficacy analyses will be conducted on data collected following the pDBL.

# 8.1.3 Type 1 error control

Comparisons of BDA MDI 80/180 µg versus AS MDI and BDA MDI 160/180 µg versus AS MDI for the primary endpoint, time to first severe exace pation using the efficacy estimand, will be conducted using Hochberg's step-up method (Hochberg 1988).

The type-I error will be controlled for secondary endpoint treatment comparisons via a hierarchical testing procedure. The following secondary endpoints will be tested under the efficacy estimand in the following sequential order, grouped by secondary endpoint:

Annualized severe exacerbation rate 4

- BDA MDI 160/180 μg versus ΔS MDI 180 μg
- BDA MDI 80/180 μg versus AS MDI 180 μg

Total annualized dose of systemic corticosteroid

- BDA MDI 160/300 μg versus AS MDI 180 μg
- BDA MDL 20/180 μg versus AS MDI 180 μg

Asthma Control Questionnaire-5 (ACQ-5) change from baseline responder analysis at Week 24

BDA MDI 160/180 μg versus AS MDI 180 μg

SDA MDI 80/180 μg versus AS MDI 180 μg

Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12) change from baseline responder analysis at Week 24

- BDA MDI 160/180 μg versus AS MDI 180 μg
- BDA MDI 80/180 μg versus AS MDI 180 μg

Statistical tests for the secondary analyses will be conducted at the 5% level of significance (2-sided). Inference for a test in the defined order is dependent on statistical significance been achieved in the preceding tests, if this is not achieved then nominal p-values will be provided. As per the primary analysis, comparisons of BDA MDI 160/180 versus AS MDI will exclude the pediatric population, whilst comparisons of BDA 80/180 versus AS MDI will include all ages.

Statistical significance can only be claimed on the key secondary endpoints of a statistically significant treatment effect is observed on both BDA MDI 160/180 µg and BDA MDI 80/180 µg versus AS MDI for the primary endpoint of time to first severe exacerbation.

# 8.2 Sample size estimate

A sample size of 1000 adult and adolescent subjects per treatment group and observation of the 570 first severe exacerbation events provides this study with 87% power to observe a 25% reduction in the risk of severe exacerbation with at least 2 dose of BDA MDI versus AS MDI assuming the Hochberg procedure (Hochberg 1988) for multiple testing and a 2-sided significance level of 5%.

In addition, up to 100 subjects in the 4 to 11 wear age group with moderate to severe asthma will be randomized with approximately 50 subjects randomized to the AS MDI group and 50 subjects randomized to the low dose ADA MDI group only.

# 8.3 Definitions of analysis sets

# 8.3.1 Full analysis set 🔊

The full analysis set (FAS) defined as all subjects who are randomized to treatment and take any amount of IP. Subjects will be analyzed according to the treatment they were assigned at randomization.

All efficacy analyses will be conducted in the FAS.

The efficacy and attributable estimand will include all data obtained up to pDBL, before subjects discontinue randomized treatment and/or before a change in maintenance therapy for lack of estima control. The effectiveness estimand will utilize all observed data up to randomized treatment discontinuation, regardless of whether subjects experience a change in maintenance therapy for lack of asthma control. The de facto estimand will utilize all observed data, including postIP discontinuation data, regardless of a change in maintenance therapy.

# 8.3.2 Safety analysis set

The safety analysis set is defined as all subjects receiving any amount of the IP. Subjects will be classified on the basis of treatment they actually received. If a subject receives more than 1 IP, he or she will be summarized according to the treatment the subject received the most. All safety summaries will be based on the safety analysis set.

## 8.4 Violations and deviations

Important protocol deviations will be listed and summarized by randomized treatment group. A per-protocol analysis excluding subjects with significant protocol deviations is not planned.

All subjects who failed any inclusion/exclusion criteria will be listed along with details of the failed criteria. This information will also be summarized in terms of the otimber and percentage of subjects failing any of the inclusion/exclusion criteria and will be based on the FAS.

# 8.5 Outcome measures for analyses

# 8.5.1 Primary efficacy analysis

The primary analysis will include all data obtained up to DBL, before subjects discontinue randomized treatment and/or before a change in maintenance therapy for lack of asthma control and will use the FAS, in accordance with the primary estimand (Section 8.1.1).

# 8.5.1.1 Derivation of time to first over asthma exacerbation

Time to first severe asthma exacerbation will be calculated as the time from randomization until the start date of the first severe asthma exacerbation:

Start date of first severe asthma excerbation - Date of randomization (Visit 2) +1

Subjects not having any severe asthma exacerbation will be censored at the date of their latest follow-up or EOS, for subjects who discontinue IP/have a change in maintenance therapy for lack of asthma control, the earliest of either day of discontinuation or day there was a change to maintenance therapy.

# 8.5.2 Secopdary efficacy analyses

The secondary analyses will include all data obtained up to the pDBL, before subjects discontinue randomized treatment and/or before a change in maintenance therapy for lack of asthma control and will use the FAS, in accordance with the primary estimand (see Section 8.1.1).

## 8.5.2.1 Derivation of annualized severe asthma exacerbation rate

For the production of summary statistics, the raw annualized severe asthma exacerbation rate will be calculated according to the following formula:

Annualized severe exacerbation rate=\sumber of severe exacerbations \*365.25/\sumber follow-wg, where the summations are over all subjects within a treatment arm.

For subjects who do not discontinue IP or do not receive a change in maintenance the apy for lack of asthma control, follow-up is calculated as:

[Date of latest follow-up or EOS] – [date of randomization (Visit 2)] – [cumulative duration of severe exacerbation(s)] + 1.

Otherwise, follow-up is calculated as the date of earliest occurrence of either IP discontinuation or change in maintenance therapy for lack of asthma control:

[Date of IP discontinuation/change in maintenance therapy] A [date of randomization (Visit 2)] - [cumulative duration of severe exacerbation(s)] + A.

# 8.5.2.2 Derivation of total systemic corticos drois exposure

Total systemic corticosteroid (SCS) exposure reported as the total annualized dose will be calculated for each subject as the sum of the current ative doses of corticosteroid divided by the duration of time (years) the subject was at the study, from randomization and up to treatment discontinuation.

Each SCS will be normalized to the empotent dose of prednisone (mg) before calculating the annualized total dose.

# 8.5.2.3 Derivation of Asthma Control Questionnaire-5 variables

All 5 symptom questions are assessed on a 7-point scale (0=good control; 6=poor control). The overall score is the mean of the 5 symptom items. At least 4 out of the 5 symptom items are needed to provide an ACQ-5 score.

The minimal important difference (MID) in ACQ-5 score is estimated to be 0.5 (Juniper 2005). On the basis of the MID, responders at Week 24 are defined as subjects achieving a decline from baseline of at least 0.5:

- Responder: (Week 24 baseline) ≤-0.5
- Nonresponder: (Week 24 baseline) >-0.5

Clinical Study Protocol, Version 4.0 Budesonide/albuterol (BDA) – AV003

Subjects who discontinue treatment for any reason or receive a change in maintenance therapy for lack of asthma control before Week 24 will be classified as nonresponders. Baseline is defined as the most recent non-missing score before and including randomization (Visit 2).

A similar analysis will be conducted at Week 12. This will be considered an exploratory endpoint.

Additionally, changes from baseline ACQ-5 overall score at Week 12 and Week 24 will be categorized into the exploratory 3-level factor:

- Improvement: (Week 24 baseline) ≤-0.5
- No Change: -0.5 < (Week 24 baseline) < 0.5</li>
- Worsening: (Week 24 baseline) ≥0.5

The interviewer-administered version will be implemented for children aged 4 to 10 years. As the ACQ-5 is not validated for children less than 6 years old; that for subjects who are 4 or 5 years of age will be excluded from the analyses of ACQ-5 endpoints.

# 8.5.2.4 Derivation of Asthma Quality of Life Questionnaire +12 and Pediatric Asthma Quality of Life Questionnaire yastables

As described in Section 5.1.2, there will be separate questionnaires for both adults and children. Both sets of questionnaires will be analyzed a similar manner.

AQLQ consists of 32 questions in 4 domains and PAQLQ consists of 23 questions in 3 domains. Both are assessed on separate 7-point Likert scales from 1 to 7, with higher values indicating better health-related quality of life.

For overall health-related quality of life and for each of the domains, the MID has been determined to be a change in score of 0.5 (Juniper 1994). On the basis of the MID, responders at Week 24 are defined as subjects achieving an increase from baseline of at least 0.5:

- Responder: (Week 24 baseline) ≥0.5
- Nonresponder: (Week 24 baseline) <0.5</li>

Subjects who discontinue treatment before Week 24 for any reason will be classified as nonresponders. Baseline is defined as the most recent non-missing score before and including randomization (Visit 2).

similar analysis will be conducted at Week 12. This will be considered an exploratory endpoint.

As the PAQLQ is not validated for children less than 7 years of age, data for subjects who are aged 4 to 6 years will be excluded from the analyses of PAQLQ endpoints.

# 8.5.3 Exploratory analyses

The exploratory analyses will include all data obtained up to the pDBL, before subjects discontinue randomized treatment and/or before a change in maintenance therapy for lack of asthma control and will use the FAS, in accordance with the primary estimand (see Section 8.1.1).

## 8.5.3.1 Derivation of deterioration of asthma variables

Time to first deterioration of asthma and the raw deterioration of asthma rate will be calculated in a similar way as to time to first severe asthma exacerbation (see Section 8.5.1.1) and the raw annualized severe asthma exacerbation rate (see Section 8.5.2.1).

# 8.5.3.2 Derivation of time to treatment discontinuation or change in maintenance therapy for lack of asthma control

Time to treatment discontinuation or change in maintenance therapy for lack of asthma control will be calculated as the time from randomization with the earliest of treatment discontinuation/change in maintenance therapy for lack of asthma control:

Date of IP discontinuation/change in main  $\hat{p}$  therapy –date of randomization (Visit 2) +1

Subjects not having prematurely discontinued treatment or receiving a change in maintenance therapy will be censored at the latest follow-up or EOS.

# 8.5.3.3 Derivation of Asthma Control Test responder variable

The MID in ACT score is estimated to be 3 (Schatz 2009). On the basis of the MID, the responders at Week 24 are defined as subjects achieving an increase from baseline of at least 3:

- Responder: (Week\$24 baseline) ≥ 3
- Nonresponder (Week 24 baseline) < 3</li>

Subjects who discontinue treatment for any reason or receive a change in maintenance therapy for lack of as toma control before Week 24 will be classified as nonresponders. Baseline is defined as the most recent non-missing score before and including randomization (Visit 2).

# 8.5.3 Derivation of other eDiary variables

# Symptom-free days

A symptom-free day is defined as the fulfillment of both of the following criteria:

- A day and night with no asthma symptoms (ie, asthma symptom score=0)
- A night with no awakenings due to asthma symptoms

## "As needed"-free days

An "as needed"-free day is defined as a day and night with no use of IP

## Asthma control days

An asthma control day is defined as the fulfillment of all of the following criteria

- A day and night with no asthma symptoms (ie, asthma symptom score

A night with no awakenings due to asthma symptoms
A day and night with no use of "as needed" medication
8.5.3.5 Inhaled corticosteroid exposure
Additional inhaled corticosteroid exposure from BDA MSS will be calculated as the total daily number of puffs of randomized treatment. number of puffs of randomized treatment.

orized into [low, medium, high] daily steroid Background maintenance therapy will be cated dose. Maintenance therapy categorizations will be based on prescribed daily dose of maintenance therapy steroids.

## Methods for statistical analyses 8.6

All tests will be 2-sided and at 5% level of significance unless otherwise stated. Adjustment will be made using the Hochberg procedure (Hochberg 1988) for the primary endpoint treatment comparisons.

In addition to the analyses described below, all variables will be summarized descriptively where appropriate.

### Analysts of the primary variable 8.6.1

The primary analysis will target the efficacy estimand in the FAS population. The primary variable, time to first severe asthma exacerbation, will be analyzed using a Cox proportional hazards regression model to compare treatment arms. The model will be adjusted for the random zation stratification factors (age group  $\geq 4$  to  $11, \geq 12$  to  $17, \geq 18$ ); region (North America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and not have prior severe exacerbations (1, >1) in the 12 months prior to screening (Visit 1) plus any severe exacerbation event experienced during the screening period and key covariates of interest with more detail to be provided in the SAP. The summary measure to compare

treatments is the estimated hazard ratio which will be presented with the corresponding 95% confidence interval and p-value.

The planned treatment comparisons for the primary analysis are:

- 1 BDA MDI 160/180 μg versus AS MDI 180 μg (superiority, primary objective)
- 2 BDA MDI 80/180 μg versus AS MDI 180 μg (superiority, primary objective)

The comparison of BDA MDI 160/180 μg versus AS MDI 180 μg will exclude the pediatric subjects (subjects aged 4 to 11 years) as they will not be randomized to BDA MDI 160/180 μg. For this analysis the age covariate will only have the 2 levels ≥12 to 17 and ≥8. However, the primary analysis for comparison of BDA MDI 80/180 μg versus AS MDI 200 μg will include subjects from all age groups.

Formally, the null and alternative hypotheses for comparisons 1 and 2 are:

H<sub>0</sub>: Hazard ratio (BDA MDI versus AS MDI)=1,

H<sub>A</sub>: Hazard ratio (BDA MDI versus AS MDI)≠1 €

All subjects who are randomized and are part of the full analysis set will be analyzed according to the strata they were allocated to in IVRS/IWRS A sensitivity analysis will be conducted based on subjects' actual strata to assess the impact of miss-stratification on the model results.

# 8.6.2 Analysis of the secondary edicacy variables

Analysis of the secondary efficacy variables will be on the FAS population. For all secondary analyses the same treatment comparisons as for the primary analysis will be conducted (see Section 8.6.1). Please see the hierarchical testing strategy for secondary endpoints (see Section 8.1.2).

# 8.6.2.1 Severe asthma exacerbation rate

Analysis of severe asthma exacerbation rate will target the efficacy estimand in the FAS population. Annualized severe asthma exacerbation rate will be analyzed using negative binomial regression to compare treatment groups. The response variable in the model will be the number of Severe asthma exacerbations. The model will adjust for (age group [≥ 4 to 11, ≥12 to 17, ≥18]); region (North America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to randomization) and key covariates of interest with more detail to be provided in the SAP.

The logarithm of the time at risk of experiencing an exacerbation will be used as an offset variable in the model. Time during an exacerbation or in the 7 days after an exacerbation will not be included in the calculation. From the negative binomial model, the annual severe asthma

exacerbation rates will be estimated, and the summary measure for the comparison of treatments will be the estimated rate ratio which will be presented with the corresponding 95% confidence interval and p-value.

The raw annualized exacerbation rate will also be summarized descriptively by treatment, using the derivation described in Section 8.5.2.1.

8.6.2.2 Asthma Control Questionnaire-5

The responder variable described in Section 8.5.2.3 at Week 24 will be analyzed using a logistic regression model to compare treatment groups. The model will be adjusted for the randomization stratification factors (age group [≥ 4 to 11, ≥12 to 17, ≥18]); region (North America, Western Europe and South Africa [Region 1] and rest of world Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to reening (Visit 1) plus any severe exacerbation event experienced during the screening period and key covariates of interest with more detail to be provided in the SAP. From the logistic regression model, treatment effects will be estimated by odds ratios and their corresponding 95% confidence intervals and p-values.

The exploratory endpoint for responder analysis at Week 2 and 3 factor categorization of ACQ-5 (Improvement; No change; Worsening) at Week 12 and Week 24 will be analyzed using an ordinal logistic regression and adjusting for the milar covariates. Full details of these analyses will be provided in the SAP.

Analysis of change from baseline in & Q-Sat Week 24 will target the efficacy estimand in the FAS population. The treatment effect for change from baseline in ACQ-5 will be estimated using a repeated measures analysis. A data up to Week 24 will be included in the model, with terms for treatment, visit, treatment visit, and baseline ACQ-5. The model will also be adjusted for the randomization stratification factors (age group  $\geq 4$  to  $11, \geq 12$  to  $17, \geq 18$ ); region (North America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to screening (Visit 1) plus any severe exacerbation event experienced during the screening period and key covariates of interest with more detail to be provided in the SAP. Visit will be fitted as a categorical variable, and the variance-covariance matrix will be assumed to be unstructured. If the procedure does not converge, then a compound symmetric variance-covariance matrix will be used instead. This model will be used to give an overall assessment of the treatment effect as well as 95 Confidence intervals.

Change from baseline will also be described descriptively for all study visits, including the EOS visit PDV and the safety follow-up telephone contact.

The all the scenarios above, baseline is defined as the most recent score before and including randomization (Visit 2).

## Asthma Quality of Life Questionnaire +12 and Pediatric Asthma Quality of 8.6.2.3 Life Questionnaire

The responder analysis will be conducted in the same way as ACQ-5 (Section 8.6.2.2). The exploratory endpoint for responder analysis at Week 12 will also be analyzed in a similar way.

The domain scores as well as the overall scores are calculated from the unweighted arithmetic means of the individual question scores. The treatment effect for change from baseline in AQLQ+12 and PAQLQ overall scores up to Week 24 will be estimated in the same way as ACQ-5, using a repeated measures analysis.

Change from baseline will also be described descriptively for all study visits including the EOS visit/PDV and safety follow-up telephone contact for each of the domains and the overall scores.

In all the scenarios above, baseline is defined as the most recent score before and including randomization (Visit 2).

### 8.6.2.4 Total systemic corticosteroid exposure

The total systemic corticosteroid exposure as total annualized dose of SCS (mg/year) will be presented descriptively by treatment. A companison in total annualized SCS dose between BDA MDI 80/180 vs AS MDI 180 and BDA MDI 180 vs AS MDI 180 will be analyzed using a Wilcoxon rank sum test and associated a Values will be presented along with the descriptive summary.

Additionally, the total SCS exposure with be summarized descriptively as the total number of days with SCS treatment due to asthmat for all subjects. A similar descriptive summary will be done for all subjects who administered at least 1 dose of SCS during the study.

### Analysis of safety variables 8.6.3

The safety analyses will include all data obtained before subjects discontinue randomized treatment and will use the safety analysis set.

### 8.6.3.1 Adverse events

Adverse eventa will be summarized by treatment group, system organ class and preferred term assigned to the event by the Medical Dictionary for Regulatory Activities. Adverse events will also be listed for each subject.

# Vital signs

Pressure. Measurements should be taken in the sitting position after at least 10 minutes of rest.

Clinical Study Protocol, Version 4.0 Budesonide/albuterol (BDA) – AV003

Baseline is defined as the most recent non-missing measurement before and including randomization (Visit 2).

### 8.6.3.3 Clinical chemistry and hematology

Clinical chemistry, hematology; and morning serum cortisol assessments will be summarized by treatment group and Visit and will also be listed by subject.

Baseline is defined as the most recent non-missing measurement before and including randomization (Visit 2)

randomization (Visit 2).

### 8.6.3.4 Concomitant medication

The number and percentage of subjects who take allowed concomitant medications, and those who take disallowed concomitant medications during the study, will be resented by treatment group.

### 8.6.4 Analysis of exploratory variables

The treatment comparisons in the secondary analyses given below are compared in the same way as the primary analysis.

### 8.6.4.1 Deterioration of asthma

Annualized deterioration of asthma and time of first deterioration of asthma will be analyzed in the same way as the time to first severe assuma exacerbation (Section 8.6.1) and annualized severe asthma exacerbation rate (Sec

### 8.6.4.2 Prebronchodilator FEV1

The treatment effect for change from baseline in FEV1 (mL) will be estimated using a MMRM analysis. FEV1 data from all visits up to Week 24 will be included in the model, with terms for treatment, visit and treatment sist with baseline FEV1 included as a covariate. The model will be adjusted for the randomization stratification factors (age group  $[\ge 4$  to  $11, \ge 12$  to  $17, \ge 18]$ ); region (North America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to screening (Visit 1) bus any severe exacerbation event experienced during the screening period and key covariate of interest with more detail to be provided in the SAP. Visit will be fitted as a categorical variable, and the variance-covariance matrix will be assumed to be unstructured. If the procedure does not converge then a compound symmetric variance- covariance matrix will be used instead. This model will be used to give assessments of the treatment effect as well as 95% confidence intervals at Week 12 and Week 24.

Reline is defined as the most recent non-missing measurement before and including Vandomization (Visit 2).

## 8.6.4.3 Morning peak expiratory flow

The mean value of change from baseline in morning PEF data during treatment will be analyzed by analysis of covariance with treatment as a factor and, baseline morning PEF score as a continuous covariate. The model will also be adjusted for the randomization stratification factors (age group [ $\geq 4$  to 11,  $\geq 12$  to 17,  $\geq 18$ ]); region (North America, Western Europe and South Africa [Region 1] and rest of world [Region 2]); and number of prior severe exacerbations (1, >1) in the 12 months prior to screening (Visit 1) plus any severe exacerbation event experienced during the screening period and key covariates of interest with prove detail to be provided in the SAP. The summary measure for the comparison of treatments will be the estimated mean difference, presented with the corresponding 95% confidence enterval.

Additionally a repeated measures analysis will be conducted and will be partitioned into 4-weekly time intervals across the randomized treatment period. The adalysis model will additionally include time point and treatment\*time point as factors and associated p-value.

Change from baseline in morning PEF will also be summarized for each subject by treatment group using summary statistics.

For all scenarios above, baseline morning PEF is defined as the average during the 10 days prior to randomization (Visit 2) during run-in. Morning PEF will be captured via the eDiary.

# 8.6.4.4 Other eDiary variables

Evening PEF, reliever therapy use, asthma symptoms (day, night, and total), night-time awakenings due to asthma symptoms, symptom-free days, "as needed"-free days and asthma control days will be analyzed in the same way as the morning PEF.

Baseline is defined as the average dring the 10 days prior to randomization (Visit 2) during run-in.

# 8.6.4.5 Time to treatment discontinuation or change in maintenance therapy for lack of asthma control

Time to treatment discontinuation or change in maintenance therapy for lack of asthma control will be analyzed apper the primary analysis described in Section 8.6.1.

## 8.6.4.6 Asimma Control Test

The ACT/C ACT will be summarized as per the secondary analysis of change from baseline and responder analysis in ACQ-5 in Section 8.6.2.2.

Baseline is defined as the most recent non-missing score before and including randomization Visit 2).

a randomized treatment will be summaries of the main daily number of subgroups of background maintenance therapy

, medium, high] daily dose.

3.0.5 Subgroup analysis

The assessment of treatment effect will be investigated in the stratification variable and other clinically important subgroups and will be defined in more detail in the SAP.

1.6.6 Sensitivity analysis

6.6.1 Tipping point and ultiple important subgroups and will be defined in more detail in the same of the stratification variable and other clinically important subgroups and will be defined in more detail in the same of the stratification variable and other clinically important subgroups and will be defined in more detail in the same of the stratification variable and other clinically important subgroups and will be defined in more detail in the same of the stratification variable and other clinically important subgroups and will be defined in more detail in the same of the stratification variable and other clinically important subgroups and will be defined in more detail in the same of the s

Multiple imputation tipping point analysis under the missing net at random assumption will be conducted. For subjects in the BDA MDI groups, this method will impute missing values poststudy discontinuation/change in maintenance for lack of asthma control assuming they were more likely to have a severe asthma exacerbation event than as implied under the missing at random assumption. The tipping point analysis will look at by how much the event rate would need to increase for the result to become nor significant. The full details of the analysis will be specified in the SAP.

## Attributable estimand 🔏 8.6.6.2

Analysis of the attributable estimand will be conducted using data obtained before subjects discontinue randomized treatment and or before a change in maintenance therapy for lack of asthma control and will use the FAS. However, the data that is missing due to randomized treatment discontinuation and/och change in maintenance therapy will be imputed on the basis of the 95th or 5th percentile of the AS MDI prn distribution if the reason is reasonably attributable to tolerability or lack of control. The 95th percentile would apply to an endpoint for which a higher value is worse outcome while the 5th percentile would apply to an endpoint for which a higher value a better outcome. More detail about the computation of the attributable estimand will be provided in the SAP.

### 8.6.6.3 E**G**éctiveness estimand

Analysis of the effectiveness estimand will be conducted in the FAS in which all observed data will be wilized regardless of whether subjects experience a change in maintenance therapy for lackof asthma control.


COVID-19 pandemic impacts

As the trial is on-going during COVID-19 pandemic, it will be necessary to evaluate and potential intercurrent events due to COVID-19 and quantify their impact on the efficiency and safety profile of the study IP.

As a minimum, the number of missed visite to conducted will be summer roups. When groups. Where appropriate, the subject level data for missed visits and sessments will be listed along with the corresponding link to COVID-19, as recorded in the RF. It is not anticipated that missing data and premature withdrawals due to COVID-19 will be related to randomized treatment. Therefore, missing data due to COVID-19 will be assumed missing at random in accordance with the efficacy estimand. If further sensitivity malyses are deemed necessary following a blinded review of missing efficacy due to COVID-19, further details will be provided in the SAP, prior to database lock and unDlinging.

Similarly, as a minimum, the number of schedule safety assessments missed due to COVID-19 will be summarized descriptively by treatment groups. Subjects with suspected or confirmed diagnosis of COVID-19, and/or COVID-19 related AEs and SAEs will be summarized descriptively. Subject evel istings of missed scheduled safety assessments and

## 9 STUDY AND DATA MANAGEMENT

## 9.1 Training of study site staff

Before the first subject is entered into the study, a designated representative will review and discuss the requirements of the Clinical Study Protocol and related documents with the investigational staff and also train them in any study specific procedures and the Rave WBDC system(s) utilized.

The investigator will ensure that appropriate training relevant to the study is given all of these staff, and that any new information relevant to the performance of this study is forwarded to the staff involved.

The investigator will maintain a record of all individuals involved in the study (medical, nursing, and other staff).

# 9.2 Monitoring of the study

During the study, the Sponsor or a designated representative will have regular contacts with the study site, including visits to:

- Provide information and support to the investigator(s)
- Confirm that facilities remain acceptable
- Confirm that the investigational team is a thering to the Clinical Study Protocol, that data
  are being accurately and timely resorded in the eCRFs, that biological samples are handled
  in accordance with the Laboratory Manual, and that IP accountability checks are being
  performed
- Perform source data verification (a comparison of the data in the eCRFs with the subject's
  medical records at the hospital or practice, and other records relevant to the study)
  including verification of informed consent/assent of participating subjects. This will require
  direct access to all original records for each subject (eg, clinic charts)
- Ensure all SAEs and AEs have been captured and reported correctly, providing oversight of subject safety while on study
- Verify the confect storage, handling, dispensation, and return of all IP
- Ensure wiredrawal of informed consent/assent to the use of the subject's biological samples
  is reported and biological samples are identified and disposed of/destroyed accordingly, and
  the action is documented, and reported to the subject

The designated representative will be available between visits if the investigator(s) or other staff the center needs information and advice about the conduct of the study.

Data entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need available.

Definition of what constitutes source data can be found in the Source Data Agreement, agreed with each investigator before site initiation with each investigator before site initiation.

### 9.2.2 Study agreements

The investigator/participating center should comply with all the terms, conditions, and obligations of the Clinical Study Protocol, or equivalent, for this study.

Clinical Trial Agreements with the investigator/participating center should be in place before any study-related procedures can take place, or subjects are enrolled.

### 9.2.3 Archiving of study documents

in the Clinical Trial Agreement. The investigator follows the principles outlined

# 9.3

All randomized subjects who do not prematurely discontinue will have a minimum of 24 weeks of treatment. The study treatment period will continue (extension phase) until the required 570 first severe exacerbation events, as defined per protocol, have been reached; and the last subject has completed 24 weeks of treatment. The EOS visit will be planned once the 570 first severe exacerbation events occur. If a subject's treatment is ≥24 weeks then the subject's EOS visit will occur at their next scheduled clinic visit. Once the PCD has been reached, any ongoing subject ≥24 weeks will return to complete their EOS visit at their next scheduled clinic visit. The safety follow-up delephone contact will occur 2 weeks (±4 days) after EOS or PDV, if applicable. The encof the study is defined as "the last visit of the last subject undergoing the study".

The study may be terminated at individual centers if the study procedures are not being performed according to Good Clinical Practice (GCP), or if recruitment is slow. The Sponsor may also terminate the entire study prematurely if concerns for safety arise within this study or in ny other study with BDA MDI.


The data collected through third party sources will be obtained and reconciled against study. The data from third parties will be transferred in accordance with data transfer specificant and reconciled in accordance with the Data Management Plan.

Adverse events and modification.

the latest version of the Medical Dictionary for Regulatory Activities at the time of database lock. Medications will be classified according to the World Health Organization Drug Dictionary. All coding will be performed by the Medical Coding Team at

Data queries will be raised for inconsistent, impossible, or missing data. All entries to the study database will be available in an audit trail.

The data will be validated as defined in the Data Management Plan. Quality control procedures will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. The Data Management Plan will also clarify the roles and responsibilities of the various functions and personnel involved by the data management process.

Serious AE reconciliation reports are produced and reconciled with the applicable Safety and Pharmacovigilance Separament safety database and/or the investigational site.

# Management of external data

Data Management will set up import agreements with third party data sources, to ensure external data is integrated in line with applicable data standards.

# Primary outcome database lock

When all required 570 art severe exacerbation events have occurred and the last adult subject has completed 24 weeks of treatment and safety follow-up, the data cleaning should be completed for the Frimary outcome database lock. Database lock will occur once all data have been coded, validated, signed, and locked, and clean file has been declared. Data will be unblinded at the primary outcome database lock.

# Final database lock

The tudy treatment period will continue for children (4 to 11 years) and adolescents (12 to ₹Years) who have not completed 24 weeks of treatment by the time of the primary outcome database lock. The safety follow-up telephone contact will occur 2 weeks (±4 days) after EOS The bother little backet of the land of th

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/GCP and applicable regulatory requirements.

10.2 Subject data protection

The informed consent/assent form will incorporate (or, in some cases 1 separate document incorporatino) wonders are privated.

privacy legislation.

Subjects will be assigned a unique identifier by the Sponsor. Any subject records or datasets that are transferred to the Sponsor will contain the identifier only; specified names or any information which would make the subject identifiable will not be transferred. Subjects must be informed that his/her personal study-related data will be used to the Sponsor in accordance with local data protection law. The level of disclosure must also be explained to the subject. Subjects must also be informed that his/her medical records may be examined by study monitors, clinical quality assurance auditors, or other authorized personne appointed by the Sponsor, by appropriate EC members, and by inspectors from regulatory authorities.

### Ethics and regulatory reflex 10.3

An EC should approve the final Clinical Study Protocol, including the final version of the informed consent/assent form and any other written information and/or materials to be provided to the subjects. The investigator will sure the distribution of these documents to the applicable EC and to the study site staff.

The opinion of the EC should be given in writing. The investigator should submit the written approval to the Sponsor or designated representative before enrollment of any subject into the study.

The EC should approve all advertising used to recruit subjects for the study.

The Sponsor or designated representative should approve any modifications to the informed consent/asset form that are needed to meet local requirements.

If required by local regulations, the Clinical Study Protocol should be re-approved by the EC annually

Final version of the informed consent/assent form, is approved by the national regulatory Sefore enrollment of any subject into the study, the final Clinical Study Protocol, including the

- The Sponsor or designated representative handles the distribution of any of these documents to additional regulatory authorities.

  The Sponsor or designated representative will provide regulatory authorities, ECs, and investigators with safety updates/reports according to local requirements.

  10.4 Informed consent/assent

  The investigator(s) at each center will:

   Ensure each subject and/or parent/legal representative (as applicable) is given full and adequate oral and written information about the nature, purpose possible risks, and benefit of the study

   Ensure each subject and/or parent/legal representative (as applicable) is given full and adequate oral and written information about the nature, purpose possible risks, and benefit of the study
  - Ensure each subject and/or parent/legal representative is notified that they are free to discontinue from the study at any time
  - Ensure that each subject and/or parent/legal representative is given the opportunity to ask questions and allowed time to consider the information provided
- Ensure each subject and/or parent/legal representative provides signed and dated informed consent/assent before conducting any procedure specifically for the study
- Ensure the original, signed informed consent/assent form(s) is/are stored in the investigator's study file
- Ensure a copy of the signed informed consent/assent form is given to the subject
- Ensure that any incentives for so jects who participate in the study as well as any provisions for subjects harmed as a consequence of study participation are described in the informed consent/assent form that is approved by an EC

# Changes to the clinical study protocol and informed consent/assent 10.5

Study procedures will not be changed without the mutual agreement of the international coordinating in estigator and the Sponsor.

If there are any substantial changes to the Clinical Study Protocol, then these changes will be documented in a new version of the study protocol.

The new version of the Clinical Study Protocol is to be approved by the relevant EC and if applicable, also the national regulatory authority, before implementation. Local requirements are to be followed for new versions of Clinical Study Protocols.

If a change to a Clinical Study Protocol requires a change to a center's informed consent/assent of form, the Sponsor and the center's EC are to approve (or a notification to the national authority is submitted where applicable for) the revised form is to the national authority is submitted where applicable for the revised form is to the national authority is submitted where applicable for the revised form is to the national authority is submitted where applicable for the revised form is to the national authority is submitted where applicable for the revised form is to the national authority is submitted where applicable for the national authority is submitted where a national author and a national authority is submitted where a national authority

As of the Clinic
Section 10.3.

Jool requires a change to a
s EC are to approve (or a notit
plicable for) the revised informed

Attives of the Sponsor, a regulatory authority, or an.
the center, including source data ventication. The purpo
systematically and independently examine all study-related to determine whether these activities were conducted, data erre a
ately reported according to the Clinical Study Protocol, Gest, guidel
applicable regulatory requirements. The investigator will contact the Sp.
ediately if contacted by a regulatory agency about an inspection at the center

And Adams to the Clinical Study Protocol, Gest, guidel
applicable regulatory agency about an inspection at the center

And Adams to the Clinical Study Protocol, Gest, guidel
applicable regulatory requirements. The investigator will contact the Sp.
adams to the Clinical Study Protocol, Gest, guidel
applicable regulatory requirements. The investigatory requirements are applicable regulatory requirements. The investigatory requirements are applicable regulatory requirements. The 10.6 Audits and inspections

Authorized representatives of the Sponsor, a regulatory authority, or an EC may perform audits or inspections at the center, including source data verification. The or inspections at the center, including source data verification. The purpose of an audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, data were recorded, analyzed, and accurately reported according to the Clinical Study Protocol, GCB, guidelines of the ICH, and any applicable regulatory requirements. The investigator wilk contact the Sponsor


## 11 LIST OF REFERENCES

- American Academy of Allergy Asthma and Immunology (AAAAI). COVID-19 and Asthma: What Patients Need to Know. 04 Jun 2020. Accessed 19 Jun 2020. https://www.aaaai.org/conditions-and-treatments/library/asthma-library/covid-asthma
- Cooper PR, Panettieri RA. Steroids completely reverse albuterol-induced β2-adrener or receptor tolerance in human small airways. J Allergy Clin Immunol 2008;122(4):394-740.
- 3. Hochberg Y. A sharper Bonferroni procedure for multiple tests of significance. Biometrika 1988;75(4):800-802.
- Global Initiative for Asthma. Global strategy for asthma management and prevention. 2018. Available from: https://ginasthma.org/wp-content/uploads/2018/04/wms-GINA-2018-report-V1.3-002.pdf.
- Investigator Brochure Edition 2.0. Budesonide/Albuterol Sulfate Pressurized Inhalation Suspension (BDA MDI, PT027); Budesonide Pressurized Inhalation Suspension (BD MDI, PT008); Albuterol Sulfate Pressurized Inhalation Suspension (AS MDI, PT007), 20 September 2019.
- Juniper EF, Svensson K, Mörk AC, Ståhl E, Messurement properties and interpretation of three shortened versions of the asthma control questionnaire. Respir Med 2005;99(5):553-558.
- Juniper EF, Guyatt GH, Willan A Griffith LE. Determining a minimal important change in a disease-specific quality of life questionnaire. J Clin Epidemiol 1994;47:81-87.
- Mendes ES, Horvath G, Camp & M, Wanner A. Rapid corticosteroid effect on β(2)adrenergic airway and airway vascular reactivity in patients with mild asthma. J Allergy Clin Immunol 2008;121(3):700-704.
- Mendes ES, Cadet LoArana J, Wanner A. Acute effect of an inhaled glucocorticosteroid on albuterol-induced bronchodilation in patients with moderately severe asthma. Chest 2015;147(4):1637-1042.
- O'Byrne RM, Bisgaard H, Godard PP, Pistolesi M, Palmqvist M, Zhu Y, et al. Budesoude/formoterol combination therapy as both maintenance and reliever medication in astima. Am J Respir Crit Care Med 2005;171(2):129-136.
- 11. O'Byrne PM. Acute asthma intervention: insights from the STAY study. J Allergy Clin Immunol 2007;119(6):1332-1336.

- Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the asthma control test. J Allergy Clin Immunol 2009;124:718-723.

  Tattersfield AE, Postma DS, Barnes PJ, Svensson K, Banar C.

  Exacerbations of asthma: a descriptive international Study. 12. Rabe KF, Atienza T, Magyar P, Larsson P, Jorup C, Lalloo UG. Effect of budesonide in
- 13. Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally
- , Larsson P, Jorup C, \( \times \) . for reliever therapy in ast. ady. Lancet 2006;368(9537):7-,

  , Yarlas AS, Hanlon J, Watson ME, Jha. of the asthma control test. J Allergy Clin In.

  ., Postma DS, Barnes PJ, Svensson K, Bauer CA, O'By. as of asthma: a descriptive study of 425 severe exacerbation. all Study Group. Am J Respir Crit Care Med 1999;160(2):594. Standard of the study of 425 severe exacerbation and Study Group. Am J Respir Crit Care Med 1999;160(2):594. Standard of the study of 425 severe exacerbation and Study Group. Am J Respir Crit Care Med 1999;160(2):594. Standard of the standard of 14. Tattersfield AE, Postma DS, Barnes PJ, Svensson K, Bauer CA, O'Byrne PM al.

  Exacerbations of asthma: a descriptive study of 425 severe current.

# 12 SUMMARY OF CHANGES

# 12.1 Changes made to Version 3.0

| Section | Changes made to Version 3.0, 21 July 2020 to |
|---|---|
| | develop global amendment, Version 4.0, |
| | Changes made to Version 3.0, 21 July 2020 to develop global amendment, Version 4.0, 08April 2021 |
| | ,O` |
| Cover page/Version History | Date and version changed; updated sponsor address; |
| | brief summary of amendment added. |
| Clinical Study Protocol Synopsis | Updated the estimated date of last subject completed |
| | from Q3 2021 to Q1 2022. |
| Clinical Study Protocol Synopsis | Clarification that up to 100 subjects in the 4 to 11-year |
| 3.3 Subject enrollment and | age group with moderate to severe asthma will be |
| randomization; | randomized. |
| 8.2 Sample size estimate | rio <sup>f</sup> |
| - | 4B. |
| Clinical Study Protocol Synopsis | Clarification that the treatment period will continue |
| 1.2 Rationale for study design, | until the lost adout subject has completed 24 weeks of |
| doses, and control groups, | Clarification that the treatment period will continue until the less adult subject has completed 24 weeks of treatment |
| 1.4 Study design; | G it's |
| Table 1, footnote c; | OF MO |
| 4.2 Randomization/treatment | E. B. |
| period/extension phase | in <sup>©</sup> |
| Clinical Study Protocol Symansis | Clarification that padiatria subjects will continue until |
| Chinical Study Protocol Synopsis | Clarification that pediatric subjects will continue until<br>24 weeks of treatment have been reached for each |
| 4 | pediatric patient, defined as the final completion date. |
| Clinical Study Protocol SynOpsis; | Clarification that the primary efficacy analysis will |
| 8.5.1 Primary efficacy agalysis | include all data up to the PCD. |
| J. J | |
| Clinical Study Protocol Synopsis; | Clarification that the secondary efficacy analysis will |
| 8.5.2 Secondary efficacy analyses | include all data up to the PCD. |
| 1.2 Rational@for study design; | Clarification that not all pediatric subjects will have |
| doses, and control groups; | 24 weeks of treatment at time of PCD. |
| 1.4 Stady design | |
| all' | |

|---|---|
| | develop global amendment, Version 4.0, |
| | 08April 2021 |
| | 0014PII 2021 |
| 3.1 Inclusion criteria #6 | Clarification that subjects aged ≥12 years of age mustodemonstrate reversibility at Visit 1. |
| | demonstrate reversibility at Visit 1. |
| | <u> </u> |
| | Added the following sentence: Subjects aged |
| | 11 years of age will perform the reversibility test, but |
| | do not require demonstration of reversibility during |
| | Visit 1 and may enroll, provided documented historical |
| | reversibility within 1 year is available. Subjects aged |
| | 4 to 11 years who previously failed inclusion criterion 6 |
| | will be permitted to rescreen. Each subject may |
| | re-screen only once. |
| | 0 |
| 3.1 Inclusion criteria #17, | Added additional forms of birth control: a condom with |
| subbullet ii | spermicide, atrapterine device (IUD), or intrauterine |
| Subbunet n | hormone-celeasting system (IUS). |
| | normone-treasing system (103). |
| 4.1 Screening and run-in period | Updated that subjects aged 4 to 11 years of age who |
| | previously failed inclusion criterion 6 will be permitted |
| | to resoreen. |
| • | F. 6 |
| 4.2 Randomization/treatment | added that children and adolescents ongoing in |
| period/extension phase | treatment after the PCD will continue in follow-up until |
| 1 Kil | they have completed 24 weeks of treatment. |
| 5.2.1 Laboratory safety | Added serum cortisol assessments along with those for |
| assessments | chemistry and hematology. |
| New section: 8.1.2 Primary | Primary outcome database lock (pDBL) will commence |
| outcome analysis(subsequent | once all randomized adults (≥18 years) have attended |
| heading numbering updated) | their EOS visit at the PCD. The analyses of primary, |
| ∑® ̃ | secondary, exploratory, and safety objectives will |
| Į "Š" | include all data up to the pDBL, which may include |
| , a <sup>1</sup> | data for children (4 to 11 years) who are still on-going |
| RIVE | in the trial and have not yet completed the 24-week |
| ă. | treatment period. |
| w. | |

|---|---|
| Section | develop global amendment, Version 4.0, |
| | 08April 2021 |
| | 00Aprii 2021 |
| | A final data base lock will occur after the pDBL, once |
| | all children have completed the EOS visit and safe |
| | follow-up. |
| | Patient level listings of data for children whewere on- |
| | going at the pDBL will be reported at the Tinal database |
| | lock. No efficacy analyses will be conducted on data |
| | collected following the pDBL. |
| | aiio |
| 8.3.1 Full analysis set | Clarification that efficacy and attributable estimand will |
| | include all data obtained up 🎓 pDBL. |
| 8.5.3 Exploratory analyses | Clarification that the exploratory analyses will include |
| | all data obtained up to OBL. |
| 8.5.3.5 Total inhaled | Headings revised: |
| corticosteroid exposure; | 0.8 |
| 8.6.4.7 Total inhaled | 8.5.3.5 Inhaled Corticosteroid exposure |
| corticosteroid exposure | 8.6.4 Tinhared corticosteroid exposure |
| | 8.0.4 minated corticosteroid exposure |
| | Text revised to describe categories for maintenance |
| <b> </b> | Therapy in addition to methods used to calculate and |
| | malyze inhaled corticosteroid exposure. |
| 8 | 8 |
| 8.6.6 Primary outcome analysis | Section removed; subsequent heading numbering |
| 4 | updated |
| *** | |
| 9.3 Study timetable and pad-of-study 9.4 Data management | Updated that all randomized subjects who do not |
| study (N) | prematurely discontinue will have a minimum of |
| ્રું | 24 weeks of treatment. |
| ø | D 14 14 4 1 5 1 D D D |
| 35 | Deleted text defining PCD. |
| , % | Once the PCD has been reached, any ongoing subject |
| KO. | ≥24 weeks will return to complete their EOS visit at |
| (\$ T | their next scheduled clinic visit |
| OM Data management | Derviced to elevify that when the last adult subject her |
| 9 A Data management | Revised to clarify that when the last adult subject has |
| <b>6</b> | completed 24 weeks of treatment and safety follow-up, |

|---|---|
| | develop global amendment, Version 4.0, |
| | 08April 2021 |
| | 8 |
| | the data cleaning should be completed for the primary |
| | the data cleaning should be completed for the primary outcome database lock. |
| | Final database lock revised to clarify that study |
| | treatment period will continue for children to |
| | 11 years) and adolescents (12 to 17 years) who have not |
| | completed 24 weeks of treatment by the time of the |
| | primary outcome database lock. |
| Throughout dogument | Additional nonsubstantial changes for administrative, |
| Throughout document | |
| | typographical, and/or grammatical corrections were |
| | made. |
| | O. |

# 12.2

| | :or |
|---|---|
| Section Changes made to Version 2.0 Changes made to Version 2.0, 29 July 2019 to develop global amendment, Version 3.0, | |
| Section | Change mixe to Version 2.0, 29 July 2019 to develop global amendment, Version 3.0, 20 July 2020 |
| Version History | Date and version changed; brief summary of omendment added. |
| Clinical Study Protocol Synopsis | Updated the estimated date of last subject completed from Q3 2020 to Q3 2021. |
| 1.3 Benefit/risk and etheral assessment | Added justification to continue study enrollment and treatment during the COVID-19 pandemic. |
| 1.5.2 Adjudication committee | Clarification that the committee will adjudicate "after medical monitoring review." |
| 2.2 Secondary Objective and<br>Clinical Study Protocol Synopsis | Updated a secondary endpoint to total "systemic" corticosteroid exposure over the treatment period. |
| 2 Exploratory Objective<br>Clinical Study Protocol Synopsis | Addition of 2 additional exploratory endpoints: |

| Section | Changes made to Version 2.0, 29 July 2019 to |
|---|---|
| | develop global amendment, Version 3.0, |
| | 21 July 2020 |
| | 21 July 2020 |
| | ACQ-5 change from baseline and responder (3-factor) analysis at Week 12 and Week 24 Inhaled corticosteroid exposure over the treatment |
| | period |
| 3.1 Inclusion criteria (item 2) and | Removed the inclusion of children ≥6 years of age in |
| Clinical Study Protocol Synopsis | Italy. |
| | Removed the inclusion of adolescent subjects ≥12 years of age in Spain. |
| | of age in Spain. |
| 3.1 Inclusion criteria (item 4) | Clarification that subjects on ICS alone or in |
| | combination with LABA are allowed to have additional |
| | maintenance medication; specified leukotriene |
| | "receptor ap agonists" are allowed. |
| | C 8 |
| 3.1 Inclusion criteria (item 5) | Update Oo reflect predicted normal FEV₁ values of ≥40 to <90% for adults and ≥60% for subjects aged 4 to |
| | Specified that subjects 4 to 17 years of age who |
| | reviously failed this inclusion criteria due to the |
| Mag | previous upper FEV <sub>1</sub> limit are permitted to re-screen once. |
| 3.1 Inclusion criteria (iten | Clarification that subjects aged 4 to 11 will be eligible |
| 00 | if they provide 2 acceptable/repeatable measurements |
| 3.1 Inclusion criteria (itent/) | for spirometry. |
| 3.1 Inclusion cris ria (item 17) | Removal of the reference to ≥50 years of age as part of |
| 5 | the definition of menopausal women. |
| 3.2 Exclusion criteria (item 25) | Specification that subjects are excluded if they had |
| 20 | been previously "randomized" in this study or another |
| 3.2 Exclusion criteria (item 25) | PT007 or PT027 study. |
| 36 Subject enrollment and | Updated the number of subjects screened from 4300 to |
| Candomization and Clinical Study | 6000. |
| Protocol Synopsis | |
| <u> </u> | |

|---|---|
| Section | |
| | develop global amendment, Version 3.0, |
| | 21 July 2020 |
| 3.5 Methods for assigning | Removed reference to screening Visit 1a. Added |
| treatment groups, 7.2 Dose and | clarification that randomization stratification will |
| treatment regimens, and Clinical | include the number of prior severe exacerbations (1, |
| Study Protocol Synopsis | >1) in the 12 months prior to screening (Visit ) "plus |
| | any severe exacerbation event experienced during the |
| | screening period." |
| 2.7 | |
| 3.11 Screen failures | Modification to allow for rescreening once in children |
| | and adolescents who failed because they did not meet |
| | the now obsolete upper FEV <sub>1</sub> opredicted limit. |
| 4 Study plan and timing of | Footnote f and applicable X" indicators were removed |
| procedures (Table 1) | due to country specific changes. Subsequent footnote |
| procedures (Table 1) | marker letters were applated. |
| | marker reners were appeared. |
| | Footnote in precedusly footnote i) was updated to |
| | remove Talk and add Argentina as requiring additional |
| | pregnancy testing. |
| | 2/2°0. |
| | cotroite m (previously footnote n) updated to reflect |
| | presicted normal FEV₁ values of ≥40 to <90% for |
| | aults and ≥60% for subjects aged 4 to 17. |
| 4.1 Semaning and min in pariod | Italy-specific information regarding full examinations |
| 4.1 Screening and run-in period 4.2 Randomization/ treatment | and pregnancy testing was removed. |
| period/extension phase, and | and pregnancy testing was removed. |
| 5.3.1 Physical examination | |
| 5.5.1 Filysical examination | |
| 5.1.8.2 COVID-19-Qnd | Addition to specify that spirometry should not be done |
| Pulmonary Function Testing | if subjects are showing signs and symptoms of |
| 235 | COVID-19 and to indicate that participants with |
| 700 | suspected COVID-19 should receive a test to confirm |
| 1,40 | diagnosis. Proper cleaning and hygiene guidance is to |
| Pulmonary Function Testing | be followed. |
| * | |
| Σ.1 Laboratory safety | Removed Italy and added "Argentina" to footnote a |
| assessments (Table 2) | (pregnancy testing requirements). |

|---|---|
| Section | develop global amendment, Version 3.0, |
| | 21 July 2020 |
| | 21 July 2020 |
| 5.3.2 Concomitant medications | Updated to indicate that previous medications should |
| | be recorded if they were taken within 3 months before |
| | screening. Added that asthma medication history will |
| | be recorded for 12 months before screening. |
| 6.3.9 COVID-19 Adverse Events | Added to provide instructions on how to manage AEs |
| | and SAEs related to the COVID-19 pandemic. |
| 7.8.1 Maintenance therapies | Addition to allow subjects receiving maintenance |
| | allergy immunotherapy (AIT) to continue their AIT. |
| | Specified that the initiation of AIT during the study is |
| | not allowed. |
| 702P-1114-111-4 | io <sup>t</sup> |
| 7.8.3 Prohibited medications | Clarification that polyclonal antibody therapy is |
| | prohibited by the use of intra-ocular monoclonal or |
| | polyclonaCantibody therapy is allowed. |
| | Clarification that the use of specific cardio-selective |
| | beta blockers in low daily doses, eg, metoprolol in |
| | allowed. |
| 8.1.2 Type 1 error control and | Actied information about hierarchical testing |
| Clinical Study Protocol Synopsis | procedures to control the type-1 error in secondary |
| 3 | endpoint analyses. Details regarding testing procedures, |
| 100 | the order of testing for secondary endpoints, and when |
| , of s | statistical significance can be claimed, are provided. |
| 8.3.1 Full analysis set | Clarification that the effectiveness estimand will utilize |
| , JQY | all observed data up to randomized treatment |
| l vos | discontinuation, regardless of whether subjects |
| , <u>`</u> | experience a change in maintenance therapy for lack of |
| Je | asthma control. Added that the de facto estimand will |
| , 2° | utilize all observed data, including post-IP |
| Ko. | discontinuation data, regardless of a change in |
| 8.3.1 Full analysis set 8.3.1 Full analysis set 8.3.1 Full analysis set 8.3.2 Derivation of annualized | maintenance therapy. |
| 8.2.1 Derivation of annualized | Updated the calculations of follow-up and IP |
| Severe asthma exacerbation rate | discontinuation/change in maintenance therapy to |
| | 1 |

|---|---|
| Section | develop global amendment, Version 3.0, |
| | , , |
| | 21 July 2020 |
| | exclude the cumulative duration of severe |
| | exclude the cumulative duration of severe exacerbation(s). Updated headings with "systemic" and replaced previous text regarding inhaled corticosteroid exposure. Specified methods to calculate and analyze total SCS exposure. |
| 8.5.2.2 Derivation of total | Updated headings with "systemic" and replace |
| systemic corticosteroid exposure, | previous text regarding inhaled corticoster exposure. |
| 8.6.2.4 Total systemic | Specified methods to calculate and analyze total SCS |
| corticosteroid exposure, and | exposure. |
| Clinical Study Protocol Synopsis | aitaito |
| 8.5.2.3 Derivation of Asthma | Definition added for 3-level factor categorization |
| Control Questionnaire-5 variables | (Improvement, No Change, and Worsening) for |
| | changes from baseline in the ACQ-5 overall scores at |
| | Weeks 12 and 24. |
| | √ .د∜ |
| 8.5.3.5 Total inhaled | Addition of ections to specify methods used to |
| corticosteroid exposure and | calculate and analyze total inhaled corticosteroid |
| 8.6.4.7 Total inhaled | exposure (C) |
| corticosteroid exposure | calculate and analyze total inhaled corticosteroid exposure in a superior control of the corticosteroid exposure in a superior control of |
| 8.6 Methods for statistical | Removed reference to "2" primary comparisons and |
| analyses | regueced with primary "endpoint treatment" |
| | comparisons. |
| 8.6.1 Analysis of the primary | Specification that analyses would target the efficacy |
| variable | estimand in the FAS population. |
| 2001 | Added statement that all subjects who are randomized |
| ank. | and are part of the full analysis set will be analyzed |
| , w° | according to the strata they were allocated to in |
| Į "Š | IVRS/IWRS. A sensitivity analysis will be conducted |
| J.S | based on subjects' actual strata to assess the impact of |
| variable used to support and | miss-stratification on the model results. |
| 8.6.1 analysis of the primary | Specified that the models for analyses of variables |
| varable, 8.6.2.2 Asthma Control | would be adjusted for the number of prior severe |
| Questionnaire-5, 8.6.4.2 | exacerbations (1, >1) in the 12 months prior to |
| Prebronchodilator FEV1, and | screening (Visit 1) "plus any severe exacerbation event |
| 8.6.4.3 Morning peak expiratory | |

|---|---|
| Section | develop global amendment, Version 3.0, |
| | , , |
| | 21 July 2020 |
| flow, and Clinical Study Protocol | experienced during the screening period", and remove references to Visit 1a. |
| Synopsis | references to Visit 1a |
| Syllopsis | references to visit 1a. |
| 8.6.2 Analysis of the secondary | Specified that analyses would be conducted on the FAS |
| efficacy variables | population. |
| | Referenced Section 8.1.2 for hierarchical testing |
| | strategy for secondary endpoints. |
| | ai <sup>©</sup> |
| 8.6.2.1 Severe asthma | Specification that analyses would target the efficacy |
| exacerbation rate | estimand in the FAS population. |
| | The number of prior severe exacerbations in the |
| | 12 months prior to "randomization" was updated as a |
| | key covariate of interest. |
| | 0, 2, |
| 8.6.2.2 Asthma Control | Addition of information for analysis of the 3-factor |
| Questionnaire-5 | categorization of ACQ-5 using ordinal logistical |
| | regression. |
| | ED JE |
| • | Specification that the analysis of change from baseline |
| | mACQ-5 at Week 24 will target the efficacy estimand |
| , de | th the FAS population. |
| 8.6.2.2 Asthma Control | Updated methods of analysis from MMRM to repeated |
| Questionnaire-5 and 8.6.2.30 Asthma Quality of Life | measures analyses. |
| Asthma Quality of Life | |
| Questionnaire +12 and Pediatric | |
| Asthma Quality of bife | |
| Questionnaire | |
| 8.6.4.3 Mortang peak expiratory | Addition of a repeated measures analysis of 4-weekly |
| flow No. | time intervals. |
| 8.6. Frimary outcome analysis | Removed "and final analysis" from heading. |

|---|---|
| | develop global amendment, Version 3.0, |
| | 21 July 2020 |
| | , |
| | Clarification of the following: when subjects will return |
| | for their EOS visits, when data cleaning should be |
| | done, and when the primary (final) analysis will occur. |
| 8.6.7.5 COVID-19 pandemic | Addition to describe statistical methods that will be |
| impacts | used to evaluate the impact of the COVID 219 pandemic |
| | on efficacy and safety variables. |
| 11 List of References | Addition of reference to the American Academy of |
| | Allergy Asthma and Immunology for information |
| | regarding COVID-19 and Ashma. |
| | 8 |
| | For Investigator Brochuse reference, updated edition |
| | and date. |
| Appendix N, COVID-19 | Addition of processes to ensure subject safety during |
| emergency measures permitted to | the COVOD-10 pandemic. Instructions for management |
| ensure subject safety | of subjects with or suspected COVID-19 infection, |
| | delayed orisits, remote visits, subject discontinuation, |
| | shipment of IP to subjects, laboratory testing, and |
| • | spinometry testing are provided. |
| Throughout document | Updated study drug to "IP" for consistency. |
| <i>'</i> !%. | Additional nonsubstantial changes for administrative, |
| *** | typographical, and/or grammatical corrections were |
| Throughout document | made. |

# 12.3 Changes made to Version 1.0

| Section A D | Changes made to Version 1.0, 11 Oct 2018 to<br>develop global amendment, Version 2.0, 29 July<br>2019 |
|---|---|
| Sersion History | Date and version changed, brief summary of amendment added. |

| Clinical Study Protocol Synopsis, | Updated the number of study sites/centers from 333 to |
|---|---|
| 1.4 Study design, 3.3 Subject | 380 and an estimated screen failure rate to a range of |
| enrollment and randomization, 4 | 30% to 50%. |
| | 30% 10 30%. |
| Study plan and timing of | Clarification on the timeframe (Visit 1 and Visit 1a) |
| procedures (footnote b in Table | and possible extension of the screening period due |
| 1), 4.1 Screening and run-in | administrative reasons or a severe asthma exacersation |
| period | event (to a maximum of 9 weeks). |
| | event (to a manimum of 5 weeks). |
| | Clarification on the use of patients' usual &-needed |
| | (prn) inhaled products and Sponsor-provided Ventolin |
| | (prn or prior to exercise) during screening. |
| | aiio |
| | Addition of the de facto estimand as a treatment policy |
| | strategy defined in the draft atternational Conference |
| | on Harmonization (ICH) 🔊 addendum. |
| 17.4.1.6 | |
| 1 Introduction | Statement clarifying that albuterol is also known under |
| | the generic name of salbutamol (the international non- |
| | proprietary name): |
| 1.2 Rationale for study design, | Provided justification of the proposed doses for |
| doses, and control groups | albateroband budesonide based on the approved label |
| , | Proventil and the dose-ranging Study PT008001 |
| • | respectively. |
| | & |
| Clinical Study Protocol Synopsis | Clarification of the maximum daily dosing recommendation for subjects and notification/eDiary |
| 1.4 Study design, 5.1.1.6.2 | recommendation for subjects and notification/eDiary |
| Symptom Reporting, 6.5 | alert to medical monitors and investigators of any |
| Overdose, and 7.2 Dose and | increased IP dosage in order to closely monitor |
| treatment regimens | treatment use with potential worsening asthma status. |
| Sy. | |
| 1.5.2 Adjudication committee | Clarification on adjudication committee events- |
| l & | recording and case definition of "worsening of asthma" |
| _ & ~ | which would necessitate adjudication committee |
| 1.5.2 Adjudication committee | review. |
| Clinical Study Protocol Synopsis<br>and 3.1 Inclusion criteria (item 2) | Specifying the inclusion of subjects 4 years of age in all |
| and 1 Inclusion criteria (item 2) | countries with the exception of Italy, Serbia, Spain, |
| ST. | Germany, Slovakia, and Ukraine. |
| £. | |

| | Specifying the inclusion of children ≥6 years of age |
|---|---|
| | only in Italy. |
| | only in runy. |
| | Specifying the inclusion of adolescent subjects ≥12 |
| | years of age only in Serbia and Spain. |
| | Specifying the inclusion of adult subjects ≥18 years of |
| | age only in Germany, Slovakia, and Ukraine. |
| | age only in definally, Stovakia, and Oktaine. |
| 3.1 Inclusion criteria (item 4) | Additional clarification that up to 20% of |
| | randomized patients will be permitted to have an |
| | additional maintenance medication (Meophylline, |
| | leukotriene, or LAMA, in addition to either ICS alone |
| | or ICS/LABA fixed dose combination). |
| | and the same of th |
| 3.1 Inclusion criteria (item 5) | Clarification that if FEV <sub>1</sub> salues are not within the |
| | permitted range at Visit 1, 1 re-test is required at Visit |
| | 1a before advancing Wisit 2 or being considered as a |
| | screen failure |
| 217.1 | C 8 |
| 3.1 Inclusion criteria (item 6) | Clarification that if reversibility is not demonstrated at |
| | Visit 1 rectest for reversibility testing is required at |
| | Visit lamefore advancing to Visit 2 or being considered |
| | a so een failure |
| 2.1 Inclusion oritorio (itam 12) | Additional appointment that the year of appears are |
| 3.1 Inclusion criteria (item 12) | additional specification that the use of spacers are |
| , to | prohibited. |
| 3.1 Inclusion criteria (items 18) | Addition of definition of complete abstinence (and that |
| and 18) | is an acceptable method of contraception only if it is |
| , sol | consistent with the preferred and usual lifestyle of the |
| , July | subject); definition of double-barrier birth control; |
| , o <sup>o</sup> | clarification on surgical sterility by vasectomy (for |
| ్డ్ | males); definition of postmenopausal status; addition of |
| JE | bilateral salpingectomy to the definition of surgical |
| , <b>%</b> | sterility; and clarification that contraceptive methods |
| and 18) and the used to support must not be used to support number of the used to support numbe | may only be recommended for adolescents who are |
| <u>\$</u> | already sexually active, and that the use of hormonal |
| King. | contraceptives must always be in consultation with a |
| at . | |
| K. | gynecologist (for females). |
| t | |

| 3.2 Exclusion criteria (item 1) | Additional specification regarding regular or occasional |
|---|---|
| 3.2 Excitation criteria (item 1) | use of oxygen. |
| | use of oxygen. |
| 3.2. Exclusion criteria (item 4) | Addition of dupilumab as an example of prohibited |
| | medication. |
| | X8" |
| 3.2 Exclusion criteria (item 21) | Additional specification that currently pregnant females |
| | will also be excluded from study participation |
| | <b>\$</b> Ø` |
| 3.2. Exclusion criteria (new item | Addition of new exclusion criterion #26: |
| 26) | experience >1 asthma exacerbation during the |
| | screening period. |
| 27364-1-611-1- | Children in the little in the little in the |
| 3.7 Methods for unblinding | Clarification that unblinding should be based on the |
| | investigator's clinical judgment (when the appropriate |
| | management and welfare of the subject requires |
| | knowledge of the treatment allocation) and that it is not |
| | required, for the investigator to inform the Sponsor or |
| | Sponsor's designed before unblinding. |
| 3.8 Restrictions | Addition of depilumab as an example of prohibited |
| | medicanon and other investigational treatments (other |
| | that the study drugs). |
| | 47.5 |
| 3.9 Treatment discontinuation by | Clarification that in case of elevated liver enzymes AST |
| subject and/or Sponsor, 6.3.8 | or ALT ≥3×ULN and total bilirubin ≥2×ULN, the |
| Hy's Law, and Appendix E Hy's | use of the IP will be suspended until the liver test values return to the normal range, and that if the liver |
| Law | 3, |
| A. C. | enzyme values become elevated again after the |
| - K | recommencement of the IP, the subject will be |
| support of ' | discontinued from IP and withdrawn from the study. |
| 9 | 4.11% 1.1.% (C.1.1) |
| 3.9 Treatment discontinuation by | Additional clarification on PDV procedures (including |
| subject and/or Sponsor, 4 Study | potential follow-up TC) for subjects who discontinue |
| plan and timing of procedures | treatment prior to EOS for any reason, and if the PDV |
| (footnote on Table 1), 4.6 | is performed at least 14 days after the last study drug |
| Follow-op | dose. |
| 4 Study plan and timing of | Additional assessments applicable to Italy ONLY; in |
| procedures (footnote f and i in | Italy, a full physical examination will be performed at |
| Table 1), 4.1 Screening and run- | all visits with additional pregnancy testing to be |
| in period, 4.2 Screening and | |
| annullment paried 5.2.1 | conducted at monthly time points in women of |
|---|---|
| enrollment period, 5.2.1 | , <u>.</u> |
| Laboratory safety assessments | childbearing potential. |
| (Table 2 notes), 5.3.1 Physical | |
| examination | 8 |
| 1.3 Benefit/risk and ethical | Addition of height assessments for all subjects at 🖎 |
| assessment, 4 Study plan and | and additional height assessments for subjects ≤\\$ |
| timing of procedures (footnote g | years of age. Additional morning serum cortises |
| | 0. |
| in Table 1), 4.1 Screening and | assessments for all subjects at specified visits |
| enrollment period, 4.2 | (Screening, Week 24, EOS and PDV). Clarification that |
| Randomization/treatment | assessments of height will continue in accordance with |
| period/extension phase, 4.3 End- | a subject's age at the time of signed informed |
| of-study visit, 4.4 Unscheduled | consent/assent. |
| visit and premature | la l |
| discontinuation visit, 5.2 Safety | Addition of urine pregnancy assessments to safety |
| assessments, 5.2.1 Laboratory | <u>~</u> |
| safety assessments (Table 2), | , dillo |
| 5.3.1 Physical examination and | 04 911Cr |
| 8.6.3.3 Clinical chemistry and | رن <i>ه</i> ر |
| hematology | 0.0 |
| | W. S. |
| 4 Study plan and timing of | Addition of urine pregnancy assessments to safety |
| procedures (footnote i in Table 1) | O' STATE OF THE ST |
| and 5.2.1 Laboratory safety | throughout the duration of the study (unless otherwise |
| assessments (Table 2) | specified). |
| 4 Study plan and timing of | Clarification on time points for dispensing and |
| procedures | collection of eDiary. |
| 4 Study plan and timing & | Addition of dispensing Ventolin at V1. |
| procedures S | Addition of dispensing ventorin at v1. |
| procedures | |
| 5.1.1 Asthma exaserbation | Clarification of deterioration of lung function with |
| 5.1.1 Asthma exacerbation definition | examples for clarity and consistency. |
| e~ | |
| 5.1.1.5 Onset and duration of | Distinction on reporting severe asthma exacerbations as |
| asthma exacerbations | separate or singular events, based on successive SCS |
| asthma exacerbations | use within 7 days (or more). |
| N. Control of the control of the con | |
| №1.1.6.1 Severe asthma | Clarification on the appropriate reporting of severe |
| exacerbation eCRF | asthma exacerbations during the screening period. |

| 5.1.1.6.2 Symptom reporting | Clarification on the appropriate reporting of asthma |
|---|---|
| | signs or symptoms. |
| 5.5.5.5.1.1.0.11.0.710 | |
| 5.1.2.1 Asthma Quality of Life | Clarification that the AQLQ+12 will be used in subjects |
| Questionnaire+12 | 12 years and older. |
| 51000 11111 1111 1111 | Clair dad Backs 311 Is 1 is 1 |
| 5.1.2.2 Pediatric Asthma Quality | Clarification that the PAQLQ will be self-administered in subjects aged 7 to 11 years. |
| of Life Questionnaire | w <sup>*</sup> |
| 5.1.8.1 Reversibility Test | Clarification that prebronchodilator PFTs hould be |
| | performed after at least 15 minutes of rest, and before |
| | administration of Ventolin. |
| | illo |
| | Removed wording that the confirmation of the FEV <sub>1</sub> |
| | measurements should be entered into the eCRF to |
| | confirm eligibility. Other san overall eligibility |
| | confirmation, there is no specific confirmation relating |
| | to this (other than overall eligibility confirmation). |
| 5.2.3 Vital sign measurements | Correction of blood pressure measurement to be taken |
| and 8.6.3.2 Vital signs | in the seated position (and not supine). |
| and 0.0.3.2 Vital signs | in the state of position (and not supine). |
| 5.3.2 Concomitant medications | Upgate es timeframe for concomitant medications to |
| | include those taken beginning within 12 months before |
| | Screening. |
| | in |
| 6.4 Reporting of serious adverse | Provision of additional reporting responsibility of |
| events | Sponsor for serious unexpected adverse drug reactions |
| 3 | related to IP. |
| ~** | |
| 6.5 Overdose, 6.7 Medication error | Clarification on the appropriate |
| error JQ* | collection/recording/reporting of an |
| , o° | Overdose/Medication Error with or without an |
| ر م | associated AE/SAE. |
| JSE . | |
| 7.8.1 Maintenance therapies and | Modification to remove the advance notification for |
| 7.8.2 Medications that may affect | investigators to notify the Sponsor with regards to any |
| reversibility and FEV1 testing | proposed maintenance therapy changes. |
| 7.3.3 Prohibited medications | Clarification/correction that inhaled short-acting |
| Ke. | anticholinergies (or short-acting muscarinic antagonists |
| 7 | [SAMA]). |

| | | Additional clarification that inhaled long-acting |
|---|---|---|
| | | anticholinergics (or LAMA), except those that were |
| | | started before screening and continued as part of |
| | | maintenance treatment are prohibited. |
| | | , gyb |
| | | Correction to reflect that nonglucocorticoid nasal |
| | | Sprays are not prohibited. |
| | Clinical Study Protocol Synopsis, | Addition of the de facto estimand as a treatment policy |
| | 8.1.1 Estimands and 8.6.7.4 De | strategy defined in the draft ICH E9 adderedum and |
| | facto estimand | specification of population analyses. |
| | | ijO <sup>1</sup> |
| | 8.5.2.2 Derivation of total | Change in how ICS and SCS are to be analyzed: ICS to |
| | corticosteroid exposure, 8.6.2.4 | be summarized as a mean daily dose; SCS to be |
| | Total corticosteroid exposure | summarized by duration of administration. |
| | Appendix D, Additional safety | Adjustment to reflect resorting investigators are highly |
| | information | encouraged to express their clinical opinion when |
| | | presented with limited or insufficient information in the |
| | | causality assessments. Further, that if the causality |
| | | assessment connot be made, these serious adverse |
| | | events with be considered to be "related". |
| | Appendix F Asthma Quality of | Applaced to April 2008 version. |
| | Life +12 Questionnaire | einos |
| | Appendix G Pediatric Asthma | Updated to January 2001 version. |
| | Quality of Life Questionnaire | |
| | ·ka | |
| | Appendix H Asthma Control | Updated to December 2002 version (and July 2011 |
| | Questionnaire-5 and -7 | version of the Interviewer-administered ACQ). |
| | Throughout document | Nonsubstantial changes for administrative, |
| | Throughout document | typographical and/or grammatical corrections. |
| | , CO | |
| | a no | |
| | Alias | |
| | al. | |
| | The | |
| . 6 | 33 | |
| ىم. | | |
| THE | | |
| • | | 111 of 159 |

Clinical Study Protocol, Version 4.0 Budesonide/albuterol (BDA) - AV003

# APPENDIX A, AVILLION PROTOCOL SIGNATURE PAGE

Avillion Signature Form for the Clinical Study Protocol

We, the undersigned, to the best of our knowledge and ability attest to the accuracy and validity of the contents of the Clinical Study Protocol.

of such application The double of the state of the



# APPENDIX C, GLOBAL INITIATIVE FOR ASTHMA (GINA, 2018)

The table below is not a table of equivalence, but of estimated clinical comparability. Categories of low, medium, and high doses are based on published information and available studies, including direct comparisons where applicable. Doses may be country-specific depending on labelling requirements, drug formulation, or inhalation device. Most of the clinical benefit from ICS is seen at low doses, and clear evidence of dose-response relationships is seldom available within dose ranges evaluated for regulatory purpose. High doses are arbitrary, but for most ICSs are those that, with prolonged use, are associated with increased risk of systemic side-effects.

The below defines the minimally acceptable documentation for inclusion. Scriteria:

- Signed and dated notes from a referring physician, including name and dose of the ICS/ICS/LABA inhaler (or names and doses, if used as separate inhalers).
- 2 Evidence of prescriptions for ICS/LABA medications that demonstrate coverage for the duration specified in inclusion criteria.

Low, Medium, and High Doses of Inhaled Corticosteroids

| Adults and advices (12 years and older) | | | |
|---|---|---|---|
| | ~~ Daliv | dosage (μg) | |
| DRUG | > rom | MEDIUM | HIGH |
| DRUG Beclometasone dipropionate (CFC) <sup>a</sup> | 200-500 | >500-1000 | >1000 |
| Beclometasone dipropionate (HF | 100-200 | >200-400 | >400 |
| Budesonide (DPI) | 200-400 | >400-800 | >800 |
| Ciclesonide (HFAX | 80-160 | >160-320 | >320 |
| Fluticasone furoate (DPI) | 100 | NA | 200 |
| Fluticasone propionate (DPI) | 100-250 | >250-500 | >500 |
| Fluticasone popionate (HFA) | 100-250 | >250-500 | >500 |
| Mone asone furoate | 110-220 | >220-440 | >440 |
| Trisacinolone acetonide | 400-1000 | >1000-2000 | >2000 |
| , 10° ci | nildren 6-11 years | | |
| Bestometasone dipropionate (CFC) <sup>a</sup> | 100-200 | >200-400 | >400 |
| Bestometasone dipropionate (CFC)* Beclometasone dipropionate (HFA) Budesonide (DPI) | 50-100 | >100-200 | >200 |
| Budesonide (DPI) | 100-200 | >200-400 | >400 |
| Budesonide (nebules) | 250-500 | >500-1000 | >1000 |

| Ciclesonide | 80 | >80-160 | >160 |
|------------------------------|---------|-----------|----------|
| Fluticasone furoate (DPI) | NA | NA | NA |
| Fluticasone propionate (DPI) | 100-200 | >200-400 | >400 |
| Fluticasone propionate (HFA) | 100-200 | >200-500 | >500 💍 |
| Mometasone furoate | 110 | ≥220-<440 | ≥440 ير% |
| Triamcinolone acetonide | 400-800 | >800-1200 | >1200 |

Abbreviations: CFC=chlorofluorocarbon propellant; DPI=dry powder inhaler; HFA=hydrofluoroalk the propellant; NA=not applicable

| Abbreviations: CFC=chlorofluorocarbon propellan propellant; NA=not applicable Beclometasone dipropionate CFC is included | If; DPI=dry powder inhaler; HFA=hydrofluoroallerae |
|---|---|
| Low Daily Doses of Inhaled Corticoster | oids for Children 5 Years aid Younger |
| DRUG | Low daily dosage (µg) <sup>a</sup><br>(age group with adequate safety and effective data) |
| Beclometasone dipropionate (HFA) | . 600 (ages ≥5 years) |
| Budesonide nebulized | ر 300 (ages ≥1 year) |
| Fluticasone propionate (HFA) | 100 (ages ≥4 years) |
| Mometasone furoate Budesonide pMDI + spacer Ciclesonide Triamcinolone acetonide Abbreviations: HFA=hydrofluoroalkane propelling | 110 (ages ≥4 years) |
| Budesonide pMDI + spacer | Not sufficiently studied in this age group |
| Ciclesonide | Not sufficiently studied in this age group |
| Triamcinolone acetonide | Not sufficiently studied in this age group |
| Subjects 5 years and younger meeting GNA or Low dose ICS + LTRA (Global Indicative for Low dose ICS + LTRA) (Global Indicative for LTRA) (Glob | |
| | 115 of 159 |

### APPENDIX D, ADDITIONAL SAFETY INFORMATION

Further guidance on the definition of a serious adverse event (SAE)

## Life -threatening

"Life -threatening" means that the subject was at immediate risk of death from the AE as it occurred or it is suspected that use or continued use of the product would result in this subject's death. "Life-threatening" does not mean that an AE occurred in a more evere form, it might have caused death (eg, hepatitis that resolved without hepatic failure).

## Hospitalization

Outpatient treatment in an emergency room is not in itself a serious AE, although the reasons for it may be (eg, bronchospasm, laryngeal edema). Hospital admissions and/or surgical operations planned before or during a study are not considered AEs if the illness or disease existed before the subject was enrolled in the study, provide that it did not deteriorate in an unexpected way during the study.

# Important medical event or medical intercention

Medical and scientific judgment should be exercised in deciding whether a case is serious in situations where important medical events thay not be immediately life-threatening or result in death, hospitalization, disability, or incapacity, but may jeopardize the subject or may require medical intervention to prevent 1 or more outcomes listed in the definition of serious. These should usually be considered as serious.

Simply stopping the suspect drug does not mean that it is an important medical event; medical judgment must be used. Examples of important medical events include but are not limited to:

- Angioedema not Severe enough to require intubation but requiring intravenous hydrocortisone treatment.
- Hepatotossicity caused by paracetamol (acetaminophen) overdose requiring treatment with N acetylcysteine.
- Intensive treatment in an emergency room or at home for allergic bronchospasm.
- Solood dyscrasias (eg, neutropenia or anemia requiring blood transfusion, etc.) or convulsions that do not result in hospitalization.
- Development of drug dependency or drug abuse.

Chip

## A guide to interpreting the causality question

When making an assessment of causality, consider the following factors when deciding if there is a "reasonable possibility" that an AE may have been caused by the drug:

- Time Course. Exposure to suspect drug. Has the subject actually received the suspect drug? Did the AE occur in a reasonable temporal relationship to the administration of the suspect drug?
- Consistency with known drug profile. Was the AE consistent with the presous knowledge of the suspect drug (pharmacology and toxicology) or drugs of the same pharmacological class? Or could the AE be anticipated from its pharmacological properties?
- De-challenge experience. Did the AE resolve or improve on supping or reducing the dose of the suspect drug?
- No alternative cause. The AE cannot be reasonably explained by another cause such as the underlying disease, other drugs, and other host open vironmental factors.
- Re-challenge experience. Did the AE reoccor if the suspected drug was reintroduced
  after having been stopped? The Sponsor would not normally recommend or support a
  rechallenge.
- Laboratory tests. A specific laboratory investigation (if performed) has confirmed the relationship.

In difficult cases, other factors could considered such as:

- Is this a recognized feature of overdose of the drug?
- Is there a known mechanism?

Causality of "related" is made if after a review of the relevant data there is evidence for a "reasonable possibility" of a causal relationship for the individual case. The expression "reasonable possibility" of a causal relationship is meant to convey, in general, that there are facts (evidence) or arguments to suggest a causal relationship.

The causality assessment is performed on the basis of the available data, including enough information to make an informed judgment. With limited or insufficient information in the case, it is highly encouraged for the reporting investigator to express his/her clinical opinion. (despite all efforts) the causality assessment cannot be made, these SAEs will be considered to be "related".

ack of ac

This Appendix describes the process to be followed to identify and appropriately report cases of Hy's Law (HL). It is not intended to be a comprehensive guide to the management cases elevated liver biochemistries.

biochemistry. In subjects who have elevated liver enzymes aspartate aminotratisferase (AST) and/or alanine transaminase (ALT) ≥ 3×ULN and total bilirubin (TBL) ≥ 25 ULN, IP will be suspended until the liver test values return to the normal range. If the ASSE, ALT or TBL reach these elevated levels again, after recommencement of IP, the subject will be discontinued from IP and withdrawn from the study. The investigator is responsible for determining whether a subject meets Potential Hy's Law (PHL) criteria at any point during the study.

The investigator participates, with the Sponsor's clinical project representatives, in review and assessment of cases meeting PHL criteria to agree whether HL criteria are met. Hy's Law criteria are met if there is no alternative explanation for the elevations in liver biochemistry other than drug induced liver injury caused by the IR.

The investigator is responsible for recording data pertaining to potential HL/HL cases and for reporting AE and SAE according to the outcome of the review and assessment in line with standard safety reporting processes. Q

### Definitions

### Potential Hy's Law

AST and/or ALT  $\ge 3 \times$  ULX combined with TBL  $\ge 2 \times$  ULN at any point during the study after the start of IP irrespective of an increase in alkaline phosphatase (ALP).

### Hy's Law

AST and/or AL⊅≥3×ULN combined with TBL ≥2×ULN, where no other reason, other than the IP, can be found to explain the combination of increases, eg, elevated ALP indicating cholestasic viral hepatitis, or another drug.

use same day) the elevation in TBL, but there is elevations in transaminases and TBL must occur. For potential HL and HL, the elevation in transaminases must precede or be coincident with (ie on the same day) the elevation in TBL, but there is no specified timeframe within which

To identify cases of PHL it is important to perform a comprehensive review of laboratory data and for any subject who meets any of the following identification criteria in isolation or in combination:

• ALT ≥3×ULN
• AST ≥3×ULN
• TBL ≥2×ULN

When a subject meets any of the identification criteria, in isolation or in continuous central laboratory will immediately send on all the significant of the identification criteria, in isolation or in continuous central laboratory will immediately send on all the inspiratory will be inspiratory w assigned to the project.

The investigator will also remain vigilant for any local laboratory reports where the identification criteria are met; where this is the case, the investigator will:

- Notify the medical monitor assigned to the project
- Request a repeat of the test (new blood traw) by the central laboratory.
- Contact the medical monitor to discuss the elevated local labs and whether these constitute an AE. Where an AE is entered due to elevations of local labs, the AE will be queried in the eCRF and elevated local lab values, units and ranges will be entered to the query response.
- When the identification criteria are met from central or local laboratory results, the investigator will without delay:
  - Determine whether the subject meets PHL criteria by reviewing laboratory reports from all previous visits (including both central and local laboratory
- The investigator will, without delay, review each new laboratory report and if the identification criteria are met, will:
  - Notify the medical monitor assigned to the project.
    - Determine whether the subject meets PHL criteria by reviewing laboratory reports from all previous visits.
  - Promptly enter the laboratory data into the laboratory eCRF.

Follow-up

Inform the medical monitor assigned to the project that the subject has not met PHL criteria. Perform follow-up on subsequent laboratory results according to the guidance. Clinical Study Protocol. Perform follow-up on subsequent laboratory results according to the guidance provided in the Clinical Study Protocol.

Potential Hy's Law criteria met

If the subject does meet PHL criteria, the investigator will:

Determine whether PHL criteria were met at any study visit before starting IP (See section below on "Actions required when Potential Hy's Law criteria are met before and after starting IP")

Notify the medical monitor assigned to the project who will then inform the central study team

The medical monitor assigned to the project will discuss the issue with the investigator to provide guidance, and agree an approach for the stody sobjects' follow-up and the continuous review of data. Subsequent to this contact the investigator will:

Monitor the subject until liver biochemistry parameters and appropriate clinical symptoms and signs return to normal or baseline levels or as ong as medically indicated

Investigate the cause of the event and serform diagnostic investigations as discussed with the medical monitor assigned to the project Por studies using a central laboratory add: This includes deciding which the tests available in the Hy's Law lab kit should be used.

Complete the 3 Liver eCRF modeles as information becomes available

If at any time (in consultation with the medical monitor assigned to the project) the PHL case meets serious criteria, report it as an SAE using standard reporting procedures.

# Review and assessment of Potential Hy's Law cases

No later than 3 Neeks after the biochemistry abnormality was initially detected, the medical monitor assigned to the project contacts the investigator to review available data and agree on whether there is an alternative explanation for meeting PHL criteria other than drug induced liver in any caused by the IP. The medical monitor assigned to the project and global safety physician will also be involved in this review with other subject matter experts, as appropriate.

instructions below. cording to the outcome of the review and assessment, the investigator will follow the If there is an agreed alternative explanation for the ALT or AST and TBL elevations, a determination of whether the alternative explanation is an AE will be made and subsequently whether the AE meets the criteria for an SAE:

If the alternative explanation is **not** an AE, record the alternative explanation on the appropriate eCRF

If the alternative explanation is an AE/SAE, record the AE/SAE in the eCRF accordingly and follow the Sponsor's standard processes

If it is agreed that there is **no** explanation that would explain the ALT or AST and TBL elevations other than the IP:

Report an SAE (report term "Hy's Law") according to the Sponsor's standard processes.

The "Medically Important" serious criterion should be used if no other serious criteria apply.

As there is no alternative explanation for the HL case, a causality assessment of "related" should be assigned.

If, there is an unavoidable delay, of over 3 weeks, in obtaining the information necessary to assess whether or not the case meets the criteria for HL, then it is assumed that there is no alternative explanation until such time as an informed decision can be made:

Report an SAE (report term "Potential Hy "Law") applying serious criteria and causality assessment as per above

Continue follow-up and review according to agreed plan. Once the necessary supplementary information is obtained, repeat the eview and assessment to determine whether HL criteria are met. Update the SAE report according to the outcome of the review amending the reported term if an alternative explanation for the liver biochemistry elevations is determined.

Actions required when Potential Hy's Law criteria are met before and after starting IP

This section is applicable to subjects who meet PHL criteria on study treatment having previously met PHL criteria at a study visit before starting IP.

At the firston study treatment occurrence of PHL criteria being met the investigator will:

Determine if there has been a significant change in the subjects' condition compared with the last visit where PHL criteria were met

If there is no significant change no action is required.

A "significant" change in the subject's condition refers to a clinically relevant change in any of the individual liver biochemistry parameters (ALT, AST, or TBL) in isolation or in combination, or a clinically relevant change in associated symptoms.

Will inform the process described in the section and process described in the section of the section of this Appendix. uncertainty.

## Actions required for repeat episodes of Potential Hy's Law

This section is applicable when a subject meets PHL criteria on stody treatment and has already met PHL criteria at a previous on study treatment visit. O

The requirement to conduct follow-up, review, and assessment of a repeat occurrence(s) of PHL is based on the nature of the alternative cause identified for the previous occurrence.

The investigator should determine the cause of the revious occurrence of PHL criteria being met and answer the following question met and answer the following question:

Was the alternative cause for the previous socurrence of PHL criteria being met found to be

the disease under study or did the subject meet PHL criteria before starting study treatment and at their first on study treatment visit as described in the section "Actions required when Potential Hy's Law criteria are met effore and after starting IP".

If No: follow the process described in the section "Potential Hy's Law criteria met" of this Appendix.

If Yes: determine if there has been a significant change in the subject's condition compared with when PHL criterfa were previously met

If there is no significant change, no action is required

If there is a significant change:

A "significant" change in the subject's condition refers to a clinically relevant change in any of the adividual liver biochemistry parameters (ALT, AST, or TBL) in isolation or in combination, or a clinically relevant change in associated symptoms. The determination of whether there has been a significant change will be at the discretion of the investigator; this Smay be in consultation with the medical monitor assigned to the project if there is any uncertainty.


## APPENDIX M, SPIROMETRY ASSESSMENT CRITERIA

### Acceptable Versus Usable Tests

Acceptable Tests must meet the following criteria:

- 1. Acceptable start of exhalation with brisk upstroke, no hesitation or false start, and back extrapolation volume <5% of forced vital capacity (FVC) or 0.150 L, which extrapolation volume greater (see example in Figure 1)
- No cough during the first second
- No valsalva maneuver
- No leak
- No obstruction of mouthpiece
- No extra breaths
- 7. Plateau achieved: ie, the volume-time curve shows no change in volume (<0.025 L) for ≥1 second, and the subject has tried to exhale for at least 6 seconds

An acceptable test meets all 7 criteria listed. This to be considered the "gold standard".

Usable spirometry tracings are those that only new criteria 1 and 2. When this occurs, repeat testing up to 8 attempts for pre-dose and 5 attempts for post-dose assessments, in an effort to obtain 3 acceptable spirograms. If only stable lests are obtained, report results based on the 3 best usable trials with observed limitations

Figure 1



The 2 largest values of FVC must be within 0.150 L of each other. The 2 largest values of FEV1 must be within 0.150 L of each other please continue collecting additional spirogrammattempts. The highest FEV1 and the production of the please continue collecting additional spirogrammattempts. The highest FEV1 and the production of the please continue collecting additional spirogrammattempts. The expanded version of the early part of a subject's volume-time spirogram, illustrating back extrapolation through the steepest part of the curve, where flow is PEF rate, to determine the new "time zero". Forced vital capacity -4.291 L; EV - 0.123 L (2.9% FVC): back extrapolation line through PEF.

### Between-Maneuver Reproducibility Criteria

### Pre-dose assessments

After 3 acceptable spirograms have been obtained, apply the following tests:

- The 2 largest values of FVC must be within 0.150 L of each other

If these criteria are met, the spirometry testing for that time point and conclude, however, if possible, please continue collecting additional spirograms to a maximum of 8 pre-dose and 5 post-dose attempts. The highest FEV1 and the highest FVC obtained at each testing time point (even if from different reproducible tracings), will be collected.

If acceptability criteria are not met, continue testine user they are met or the subject cannot/ Post-dose assessments

After 2 acceptable spirograms have been obtained, apply the following tests:

• The 2 largest values of Tive

- The 2 largest values of FVC are within 0.150 L of each other, and/or
- The 2 largest values of FEV are within 0.150 L of each other

If these criteria are met, the sprometry testing for that time point may conclude. The highest FEV<sub>1</sub> and the highest FVC btained at each testing time point (even if from different reproducible tracings), will be collected.

If acceptability/reproducibility criteria are not met, continue testing until they are met or the subject cannot/ sould not continue (maximum of 5 attempts).

The following activities were implemented in order to ensure subject safety during the global lockdown due to the COVID-19 pandemic. While global lockdown restrictions are current. Therefore, necessary are Therefore, necessary emergency measures accepted during the initial global lockdown will be permitted to protect subject safety in the event that infection rates return to levels requiring the return of government or local restrictions on movement of people and goods.

Any procedure performed outside the protocol specified requirements will be documented as a protocol deviation.

<u>Visit Management:</u>

### Visit Management:

# Out of window visits should be considered if it is necessary to **Delayed Visits** safeguard the health of the subject and site staff or enables an on-site subject visit. o If a return to lockdown announced or the site is on lockdown and cannot process a visit, if possible, visits should be rescheduled to carlie later as required to safeguard subjects and Randomzation: If a subject is in screening and cannot complete the randomization visit within 28 days due to local COVE-19 lockdown restrictions, the screening period may be extended to a maximum of 9 weeks. In the event of an extension to the screening period >28 days due to COVID-19. the following safety measurements should be repeated in advance of randomization: safety laboratory assessments, ECG, vital signs, concomitant medications, and medical/surgical history. Visit 6/Week 24: All efforts should be made to complete the associated assessments in the clinic, even if this is visit is delayed. If necessary, while waiting for the time to complete this visit, an unscheduled call and drug dispensing should be done to ensure the subject has sufficient IP during this time.

| Remote Visits | 0 | Where subjects have COVID-19 infection, the site is on lockdown, local restrictions prohibit attendance, or similar, a telephone visit should be completed. All assessments performed should be documented in the same way they would if the visit would have happened on site. |
|---|---|---|
| | 0 | Before a remote visit is performed, verbal consent must be obtained and documented in the subject's medical notes to ensure that the subject understands the implications of continuing in the study when face-to-face visits are temporarily not possible due to COVID-19 restrictions. Where possible, the investigator should ask the subject to confirm their agreement in writing either by email or via a letter. Where multiple inclinic visits will be missed, written consent of the subject will be required. |
| | 0 | If a remote visit is completed; and it is considered appropriate and safe to continue IR, this could be dispatched direct to the subject by courier. |
| | 0 | Randomization visits cannot be conducted remotely and therefore subjects in screening who do not wish to attend an on-site visit should be screen-failed as "withdrawal of consent." |
| | 0 | Remote closeout Visits where necessary for sites that have no enroyed patients. |
| Subject | 0 | Where repeated visits are likely to be missed, the site should |
| Discontinuation | ٨ | discuss with the subject and consider ongoing treatment |
| | SO. | options. Where a subject does not wish to attend further clinic |
| ું | ř | visits, a PDV visit should be scheduled and consent should be |
| (v) | | requested to perform continued remote follow-up of the subject |
| S LOS OF STATE OF STA | | "off treatment on-study" in line with global amendment 1. |
| Shipment of Drug | 0 | Subjects should provide verbal consent via a telephone call to |
| from Sife to Subjects | | use their personal details to complete the site-to-subject |
| Shipment of Drug<br>from Site to Subjects | | shipment request. Consent must be documented in the subject's medical records and preferably confirmed in writing via an email or other written means (eg, via post). |

| | Safety Labs | Where central analysis is not possible, local testing is |
|---|---|---|
| | | permitted. Lab normal ranges would need to be made available. |
| | | o In the event that routine safety lab tests are missed due to |
| | | temporary inability of subject to get to site due to COVID-1950<br>an unscheduled lab should be done at the subject's next climic |
| | | visit if possible. |
| | Spirometry | <ul> <li>The investigator should request confirmation from the subjects<br/>that they are not aware of having been exposed to COVID-19,</li> </ul> |
| | | that they are not currently infected or infectious, and should |
| | | exercise their medical judgement with respect to this |
| | | information prior to conducting spiromets assessments. Sites |
| | | should continue to follow hygiene and cleaning guidance within the manuals to minimize possible cross-contamination. |
| | | 0 |
| | Subjects with | If a subject has confirmed COMD-19 this is to be reported as |
| | confirmed<br>COVID-19 infection | an AE/SAE, but is not per sea reason to withdraw the subject. |
| | COVID-19 Infection | The investigator should determine whether the subject's IP |
| | | should continue be interrupted, or stopped in accordance with |
| | | the Clinical Study Protocol. |
| | | The investigator should continue to reassess the benefit-risk of |
| | | continued study involvement for a study subject infected with |
| | | compared once the infection has resolved and the subject is no |
| | | longer considered to be infectious. |
| | | The name on his standard on the identified as COVID 10 positive |
| | | a retest must be performed after resolution of symptoms (if |
| | - gi | present). The subject can only be considered for enrollment |
| | 8,00 | 4 weeks after having a negative result. |
| | 200 | |
| | a no | |
| | Rus | |
| | ret. | |
| ۵, | N. C. | |
| % | | |
| This | | should continue be atterrupted, or stopped in accordance with the Clinical Study Protocol. The investigator should continue to reassess the benefit-risk of continued study involvement for a study subject infected with COVID-19. In-clinic visits for this subject should only recompence once the infection has resolved and the subject is no longer considered to be infectious. For new subjects previously identified as COVID-19 positive, a retest must be performed after resolution of symptoms (if present). The subject can only be considered for enrollment 4 weeks after having a negative result. |
| | CONFIDENTIAL AND PRO | PRIETARY 159 of 159 |